

# CARTISTEM® PHASE I/IIa CLINICAL TRIAL PROTOCOL MP-0201-01

**Version 3.2** 

Date: 15 March, 2017

# CARTISTEM® PHASE I/IIa CLINICAL TRIAL PROTOCOL

CARTISTEM® 

| Name of Company: MEDIPOST Co., Ltd. Name of Product: CARTISTEM® (Allogeneic-Unrelated, Umbilical Cord Blood-Derived Mesenchymal Stem Cells, Cultured Ex vivo, Combined with sodium Hyaluronate) Protocol #: MP-0201-01 | | |
|---|---|---|
| Protocol Title | Evaluation of Safety and Exploratory Efficacy of CARTISTEM®, a Cell Therapy Product for Articular Cartilage Defects: A Phase I/IIa Clinical Trial in Patients with Focal, Full-thickness Grade 3-4 Articular Cartilage Defects of the Knee | |
| Clinical Phase | Phase I/IIa | |
| Study Overview | 2.25×10 <sup>7</sup> hUCB-MSC (0.25×10 <sup>7</sup> cells/cm <sup>2</sup> ; 0.5 n | CARTISTEM® will be administered at doses ranging from $0.5 \times 10^7$ to $2.25 \times 10^7$ hUCB-MSC $(0.25 \times 10^7 \text{ cells/cm}^2; 0.5 \text{ mL/cm}^2 \text{ with } 0.5 \times 10^7 \text{ MSC/mL})$ to patients with focal, full-thickness, Grade 3-4 articular cartilage defects of $\geq 2 \text{cm}^2$ in size. |
| | Safety: Patient safety will be assessed step-wise with increasing levels of total hUCB-MSC and HA exposure: a total of 12 patients will be enrolled and treated with CARTISTEM® to evaluate whether dose limiting toxicity (DLT) is detected. DLT is defined as toxicity or adverse event of Grade 3 or higher [80 points or higher for pain] in two or more events at the surgery site among swelling, tenderness, range of motion, and pain in any one visit. DLT is also defined as adverse drug reaction of Grade 3 or higher in the Common Toxicity Criteria Adverse Events (CTCAE), Version 4.0, with the exception of the following events and that they are unresolved for 7 consecutive days, despite medical interventions: ✓ Abnormal results in lab test (Acidosis, Hyponatremia, Hyperbilirubinemia, etc.) ✓ Fatigue, defined as not relieved by rest; limiting self-care ADL ✓ Pain, defined as severe pain; limiting self-care ADL ✓ Headache, defined as severe pain in various parts of the head, limiting self-care ADL | |
| | Fever, defined as > 40.0 degrees C (> 104.0 Initially, 6 patients with lesion sizes of 2-5 cm <sup>2</sup> w (Dosage A); if dose limiting toxicity is not detect after administration, an additional 6 patients, with | vill be enrolled and treated ted during a 12 week period |

CARTISTEM® 

| | 5 cm <sup>2</sup> , will be enrolled and treated (Dosage B) to further evaluate safety. |
|---|---|
| | Efficacy: Efficacy will be evaluated with several validated clinical outcome instruments as primary endpoints as well as non-invasive structural assessment utilizing high-resolution magnetic resonance imaging with cartilage-specific sequences as a secondary endpoint. |
| <b>Objectives:</b> | |
| Primary<br>Objective | To evaluate the safety of CARTISTEM® administration |
| Secondary<br>Objectives | To evaluate the exploratory efficacy (improvement in Clinical Scores and regeneration of defective cartilage as assessed by Radiological images) of CARTISTEM®. |
| Diagnosis and<br>Main Criteria for<br>Inclusion | <ul> <li>Patients must meet the following criteria to be eligible for the study;</li> <li>Patients with an intended- to- treat single focal, full-thickness cartilage defect (ICRS [International Cartilage Repair Society] Grade 3 or 4) of the knee as a result of ageing, trauma, or degenerative diseases.</li> <li>Age ≥ 18 years old</li> <li>Size of the articular cartilage lesion is ≥ 2 cm²</li> <li>Swelling, tenderness and active range of motion ≤ Grade II</li> <li>Joint pain: 20-mm - 60-mm on VAS (Visual Analog Scale) at the time of Screening</li> <li>Appropriate blood coagulation, kidney and liver function laboratory parameters: <ul> <li>PT(INR) &lt; 1.5, APTT &lt; 1.5 × control</li> <li>Creatinine ≤ 2.0 mg/dL, Albumin ≤ trace in urine dipstick test</li> <li>Bilirubin ≤ 2.0 mg/dL, AST/ALT ≤ 100 IU/L</li> </ul> </li> <li>Ligament instability ≤ Grade II</li> <li>Lower extremity alignment within 5 degrees of the neutral weight bearing axis</li> <li>No meniscal surgery within the past 3 months and more than 5mm of meniscal rim remaining</li> <li>Ability and willingness to fully participate in the post-operative rehabilitation program</li> <li>Subject is informed of the investigational nature of this study, voluntarily agrees to participate in the study, and signs an IRB-approved informed consent prior to performing any of the screening procedures</li> </ul> |

CARTISTEM® 

| | • Body Mass Index (BMI) ≤ 35 kg/m <sup>2</sup> |
|---|---|
| Criteria for Exclusion | <ul> <li>Patients who have been treated previously and are asymptomatic</li> <li>Avascular necrosis/ osteonecrosis</li> <li>Autoimmune or inflammatory joint disease</li> <li>History of infection within the past 6 weeks</li> <li>Surgery or radiation therapy within the past 6 weeks</li> <li>Serious medical co-morbidities, which would otherwise contraindicate surgery, as determined by the investigator</li> <li>Currently pregnant or nursing</li> <li>Psychotic diseases, epilepsy, or any history of such diseases</li> <li>Current abuse of alcohol (&gt; 10 drinks weekly) and/or regular exposure to other substances of abuse, currently an active smoker</li> <li>Chronic inflammatory articular diseases such as rheumatoid arthritis</li> <li>Enrolled in any other clinical trials within the past 4 weeks</li> <li>Administered immunosuppressants such as Cyclosporin A or azathioprine within the past 6 weeks</li> <li>Ligament instability &gt; Grade II</li> <li>Uncorrected significant lower extremity malalignment (i.e. &gt; 5 degrees)</li> <li>(sub-) Total meniscectomy (&lt;5mm rim remaining)</li> <li>Corticosteroid or viscosupplementation injection to the affected knee in the past 3 months</li> <li>Principal investigator considers inappropriate for the clinical trial due to any reasons other than those listed above</li> </ul> |
| Number of<br>Patients | 12 patients in total; 6 patients with defect sizes of 2-5 cm <sup>2</sup> followed by 6 patients with defect sizes > 5cm <sup>2</sup> |
| Number of Study<br>Centers | Two |
| Concomitant<br>Treatment | Patients should discuss any medications and therapies they are currently taking with the study doctor. Patients in this trial must not take the following drugs: glucosamine, dietary supplements used as alternative medicine to treat osteoarthritis such as chondroitin sulfate and hyaluronan, systemically administered corticosteroids (Hydrocortisone, Prednisone, Prednisolone, Methylprednisolone, Triamcinolone, Dexamethasone, Paramethasone, Betamethasone, Aldosterone, Fludrocortisone ) and immunosuppressants (Prednisone, Vincristine, Azathioprine, $\gamma$ – globulin, Cyclophosphamide, Chlorambucil, 6-mercaptopurine, Cyclophosphamide + factor XIII, Rh(D) immune globulin, ALG, Actinomycin-D, OKT3, Methotrexate) |

CARTISTEM® 



evaluate for dose limiting toxicity (DLT).

Initially, 6 patients with defect sizes of 2-5 cm<sup>2</sup> will be enrolled in Dosage A and treated with  $0.5 - 1.25 \times 10^7$  hUCB-MSC. If DLT is not detected in any patients by 3 months post-administration (time point for first clinical efficacy evaluation), then additional 6 patients with defect sizes of above 5 cm<sup>2</sup> will be enrolled in Dosage B and treated with  $> 1.25 \times 10^7 \text{ hUCB-MSC}$ to further evaluate safety.

If DLT is detected in 1 or 2 patients during Dosage A, additional 3 patients will be enrolled and assessed at Dosage A. If DLT is detected in 3 or more patients during Dosage A period, the study will be stopped.

In the absence of DLT, a total of 12 patients will, therefore, be evaluated for safety and exploratory efficacy.

**CARTISTEM®** 

| Clinical Trial<br>Material (CTM) | CARTISTEM® (human allogeneic-unrelated umbilical cord blood-derived mesenchymal stem cells, hUCB-MSC, and sodium hyaluronate) CARTISTEM® consists of approximately 7.5 x 10 <sup>6</sup> hUCB-MSC suspended in 1.5 mL medium in one vial, and 60 mg sodium hyaluronate provided as a lyophilized sponge form in a separate vial. The two vials are mixed at the surgical site. Upon admixture of the two vials, the combination forms a viscous gel, which is implanted into the articular cartilage defect. |
|---|---|
| Clinical Trial<br>Material Dosage<br>and<br>Administration | CARTISTEM® will be administered into the articular cartilage defect by open surgery at a dose of 0.5 mL/cm² based upon size of the defect. The CARTISTEM® dosage has been selected based on the results derived from nonclinical studies and prior human experience (see Investigator's Brochure for further information) |
| Surgical<br>Technique | Before application of CARTISTEM®, unstable chondral fragments are debrided using a curet and stable shoulders of healthy surrounding cartilage are created. After adequate removal of the debris, multiple holes are created across the entire articular cartilage defect with a 2~3 mm drill bit spacing the holes approximately 3~5 mm apart. CARTISTEM® is applied onto the drilled holes first, and then throughout the entire cartilage defect. |
| Post-operative rehabilitation | Patients will be started on a continuous passive motion (CPM) device on post-operative day 1 with a range of motion of 0-30 degrees initially. This will be increased by 10 degrees per day as tolerated to a maximum of 0-90 degrees. Patients will undergo CPM treatment for 6 hours per day over 6 weeks. The patient will remain touch-down weight-bearing (TDWB) for 6 weeks, and then advance to full-weight bearing during the next 6 weeks (up to week 12). The patient will refrain from high-impact activities, such as running, during the subsequent 8 to 12 weeks (week 20 – 24). |
| Reference<br>Therapy | The study does not include a reference compound. |
| Approximate Duration of Patient Participation | Each patient will undergo a 6-week screening period for eligibility and a 12-month follow-up observation period for both the primary (safety) and secondary (efficacy) evaluations following administration of CARTISTEM®. Also each patient will undergo a 24-month follow-up visit for a long term patient assessment. |

CARTISTEM® 

| Approximate<br>Duration of<br>Study | The estimated duration of the study for the primary evaluation is approximately 12 months, with an additional 12 month extension for the long-term patient assessment phase. |
|---|---|
| Safety<br>Evaluation | General General safety will be evaluated via the following assessments: AEs, routine clinical laboratory tests (hematology, clinical chemistry, and urinalysis), thrombin generation (PT and aPTT), immunogenicity tests (T cell subset), vital signs, physical exams, ECGs, and MRI for tumorigenicity. |
| | Adverse Events To assess the safety of CARTISTEM®, the course and degree of swelling, tenderness, range of motion and pain will be determined. DLT is defined as toxicity or adverse event of Grade 3 or higher [80 points or higher for pain] in two or more events at the surgery site among swelling, tenderness, range of motion, and pain, in any one visit. DLT is also defined as adverse drug reaction of Grade 3 or higher in the Common Toxicity Criteria Adverse Events (CTCAE), Version 4.0, with the exception of the following events and that they are unresolved for 7 consecutive days, despite medical interventions: ✓ Abnormal results in lab test (Acidosis, Hyponatremia, Hyperbilirubinemia, etc.) ✓ Fatigue, defined as not relieved by rest; limiting self-care ADL ✓ Pain, defined as severe pain; limiting self-care ADL ✓ Headache, defined as severe pain in various parts of the head, limiting self-care ADL ✓ Fever, defined as >40.0 degrees C (> 104.0 degrees F) for > 24 hours |
| Efficacy<br>Evaluation | Primary efficacy outcome parameters will be the postoperative changes in subjective knee function as assessed by IKDC (International Knee Documentation Committee) score at 12 months. For secondary efficacy outcome parameters, patients will answer questionnaires for pain (visual analogue scale, VAS), knee specific outcome instruments (Lysholm knee scoring, and KOOS [Knee injury and Osteoarthritis Outcome Score]). Structural information will be gathered using high-resolution (1.5 or 3 Tesla) magnetic resonance imaging (MRI). |

CARTISTEM® 

# Statistical Methods

General: all safety and efficacy endpoints will be presented for each dose cohort as well as for all patients combined. For safety evaluation, statistical homogeneity between dose groups will be performed. For efficacy evaluation, statistical comparison (difference) between dose groups will be performed.

#### 1) Safety

Safety will be demonstrated with 95% confidence intervals. Adverse events, adverse drug reactions, serious adverse events, and drop-out patients due to AE will be presented with frequency and percentage. Homogeneity between dose groups will be analyzed using person's chi-square test or Fisher's exact test. Descriptive statistics including means, medians, SD (standard deviation), minimum and maximum will be used to demonstrate the other safety endpoints.

# 2) Efficacy

Symptom improvement from the outcome instruments will be demonstrated with means and standard deviations. Efficacy results will also be analyzed for statistical significance using change from baseline at each efficacy endpoint. Statistical difference of continuous variables and categorical variables between dose groups will be compared using t-test and Fisher's exact test, respectively.

## Rationale for Study Population and Number of Patients

CARTISTEM® is administered to the defective joint cartilage region by open surgery. Due to ethical considerations, it is not possible to conduct this type of procedure in a healthy subject. Therefore, no studies in healthy subjects will be performed.

Factors such as number of subjects to acquire statistical data of the effectiveness are not considered as critical in this phase I/IIa study. A small number of subjects generally participate in this stage of clinical study. Accordingly, Dosage A is set based on dose limit of toxicity from non-clinical study and then Dosage B will be administered.

CARTISTEM® 

# **Abbreviations**

| AE | Adverse Event, Adverse Experience |
|---|---|
| ADR | Adverse Drug Reaction |
| ALP | Alkaline Phosphatase |
| ALT(sGPT) | Alanine aminotransferase (serum Glutamic Pyruvic Transaminase) |
| AST(sGOT) | Aspartate aminotransferase (serum Glutamic Oxaloacetic Transaminase) |
| BUN | Blood Urea Nitrogen |
| CK | Creatine Kinase |
| CRP | C-Reactive Protein |
| CTC | Common Toxicity Criteria |
| DLT | Dose Limiting Toxicity |
| ESR | Erythrocyte Sedimentation Rate |
| HCG | Human Chronic Gonadotropin |
| Hb | Hemoglobin Concentration |
| Hct | Hematocrit |
| ICRS | International Cartilage Repair Society |
| IKDC | International Knee Documentation Committee |
| IND | Investigational New Drug |
| KOOS Score | Knee injury and Osteoarthritis Outcome Score |
| LDH | Lactate dehydrogenase |
| MCH | Mean Corpuscular Hemoglobin |
| MCHC | Mean Corpuscular Hemoglobin Concentration |
| MCV | Mean Corpuscular Volume |
| MLR | Mixed Lymphocyte Reaction |
| MTD | Maximal Tolerated Dose |
| NCI | National Cancer Institute |
| PT | Prothrombin Time |
| aPTT | Activated Partial Thromboplastin Time |
| RBC | Red Blood Cell |
| ROM | Range of Motion |
| VAS | Visual Analogue Scale |
| WBC | White Blood Cell |

CARTISTEM® 

# **Table of Contents**

| 1 | T | itle and Development of Phase | 12 |
|---|---|---|---|
| | 1.1 | Study Title | |
| | 1.2 | Developmental Phase | 12 |
| 2 | N | ame and affiliation of principal or coordinating investigators | 12 |
| | | Name and Address of the Research Facilities | |
| | | Names and Titles of the Coordinating Investigator and the Principal Investigators | |
| | | Name and Title of the Clinical Trial Pharmacist | |
| | | Name and Address of the reviewing Institutional Review Board (IRB) | |
| 3 | | ame of the Sponsor | |
| 4 | В | ackground of the Study | 14 |
| | 4.1 | Cartilage defects | |
| | 4.2 | Investigational cellular-surgical combined interventions | 15 |
| | 4.3 | CARTISTEM® (MEDIPOST Cell Therapy Product) | 16 |
| | 4.4 | Sodium Hyaluronate | 17 |
| 5 | P | urpose of the Study | 18 |
| 6 | St | tudy Design | 19 |
| | 6.1 | Study Period | |
| | 6.2 | Subject Selection Criteria | 19 |
| | 6.3 | Number of Subjects | 21 |
| | 6.4 | Administration Dosage | 22 |
| | 6.5 | Dose Escalation | |
| | 6.6 | Definition of Maximum Permissible Dose and Method of Dose Escalation | 26 |
| | 6.7 | Expected Adverse Effects and Usage Considerations | 26 |
| | 6. | .7.1 Expected Adverse Effects | 26 |
| | 6. | .7.2 Usage Considerations | 27 |
| 7 | Ir | nvestigational Product | 27 |
| | 7.1 | Investigational Product | 27 |
| | 7. | .1.1 Trade Name | 27 |
| | 7. | .1.2 Ingredients | 27 |
| | 7. | .1.3 Property | 28 |
| | 7.2 | Route of Administration | 28 |
| | 7.3 | Return and disposal of unused investigational product | 31 |
| 8 | St | tudy Methodtudy Method | 32 |
| | 8.1 | Overview of the Study Design. | 32 |
| | 8.2 | Study Flow Chart | |
| | 8.3 | Concomitant Medications and Concomitant Non-drug Therapies | 36 |
| | 8.4 | Observation and Evaluation Items | 36 |
| | 8. | .4.1 Demographic Background and Medical History of Subjects | 36 |
| | 8. | 4.2 Concomitant Medications | 37 |
| | 8. | .4.3 Evaluation of Adverse Events & Toxicity | 37 |
| | 8. | .4.4 Laboratory Evaluations | 38 |
| | 8. | .4.5 Immunogenicity study | 38 |
| C/ | ARTIST | Page 10 | 0 of 137 |

| 8.4.6 IKDC Score | |
|-------------------------------------------|------------------------|
| 8.4.7 100-mm VAS Evaluation | 39 |
| 8.4.8 Lysholm Score | 39 |
| 8.4.9 KOOS Score | 39 |
| 8.4.10 MRI Assessment | |
| 8.5 Early Discontinuation from the Stud | ly39 |
| 9 Definition of Adverse Events | 40 |
| 9.1 Criteria for Safety Assessment | 40 |
| 10 Statistical Analysis | 41 |
| 10.1 Analysis Populations | 41 |
| 10.1.2 Efficacy Population | 41 |
| 10.2 Analysis of Safety Variables and Sta | tistical Evaluation |
| 10.2.1 Safety Variables | 41 |
| 10.2.2 Analysis of Safety Endpoints | 42 |
| 10.3 Analysis of Efficacy Variables and S | Statistical Evaluation |
| 10.3.1 Efficacy Variables | 42 |
| 10.3.2 Analysis of Efficacy Endpoin | ts |
| 11 Rehabilitation Protocol | 44 |
| 12 References | 48 |
| APPENDIX 1. IKDC score | 51 |
| APPENDIX 2. LYSHOLM SCORE | 54 |
| APPENDIX 3. KOOS KNEE SCORE | <i>2</i> 55 |
| APPENDIX 4. CTCAE(Version 4.0) | 58 |
| APPENDIX 5. IDMC charter | |

CARTISTEM® 

# 1 Title and Development of Phase

1.1 Study Title

Evaluation of Safety and Exploratory Efficacy of CARTISTEM®, a Cell Therapy Product for Articular Cartilage Defects: A Phase I/IIa Clinical Trial in Patients with Focal, Full-thickness, Grade 3-4 Cartilage Defects of the Knee

1.2 Developmental Phase

Phase I/IIa

# 2 Name and affiliation of principal or coordinating investigators

2.1 Name and Address of the Research Facilities

#### **RUSH University Medical Center**

1611 W. Harrison Street, Chicago, IL 60612

#### **Brigham and Women's Hospital**

850 Boylston St., Chestnut Hill, MA 02467

2.2 Names and Titles of the Coordinating Investigator and the Principal Investigators

Coordinating Investigator, Principal Investigator

Brian J. Cole, MD

Professor, Department of Orthopedic Surgery

Professor, Department of Anatomy and Cell Biology

Section Head of Cartilage Restoration Center

Principal Investigator

Andreas H. Gomoll, MD

Assistant Professor, Department of Orthopedic Surgery

2.3 Name and Title of the Clinical Trial Pharmacist

CARTISTEM® consists of umbilical cord blood-derived mesenchymal stem cells (hUCB-MSC; main component) suspended in a transparent pale pink medium and sodium hyaluronate

CARTISTEM® 

(device) intended for cartilage regeneration in patients with cartilage defects or injuries. Unlike other conventional investigational products, the innate biological properties of the living cells in this product limit the shelf-life of the suspension (mixture of hUCB-MSC and HA) to less than 72 hours after preparation. Therefore, the investigational product needs to be delivered to the test site on the day of the actual surgery so that the on-site preparation and administration to the patient can take place shortly after receipt of the two vialed CARTISTEM® components (hUCB-MSC and lyophilized HA). Designation of a clinical trial pharmacist is deemed unnecessary as the unused portion of the investigational product which is ordered and administered on an individual subject basis is to be returned to MEDIPOST after the surgery. Therefore, a clinical nurse is given the role of managing the investigational product under supervision of the principal investigator and the subinvestigators.

Moreover, CARTISTEM® does not require a separate compounding or preparation process of a clinical trial pharmacist as the product can be mixed and used by the principal investigator in the surgery room. Hence, it was decided that it would be acceptable to have an appropriate individual designated by the (principal) investigator order, receive the shipment of, and return the investigational product to the sponsor. Therefore, a clinical nurse is assigned the role of managing the investigational product under the supervision of the investigator.

2.4 Name and Address of the reviewing Institutional Review Board (IRB)

#### The Institutional Review Board at RUSH University Medical Center

Research and Clinical Trials Administration Office

1653 W. Congress Parkway, Chicago, IL 60612

(Mailing Address: 707 S. Wood Street, Lower Level, Chicago, IL 60612)

#### Partners Human research Committee at Brigham and Women's Hospital

116 Huntington Avenue, Suite 1002, Boston, MA 02116

(Website: http://healthcare.partners.org/phsirb)

CARTISTEM® 

# 3 Name of the Sponsor

MEDIPOST Co., Ltd.

21 Daewangpangyo-ro 644-beon-gil, Bungdang-gu, Seongnam-si, Gyeonggi-do 13494, Korea

# 4 Background of the Study

## 4.1 Cartilage defects

Chondral defects or damage to articular cartilage due to accidents, repetitive trauma or arthritis are common disorders. They are major causes of disability, as they can lead to osteoarthritis and they rarely heal spontaneously (e.g., Dragoo et al. 2003, Moore et al. 2005). As the population ages and as more young people participate in active sports, the size of the target patient group is also growing. However, despite ongoing research efforts, clinical products directed at cartilage repair remain limited.

Articular cartilage consists of hyaline cartilage and is a highly differentiated connective tissue covering joint surfaces. It is avascular and alymphatic, and it is sheltered from the immune system. It also has no nerve supply and is therefore not sensitive to early injuries. Articular cartilage also has poor repair properties because there are relatively few cells in the tissue, the metabolic rate is low, and the capacity of chondrocytes to divide and migrate within articular cartilage is restricted by the dense matrix. As a consequence, it is generally agreed that articular cartilage does not repair significantly after damage to the collagen matrix (e.g., Chang et al. 2006, Gelse et al. 2003, Hedrick and Daniels 2003, Katayama et al. 2004, Risbud et al. 2001, Wakitani et al. 2002). Therefore, damage to the tissue as a result of trauma generally progresses to osteoarthritis.

In most cases, the critical limiting step for the induction of spontaneous cartilaginous repair is incomplete and leads to the formation of fibrous, or at best fibrocartilage, tissue – a tissue intermediate of fibrous mesenchyme and cartilage, depending on the location and size of injury. Compared with the native hyaline articular cartilage, fibrous repair tissue has poor mechanical qualities and is prone to fail in the long term (Athanasiou et al. 2001, Chuma et al. 2004, Gelse et al. 2003, Guo et al. 2004, Mizuta et al. 2004, Moore et al. 2005, Otsuka et al. 1997). It is, 

therefore, desirable to develop procedures that allow for improved repair of cartilage defects, as discussed below.

#### 4.2 Investigational cellular-surgical combined interventions

Various different types of treatments are in use, such as drug therapy, arthroscopy, joint replacement surgery, marrow stimulation techniques (drilling, abrasion arthroplasty and microfracture for stimulation of local MSC), periosteal grafts, and autologous chondrocyte transplantation (Athanasiou et al. 2001, Risbud et al. 2001, Smith et al. 2005). However, conventional treatment modalities have not been able to provide complete and sustained resolution of symptoms following damage to the articular cartilage. Despite the numerous techniques available today, complete healing of damaged or defective cartilage or consistent reproduction of normal hyaline cartilage does not occur, and continuous drug administration or secondary surgeries are common. Thus, functional restoration of diseased and damaged human articular cartilage continues to remain one of the most challenging orthopedic problems and the clinical need for cartilage repair/regeneration technologies is undisputed (Athanasiou et al. 2001, Elisseeff 2004, Gelse et al. 2003, Lee et al. 2010, Smith et al. 2005, Yanai et al. 2005).

The latest attempts to develop clinically useful procedures for repairing damaged articular cartilage include the use of cells with the potential for cartilage repair. There are three potential cell types that may be utilized: chondrocytes (already used in the autologous chondrocyte transplantation technique), adult (somatic) stem cells and embryonic stem cells (Barry 2003, Browne et al. 2005, Giannoni et al. 2005, Guo et al. 2004, Otsuka et al. 1997, Yanai et al. 2005).

Chondrocyte implantation has long been considered as a potential treatment and several approaches of chondrocyte implantation are in current clinical use. Implantations of previously isolated and *in vitro* amplified autologous chondrocytes are being performed in current clinical practice. The disadvantages of this procedure are the limited proliferative capacity of adult chondrocytes, the issue of dedifferentiation in culture and required re-differentiation upon implantation, as well as the need for a 2-stage procedure for harvest and implantation.

The use of stem cells is the most recently developed and investigated method. The most promising approaches involve the introduction of MSC /cartilage precursor cells. Bone marrow

CARTISTEM® 

contains non-hematopoietic progenitor cells capable of differentiating into osteoblasts, chondrocytes and adipocytes; because those differentiated cells have mesodermal origin, their bone marrow progenitors have been designated MSC.

The umbilical cord blood is a source of hematopoietic stem cells and is used for hematopoietic stem cell transplantation in patients with diseases such as leukemia, aplastic anemia, and congenital immune deficiency that require allogeneic hematopoietic stem cell transplants. Over 5,000 cases of umbilical cord blood-derived hematopoietic stem cell transplantations have been conducted globally as of 2004, and transplant treatments using umbilical cord blood are expected to increase even further in the future. Umbilical cord blood is blood from the placenta and umbilical cord, which can be easily collected from the umbilical cord after childbirth, and therefore the collection poses no risk of harm to either the mother or the infant. Considering the present US birth rate of about 4,000,000 infants per year, umbilical cord blood is one of the most readily available and non-invasive sources of mesenchymal stem cells. The mesenchymal stem cell found in umbilical cord blood is characterized by its ability to self-replicate as well as its multipotency, or the capability to differentiate into cell lineages that compose bone, cartilage, bone marrow stroma, adipocytes, tendon, neurons, and various other tissues and organs.

Research in MSC has had a rapid acceleration over the past decade and MSC-based therapy has become one of the objects of investigation for a new branch of medicine termed regenerative medicine. This emerging technology shows great promise for producing transplantable cartilage constructs to restore the function of degenerated joints. However, current treatment options using MSC for articular cartilage repair/regeneration are still at an experimental stage of development. Studies with MSC were conducted in various animal models while currently only one clinical investigation and two case reports with MSC are available (e.g., Wakitani et al. 2002, Wakitani et al. 2010).

# 4.3 CARTISTEM® (MEDIPOST Cell Therapy Product)

CARTISTEM® is intended to be used as a single-dose cellular therapeutic agent for cartilage regeneration in human subjects with cartilage defects of the knee as a result of ageing, trauma or

CARTISTEM® 

degenerative diseases.

The CARTISTEM® drug product consists of a combination of human umbilical cord blood-derived mesenchymal stem cells (hUCB-MSC; supplied as a liquid suspension) and lyophilized sodium hyaluronate, provided in separate vials for mixing prior to administration. The packaged drug product will be shipped and stored as two vials, one vial containing approximately 7.5x106 hUCB-MSCs suspended in 1.5 mL medium (alpha-MEM) to be mixed with one vial containing 60 mg sodium hyaluronate (lyophilized). Upon admixture of the two vials, i.e. after distribution of the cells in the hyaluronate polymer, the reconstituted product (5x106 cells/mL; 40 mg/mL sodium hyaluronate) is formed as a viscous gel which is implanted into the cartilage lesion during open surgery. The initial proposed clinical dose is to be 0.5 mL/cm² (approximately 2.5x106 cells and 20 mg HA/cm²). Immune phenotype tests using flow cytometer demonstrated that the hUCB-MSCs are CD45 negative, CD14 negative, HLA-DR negative, CD29 positive, CD73 positive, CD105 positive, and CD166 positive.

hUCB-MSCs, the active ingredient in CARTISTEM®, are expected to induce the regeneration of damaged cartilage tissues by repair of the microenvironment with paracrine effects or by differentiation towards tissue-specific pathways. Sodium hyaluronate is believed to function as a medical device to provide mechanical stability to the hUCB-MSC suspension, enabling the cells to remain at the site of the implantation and not disseminate into adjacent areas.

#### 4.4 Sodium Hyaluronate

Hyaluronic acid is a natural component of the extracellular matrix in cartilage. The glycosaminoglycan is highly conserved and is widely distributed in the body. hUCB-MSCs express cell surface receptors (CD44) that bind to hyaluronic acid. Interaction between cells and the extracellular matrix regulates many biological processes that are important to cartilage homeostasis and repair, including cell attachment, growth, differentiation, and survival (Marcacci et al. 2005, Risbud et al. 2001).

Since the 1970's, hyaluronic acid has been clinically used as a chondroprotective agent (Caplan and Dennis 2006, Watterson and Esdaile 2000). In addition, sodium hyaluronate has been

CARTISTEM® 

FDA approved for the treatment of osteoarthritis of the knee since 1997 (as an orthopedic device – e.g. ORTHOVISC® High Mol, SUPARTZ® Dispo, SYNVISC® (Hylan G-F 20) and HYALGAN®). In 2003, HA was approved for injection into the mid to deep dermis for correction of moderate to severe facial wrinkles and folds (such as nasolabial folds). In all cases, the FDA has regulated the products as medical devices.

The sodium hyaluronate in the CARTISTEM® product is believed to provide a stabilizing function to the MSC enabling them to remain at the site of the implant and not spill over into adjacent areas. In fact, sodium hyaluronate (and its derivatives) has proven to be an ideal molecule for use in the delivery of cellular therapies such as autologous chondrocytes or MSC in cartilage repair helping to keep the implanted cells in place (e.g., Elisseeff 2004, Marcacci et al. 2005, Risbud et al. 2001). In addition, hyaluronic acid has been shown to be both non-toxic and biocompatible (Kasahara et al. 2008). Thus, sodium hyaluronate was considered highly desirable for use as a scaffold in CARTISTEM®. There is currently no evidence that the presence of sodium hyaluronate contributes in any way to the inherent activity of the implanted MSC. Therefore, MEDIPOST considers the sodium hyaluronate to be a device in the final administered CARTISTEM®.

# 5 Purpose of the Study

The primary objective of the proposed single-center phase I/IIa study is to evaluate the safety of CARTISTEM®, an allogeneic-unrelated mesenchymal stem cell (hUCB-MSC) suspension mixed with sodium hyaluronate, at doses ranging from  $0.5 \times 10^7$  to  $2.25 \times 10^7$  hUCB-MSC in patients with articular cartilage defects that are equal or greater than  $2 \text{cm}^2$ .

The secondary objective of the study is to evaluate the efficacy (regeneration of defective cartilage and decrease of pain) of CARTISTEM®.

CARTISTEM® will be administered, as a function of the defect size, at a cell density of  $0.25 \times 10^7$  cells/cm² (0.5 mL/cm² with  $0.5 \times 10^7$  hUCB-MSC/mL) directly into the articular cartilage defect by open surgery.

CARTISTEM® 

A total of 12 patients, initially 6 patients with defect sizes of 2 to 5 cm<sup>2</sup> (Dosage A) followed by an additional 6 patients with defect sizes of above 5 cm<sup>2</sup> (Dosage B), will be enrolled sequentially in 2 groups in order to evaluate whether dose-limiting toxicity (DLT) is detected.

Each patient will undergo a 6-week screening period for eligibility and a 12-month follow-up observation period for both the primary (safety) and secondary (efficacy) endpoints of the study. There is an additional long term follow-up observation visit at 24 months. The estimated total duration of the study is approximately 24 months.

Prior to administration of CARTISTEM®, the defect will undergo debridement, and following appropriate preparation, perforation of the subchondral plate.

CARTISTEM® is applied directly onto the entire defect site.

For use at the clinical site, CARTISTEM® will be provided as a cell suspension and lyophilized sodium hyaluronate in separate glass vials.

In terms of post-operative rehabilitation, patients will be started on a continuous passive motion (CPM) device on post-operative day 1 and refrain from high-impact activities such as running for 20 to 24 weeks.

# 6 Study Design

- 6.1 Study Period
  - 1) 24 months from approval of the clinical trial protocol
  - 2) Recruiting period: 7 months
  - 3) Follow-up period: 12 months from baseline (week 0) to final visit
  - 4) Long term follow-up visit: 24 months following administration of CARTISTEM®
- 6.2 Subject Selection Criteria
  - 1) Inclusion Criteria
  - A. Patients with an intended- to- treat single focal, full-thickness cartilage defect (ICRS [International Cartilage Repair Society] Grade 3 or 4) of the knee as a result of ageing,

CARTISTEM® 

trauma, or degenerative diseases

- B. Age  $\geq$  18 years old
- C. Size of the articular cartilage lesion is  $\geq 2 \text{ cm}^2$
- D. Swelling, tenderness and active range of motion ≤ Grade II
- E. Joint pain: 20-mm 60-mm on VAS (Visual Analog Scale) at the time of Screening
- F. Appropriate blood coagulation, kidney and liver function laboratory parameters:
  - ✓ PT(INR) < 1.5, APTT <  $1.5 \times control$
  - ✓ Creatinine  $\leq$  2.0 mg/dL, Albumin  $\leq$  trace in urine dipstick test
  - ✓ Bilirubin  $\leq 2.0 \text{ mg/dL}$ , AST/ALT  $\leq 100 \text{ IU/L}$
- G. Ligament instability ≤ Grade II
- H. Lower extremity alignment within 5 degrees of the neutral weight bearing axis
- I. No meniscal surgery within the past 3 months and more than 5mm of meniscal rim remaining
- J. Ability and willingness to fully participate in the post-operative rehabilitation program
- K. Subject is informed of the investigational nature of this study, voluntarily agrees to participate in the study, and signs an IRB-approved informed consent prior to performing any of the screening procedures
- L. Body Mass Index (BMI)  $\leq 35 \text{ kg/m}^2$
- 2) Exclusion Criteria
- A. Patients that have been treated previously and are asymptomatic
- B. Avascular necrosis / osteonecrosis
- C. Autoimmune or inflammatory joint disease
- D. History of infection within the past 6 weeks
- E. Surgery or radiation therapy within the past 6 weeks
- F. Serious medical co-morbidities which would otherwise contraindicate surgery, as determined by the investigator
- G. Currently pregnant or nursing
- H. Psychotic diseases, epilepsy, or any history of such diseases

CARTISTEM® 

- I. Current abuse of alcohol (> 10 drinks weekly) and/ or regular exposure to other substances of abuse; currently an active smoker
- J. Chronic inflammatory articular diseases such as rheumatoid arthritis
- K. Enrolled in any other clinical trials within the past four weeks
- L. Administered immunosuppressants such as Cyclosporin A or azathioprine within the past 6 weeks
- M. Ligament instability > Grade II
- N. Uncorrected significant lower extremity malalignment (i.e. > 5 degrees)
- O. (Sub-) Total meniscectomy (<5mm rim remaining)
- P. Corticosteroid or viscosupplementation injection to the affected knee in the past 3 months
- Q. Principal investigator considers inappropriate for the clinical trial due to any reasons other than those listed above

#### 6.3 Number of Subjects

1) Estimated Number of Patients

This study requires 12-18 patients (6-9 patients per arm depending on rate of DLT) for two different dose ranges (Dosage A: defect sizes of 2-5 cm<sup>2</sup> and Dosage B: defect sizes of above 5 cm<sup>2</sup>).

2) Target Number of Subjects and Rationale

This is a phase I/IIa clinical trial to evaluate safety and exploratory efficacy of the investigational drug product. Therefore, it is not considered critical to base the number of subjects on formal statistical power calculations. Six patients at each dose cohort enrolled sequentially are considered sufficient for this study. This study will be performed with two dose ranges, on the basis of existing pre-clinical test results. Initially, 6 patients with defect sizes of 2-5 cm<sup>2</sup> will be enrolled in Dosage A. If no DLT is seen during Dosage A, another 6 patients with larger defect sizes (above 5 cm<sup>2</sup>) will be recruited for Dosage B of the study. There could be a need for an intermediate dose or up to 6 additional patients, based on the rate of DLT seen.

CARTISTEM® 

#### 6.4 Administration Dosage

#### 1) Initial Administration Dosage and Rationale

It is somewhat well understood by developers and regulators of living cell therapies that for products like CARTISTEM® administered locally into an anatomical defect there is no simple extrapolation of a safe starting dose in humans based primarily upon body surface area calculations derived from animal studies.

In addition, dose determinations in this clinical setting should take into account the surface area of the cartilage defect such that all NOAEL values should be converted into a unit quantity (cells/cm<sup>2</sup>) at the application site. This approach applies to most therapeutics administered into anatomical compartments that have little subsequent distribution outside of the compartment; it is recommended that doses are normalized between species according to the compartmental volumes and amount of the therapeutic product.

Support for the range of CARTISTEM® doses  $(0.5 \times 10^7 \text{ cells to } 2.25 \times 10^7 \text{ cells})$  to be evaluated for safety and efficacy in this phase I/IIa study comes from both preclinical studies and clinical results in humans (comprised of a completed Phase I/II study in Korean patients with articular cartilage defects (N=7) and an ongoing Phase III study in Korean patients (N=50), as follows:

NOAELs for CARTISTEM® have been determined in the rat (Study No. B04001; NOAEL =  $3x10^7$  cells per mL; >  $1x10^7$  cells per cm²) and the rabbit (Study No. B04004; NOAEL =  $1.5x10^7$  cells per mL; >  $0.3x10^7$  cells per cm²); however, it is possible that the design of these studies did not allow for a proper assessment of the NOAEL due to limitations on the density of cells administered, and an overall very low toxicity of the hUCB-MSC in the species examined.

No treatment-related SAEs have been reported in seven patients who participated in a phase I/II Korean study and 50 patients currently enrolled in an ongoing phase III Korean study; all of these patients have received single administrations of  $0.25 \times 10^7$  cells/cm<sup>2</sup> (0.5 ml/cm<sup>2</sup> with  $0.5 \times 10^7$  MSC/mL) up to a maximum of  $2.25 \times 10^7$  total MSC; this number of cells represents a much higher dose than the NOAEL ( $10 \times 10^7$  MSC per mL) derived from

CARTISTEM® 

Study B04001 (GLP repeat-dose toxicology study in rats).

Based on these findings (for further discussion, please see the Investigator's Brochure), MEDIPOST has selected a single administration of CARTISTEM® at  $0.25 \times 10^7$  cells/cm<sup>2</sup> (0.5 mL/cm<sup>2</sup> with  $0.5 \times 10^7$  hUCB-MSC/mL), with both the volume and total number of hUCB-MSC administered to patients being a function of the defect size.

Similar products available on the market include CARTICEL® manufactured by Genzyme Biosurgery, an autologous cultured chondrocyte product approved by the US-FDA. Clinical studies of CARTICEL® were conducted at dose levels ranging from 0.64×10<sup>6</sup> cells/cm² up to 3.3×10<sup>6</sup> cells/cm² for the 1.2×10<sup>7</sup> cells/0.4mL product. Meanwhile, Chondron, the autologous chondrocyte regeneration therapy of Cellontech, Korea, is a 1.2×10<sup>7</sup> cells/0.4mL product which is applied at a ratio of 0.1 mL for every 1 cm² of cartilage defect. For cartilage defects greater than 4 cm² in size, the entire vial is administered.

Both CARTICEL® and Chondron are autologous chondrocyte therapies, with limits in cell proliferation and maximum number of cells that can be achieved in the defect. In other words, the limited cell number is a challenge and it is difficult to determine a constant cell concentration per unit area in larger defect sizes. Also, there are potentially large differences in cell potency since the starting materials/living cells are derived in a patient-specific manner and, therefore, typically vary greatly from patient to patient.

CARTISTEM® can be differentiated from these two products because it is an off-the-shelf allogeneic-unrelated cellular therapy that allows a consistent application of the most effective cell concentration per area of defect throughout the entire lesion with a constant cell concentration.

Against this background, the most scientific and logical approach for the study would be to perform the clinical trial using two different cell concentrations of  $0.5 \times 10^7$  cells/mL and  $1.0 \times 10^7$  cells/mL. However, it was deemed ethically inappropriate to subject a treatment group to a relatively-less effective dose. Therefore, a single cell concentration expected to be the more effective of the two was first chosen through a preclinical study and adopted for CARTISTEM®

this clinical trial. The total volume of administration was determined by size of the lesion.

CARTISTEM<sup>®</sup>, consisting of mesenchymal stem cells and sodium hyaluronate, will be applied at a dose of 0.5 mL/cm<sup>2</sup>. The administered dose is, therefore, a function of the defect size. It will be administered into the cartilage defect by open surgery.

The following chart provides determination of CARTISTEM® dosage relative to the defect size (derived from nonclinical studies and prior human experience):

| Study<br>Phase | <b>Defect Size</b> | Volume of Dose | Total Cell Number<br>(hUCB-MSC) | Device Dosage<br>(Sodium hyaluronate) |
|---|---|---|---|---|
| | 2 cm <sup>2</sup> 1.0 | | $0.5 \times 10^7$ cells | 40 mg |
| A | 3 cm <sup>2</sup> | 1.5 mL | $0.75 \times 10^7$ cells | 60 mg |
| 71 | 4 cm <sup>2</sup> | 2.0 mL | $1.0 \times 10^7$ cells | 80 mg |
| | 5 cm <sup>2</sup> | 2.5 mL | $1.25 \times 10^7$ cells | 100 mg |
| | 6 cm <sup>2</sup> | 3.0 mL | $1.5 \times 10^7$ cells | 120 mg |
| В | 7 cm <sup>2</sup> | 3.5 mL | $1.75 \times 10^7$ cells | 140 mg |
| | 8 cm <sup>2</sup> | 4.0 mL | $2.0 \times 10^7$ cells | 160 mg |
| | 9 cm <sup>2</sup> ~ | 4.5 mL ~ | $2.25 \times 10^7 \text{ cells} \sim$ | 180 mg ~ |

#### 6.5 Dose Escalation

This clinical trial will employ the following dose escalation scheme:

A total of 12-18 patients will be enrolled and treated with CARTISTEM® for dose limiting toxicity (DLT) evaluation. Initially, 6 patients with lesion sizes of 2 – 5 cm² will be assigned to Dosage A and treated with 0.5 – 1.25x10<sup>7</sup> MSCs; if dose limiting toxicity is not observed at the 3 month time point for the first clinical efficacy evaluation, then another 6 patients with lesion sizes of above 5 cm² will be assigned to Dosage B and treated with more than 1.25 x 10<sup>7</sup> MSCs for further safety evaluation. If a DLT occurs to one or two patients of the group treated with the dosage A, 3 more patients will be assigned to dosage A. If DLT happens to 3 of the patients who were treated with the dosage A or above, this study will be halted and the FDA and IRB will be notified. The Independent Data Monitoring Committee will perform a comprehensive review of safety (see Section 9.1).

CARTISTEM® 

If no DLT occurs to any of the dosage A patients, another 6 patients with larger defect sizes will be enrolled and assigned to dosage B. In case of no DLT observed, a total of 12 patients will be enrolled for safety and efficacy evaluation. However, 18 patients could be enrolled if DLT occurs to two patients. If DLT occur 3 or more patients treated with Dosage B, this study will be halted and the FDA and IRB will be notified. The Independent Data Monitoring Committee will perform a comprehensive review of safety (see Section 9.1).



CARTISTEM® 

**Dose Limiting Toxicity (DLT):** DLT is defined as toxicity or events of Grade 3 or higher (80 points or higher against pain) in two or more events at the surgery site among swelling, tenderness, range of motion, and pain in any one visit. DLT is also defined as adverse drug reaction of Grade 3 or higher in the Common Toxicity Criteria Adverse Events (CTCAE), Version 4.0, with the exception of the following events and that they are unresolved for 7 consecutive days, despite medical interventions:

- ✓ Abnormal results in lab test (Acidosis, Hyponatremia, Hyperbilirubinemia, etc.)
- ✓ Fatigue, defined as not relieved by rest; limiting self-care ADL
- ✓ Pain, defined as severe pain; limiting self-care ADL
- ✓ Headache, defined as severe pain in various parts of the head, limiting self-care ADL Fever, defined as > 40.0 degrees C (> 104.0 degrees F) for > 24 hours

<u>Maximum Tolerated Dose (MTD):</u> If DLT occurs in 2 or fewer patients at the Dosage B level, the MTD will be Dosage B. If DLT occurs in 3 or more patients treated with Dosage B then the MTD will be Dosage A. If DLT occurs in 3 patients treated with Dosage A then the MTD will not have been determined in this study design.

#### 6.7 Expected Adverse Effects and Usage Considerations

#### 6.7.1 Expected Adverse Effects

There has not been any expected adverse effect that is directly related to the administration of CARTISTEM®, however, mild increase in temperature, pain, nausea, and headache may occur in a response to the administration of allogenic mesenchymal stem cells. In general, adverse effects that may be observed following arthrotomy accompanied by the use of anesthesia include the followings:

- Implant site pain, pruritus, and warmth
- Nausea

**CARTISTEM®** 


- Constipation
- Dyspepsia
- Headache
- Dysuria
- Dizziness

#### 6.7.2 Usage Considerations

- 1) Sterility should be strictly maintained as the product involves injection into human knee joint cavity.
- 2) Should any serious adverse events occur during the administration period or within 14 days after final injection, the principal investigator must, regardless of whether or not the adverse reaction is thought to be related to the study drug, report the incident to the clinical trial review committee and MEDIPOST Co., Ltd. personnel within 24 hours of occurrence.
- 3) This drug should not be administered intravenously.
- 4) Before mixing the constituting substances of the drug, tap the vial with the fingers to make sure that the cells and the preserving solution mix properly. Do not vortex.
- 5) In order to prevent the intrusion of any foreign materials into the syringe, wipe the needle point and insertion area of the vial with ethanol before inserting the needle into the vial.

# 7 Investigational Product

7.1 Investigational Product

#### 7.1.1 Trade Name

**CARTISTEM®** 

#### 7.1.2 Ingredients

- hUCB-MSCs: Human umbilical cord blood-derived mesenchymal stem cell suspension in pale pink and transparent medium
- Sodium hyaluronate: white or gray-white lyophilized sponge form

CARTISTEM® 

# 7.1.3 Property

A viscous gel matrix formed by mixing umbilical cord blood-derived mesenchymal stem cell suspension and white lyophilized sodium hyaluronate

#### 7.1.4 Storage and Handling Conditions

- Storage condition: 2 10 °C (36 50 °F)
- Shelf-life of hUCB-MSC suspension: 72 hours from the time of manufacturing
- CARTISTEM® after combining with sodium hyaluronate is recommended to use within 12 hours from time of the combination.

#### 7.2 Route of Administration

- 7.2.1. Anesthetize a patient.
- 7.2.2. Gently finger-tap hUCB-MSC vial to mix and transfer 1.5 mL of the cell suspension using a sterile syringe to the HA vial. Gently mix using a sterile spatula and leave the mixture stationary until the sodium hyaluronate is completely swollen for at least 30 minutes at room temperature.
  - 7.2.3. Perform arthroscopy to obtain more accurate measurement of the defect size.
- 7.2.4. Expose the cartilage defect through routine knee arthrotomy, based on defect location (medial or lateral parapatellar arthrotomy).

CARTISTEM® 



7.2.5. Debride the cartilage defect back to stable shoulders using a curet to remove any unstable or degenerated (soft and fissured) cartilage, following standard guidelines as used for microfracture or autologous chondrocyte implantation. After debridement, measure size of the defect to calculate required the dose of CARTISTEM®.

CARTISTEM® 



- 7.2.6. Create multiple holes across the entire base of the articular cartilage defect with a 2~3mm drill bit spacing the holes approximately 3~5 mm apart. If active bleeding is encountered, the defect may be packed with epinephrine soaked sponges. Alternatively, thrombin (5000 Units) or thrombin spray may be used. The defect base should be without any active bleeding at the time of implantation.
  - 7.2.7. Fill the holes with CARTISTEM® first and across the entire cartilage defect.
  - 7.2.8. Deflate the tourniquet, achieve hemostasis, and close the wound.
  - 7.2.9. Put a knee immobilizer and a standard cold-therapy device onto the leg of a patient.

CARTISTEM® 



# 7.3 Return and disposal of unused investigational product

After administration of CARTISTEM®, the amount of any empty containers or remaining drug shall be documented on a designated form and returned to the Contract Manufacturing Organization (CMO).

The CMO will then verify the amount of any remaining drugs indicated on the form and store them frozen for one year after its receipt of the returned investigational product. Thereafter, the CMO will dispose the returned drug per its operating procedure.

CARTISTEM® 

# 8 Study Method

8.1 Overview of the Study Design

This study is a phase I/IIa open-label clinical trial with the objective of assessing the safety and exploratory efficacy of a single administration of CARTISTEM®, an allogeneic-unrelated umbilical cord blood-derived mesenchymal stem cell product, in patients with articular cartilage defects.

CARTISTEM® 

# 8.2 Study Flow Chart

| | Screening (Week – 6~Week 0) | Baseline (Day -2) (±2d) | Treatment (Day 0) | Week 2 (±5d) | Week 4 (±5d) | Week 8<br>(±5d) | Week 12<br>(±7d) | Week 24<br>(±14d) | Month 12 (±30d) | Month 24 (±30d) |
|---|---|---|---|---|---|---|---|---|---|---|
| Visits | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Informed Consent | • | | | | | | | | | |
| Physical Examination <sup>1)</sup> | • | | | • | • | • | • | • | • | • |
| Medical History,<br>Medication History <sup>1)</sup> | • | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | • | | | | | | | | | |
| Pregnancy Test (Serum HCG) | • | • | | | | | | | | |
| Vital Signs/Temperature | • | • | • | • | • | • | • | • | • | • |
| Laboratory Tests <sup>2)</sup> | <b>3</b> ) | | | <b>4</b> ) | • | • | • | • | • | |
| Immunogenicity tests (T cell subset) | <b>•</b> 5) | | | | | | | • | | • |
| X-ray of the Joint | • | | | | | | | | | |
| MRI (T2 mapping) | <b>6</b> ) | | | | | | | • | <b>1</b> 7) | <b>1</b> 7) |
| Administration of the Investigational Product <sup>8)</sup> | | | • | | | | | | | |
| IKDC Score <sup>9)</sup> | • | • | | | • | • | • | • | • | • |

CARTISTEM® 

| | Screening (Week – 6~Week 0) | Baseline<br>(Day -2)<br>(±2d) | Treatment (Day 0) | Week 2 (±5d) | Week 4 (±5d) | Week 8 (±5d) | Week 12 (±7d) | Week 24 (±14d) | Month 12 (±30d) | Month 24 (±30d) |
|---|---|---|---|---|---|---|---|---|---|---|
| Lysholm Score | | • | | | • | • | • | • | • | • |
| KOOS Score | | • | | | • | • | • | • | • | |
| 100-mm VAS<br>Evaluation <sup>10)</sup> | | • | | <b>1</b> 11) | • | • | • | • | • | • |
| Check for Concomitant<br>Medications | | • | | • | • | • | • | • | • | • |
| Check for Adverse<br>Events/Toxicity | | | | • | • | • | • | • | • | • |

- 1) Name, gender, date of birth, address, height, body weight, medical history, concomitant medications
- 2) Hematology: Hematocrit, Hemoglobin, MCV, MCH, MCHC, RBC, WBC, Platelet, Differential count (Neutro, Eosino, Baso, Lympho, Mono)

Blood Chemistry: GOT (AST), GPT (ALT), Alkaline Phosphatase, Glucose, Urea (BUN), Creatinine, Direct bilirubin, CK, LDH, Uric acid, Albumin, and Total Protein

Blood Coagulation: PT, aPTT

Electrolytes: Sodium, Potassium, Chloride

Urinalysis: Color, Specific gravity, pH, Leucocytes, Nitrite, Protein, Glucose, Ketone, Urobilinogen, Bilirubin, RBC, Microscopy

- 3) Lab test at Screening can be used as the pre-treatment baseline.
- 4) Lab Tests for patient at Week 2 can be omitted if the lab tests within the window period for Week 2 (i.e. 9 to 19 days after operation) are available.
- 5) Immunogenicity test at Screening can be used as the pre-treatment baseline.
- 6) MRI (T2 mapping) performed for at Screening may be skipped if MRI (T2 mapping) within the past 6 months is available. MRI (T2 mapping) at Screening can be used as the pre-treatment baseline.
- 7) MRI performed at Week 24 and Months 12 and 24 will also evaluate for tumorigenicity at focal lesion of the knee administration

CARTISTEM® 

site.

- 8) Administration of the Investigational Product: 500 µL/cm<sup>2</sup> of defect size
- 9) From baseline to Week 24, only subjective knee evaluation form must be filled in.
- 10) Use of NSAIDs must be discontinued for 6 weeks prior to treatment and may be resumed following the treatment. Use of NSAIDs and any other analgesics must be discontinued for 48 hours and 24 hours, respectively, prior to VAS evaluation at Weeks 4, 8, 12, and 24, and Months 12 and 24.
- 11) Patient may be allowed to take analgesics within 24 hours prior to VAS evaluation at Week 2.

The subject must visit the center on the scheduled visitation date $\pm 5$  days for Week 2, 4, and 8;  $\pm 7$  days for Week 12,  $\pm 14$  days for Week 24 after the administration of the investigational product. For the long term follow-up patient assessment, the subject must visit the center on the scheduled visitation date $\pm 30$  days at Months 12 and 24.

CARTISTEM® 

#### 8.3 Concomitant Medications and Concomitant Non-drug Therapies

Concomitant treatment with systemic corticosteroids or immunosuppressants is not permitted, but co-administration of any other drugs that have no effect on the efficacy assessment is allowed. If there is a concomitant medication, the name of the drug's active ingredient (name of the product in case of a combination drug), dosage, starting/ending date of administration, and the reasons for administration are to be recorded on the case report form (CRF). Information on any concurrent therapies (ex: physiotherapy) are also required to be documented on the CRF (type, duration, etc.). All concomitant medications and therapies are to be recorded at baseline and during the trial.

The following drugs are not permitted: glucosamine, dietary supplements used as alternative medicine to treat osteoarthritis such as chondroitin sulfate and hyaluronan, systemically administered corticosteroids (Hydrocortisone, Prednisone, Prednisolone, Methylprednisolone, Triamcinolone, Dexamethasone, Paramethasone, Betamethasone, Aldosterone, Fludrocortisone ) and immunosuppresant (Prednisone, Vincristine, Azathioprine,  $\gamma$ – globulin, Cyclophosphamide, Chlorambucil, 6-mercaptopurine, Cyclophosphamide + factor XIII, Rh(D) immune globulin, ALG, Actinomycin-D, OKT3, Methotrexate

#### 8.4 Observation and Evaluation Items

#### 8.4.1 Demographic Background and Medical History of Subjects

The patients will be screened by survey of demographic background and medical history to determine their eligibility for enrollment.

- ✓ Demographic background: the patient's initials, date of birth, age, gender, body weight, height, ethnicity, etc.
- ✓ Medical history: the patient's current or past diseases of substantial significance
- ✓ Vital Signs and Physical Examination: vital signs will be monitored and recorded at screening, after administration of the investigational product, and at each follow-up visit.
- ✓ Vital signs: blood pressure, pulse
- ✓ Physical examinations: general condition, nutritional condition, skin/mucosa, eye, ENT, thyroids, lungs, cardiovascular system, abdomen, kidney, spine/extremities,

CARTISTEM® 
peripheral circulation, neuro-psychiatric system, lymphatic system, etc

#### 8.4.2 Concomitant Medications

Each participating subject must be inquired at baseline and throughout the treatment period and at each follow up visit whether he or she is on any concomitant medications. And detailed information of the medication such as the name of the drug's active ingredients (name of the product for a combination drug), dosage, start and end dates of the administration, and a reason for the administration should be documented on case report form.

#### 8.4.3 Evaluation of Adverse Events & Toxicity

Any adverse events (AE) or toxic reactions of each participating subject will be evaluated throughout the course of the study and at each follow up visit (from Day -2 to the end-of-study visit). Any adverse events or serious adverse events will be managed, investigated, and reported according to the procedures described in the following sections:

## ✓ Adverse Events

When an adverse event is either observed by the investigator or reported by a subject, the investigator, regardless of the relationship of the AE to the investigational product, will record name and type of the adverse event, the severity, dates of onset and resolution of the event, the investigator's opinion on the relationship between the investigational product and the adverse event, and whether or not the event was an SAE (serious adverse event) on the case report form (CRF).

The principal investigator or the trial coordinator will carry out follow-up observations for all subjects with adverse events until the symptoms subside and the abnormal clinical test results are returned to normal, or until a satisfactory explanation can be given for the observed changes. If and when there is such a request from the sponsor, a progress report on the adverse event will be submitted to the trial coordinator.

# ✓ Serious Adverse Events

A serious adverse event is defined as any untoward medical occurrence at any dose that causes death, life-threatening condition, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another important medical event (see below).

CARTISTEM® 

Important medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in in-patient hospitalization, or development of drug dependency or drug abuse. If a serious adverse event occurs, the investigator must, regardless of the relationship of the SAE to the investigational product/treatment, report the event to the responsible Institutional Review Board/Independent Ethics Committee and to the sponsor within 24 hours of awareness of the event by the investigator or, at the latest, by the next working day.

If an unexpected fatal or life-threatening adverse event occurs, the sponsor must report to the FDA by telephone or fax within seven days and report in writing of unexpected and serious adverse events within 15 days as required under 21CFR312.32.

# 8.4.4 Laboratory Evaluations

Laboratory evaluations will be performed at screening, after final administration of the investigational product and at every follow-up visit.

- 1) Hematology: Hematocrit, Hemoglobin, MCV, MCH, MCHC, RBC, WBC, Platelet, Differential count (Neutro, Eosino, Baso, Lympho, Mono)
- 2) Blood Chemistry: GOT(AST), GPT(ALT), Alkaline Phosphatase, Glucose, Urea(BUN), Creatinine, Direct bilirubin, CK, LDH, Uric acid, Albumin, Total Protein
- 3) Blood coagulation test: PT, aPTT
- 4) Electrolytes: Sodium, Potassium, Chloride
- 5) Urinalysis: Color, Specific gravity, pH, Leucocytes, Nitrite, Protein, Glucose, Ketone, Urobilinogen, Bilirubin, RBC, Microscopy

# 8.4.5 Immunogenicity study

T cell subset for immunogenicity evaluations will be performed at Screening, at 24-week 12-month, and 24-month visit.

#### 8.4.6 IKDC Score

CARTISTEM® 

The subjects will undergo a self-assessment of knee function using IKDC subjective knee evaluation score before and after the drug administration in order to determine the efficacy of the investigational product. The IKDC assessment will be performed at the 4, 8, 12, 24 weeks and 12 and 24 months after the drug treatment in an exploratory fashion but the IKDC score from the 12 month time point will be used as a primary result of the post-operative change.

#### 8.4.7100-mm VAS Evaluation

The subjects will undergo a self-assessment of joint pain using 100 mm VAS before and the 2, 4, 8, 12, 24 weeks and 12 and 24 months after the drug administration for the efficacy evaluation. Use of NSAIDs must be discontinued for 6 weeks prior to treatment and may be resumed following the treatment. Use of NSAIDs and any other analgesics must be discontinued for 48 hours and 24 hours, respectively, prior to VAS evaluation at Weeks 4, 8, 12, and 24, and Months 12 and 24. Patient may be allowed to take analgesics within 24 hours prior to VAS evaluation at Week 2.

#### 8.4.8 Lysholm Score

The subjects will undergo a self-assessment of knee function using Lysholm Score before and the 4, 8, 12, 24 weeks and 12 and 24 months after the drug administration for the efficacy evaluation.

#### 8.4.9 KOOS Score

The subjects will undergo a self-assessment of knee function and knee-related quality-of-life (QoL) using KOOS Score before and the 4, 8, 12, 24 weeks and 12 and 24 months after the drug administration for the efficacy evaluation.

#### 8.4.10 MRI Assessment

Structural information will be gained using high-resolution (1.5 or 3 Tesla) magnetic resonance imaging (MRI) at Screening, week 24, month 12, and month 24 in order to evaluate the clinical symptom improvement. The MRI evaluations at week 24, month 12 and month 24 will also evaluate for tumorigenicity at focal lesion.

#### 8.5 Early Discontinuation from the Study

Drop-out or withdrawal of a subject from the study can be determined at any time point during the study period by reporting to the trial coordinator or the principal investigator.

CARTISTEM® 

Should a patient voluntarily decide to withdraw, the decision will be respected and accepted without any questions.

Purpose of this study is to evaluate the safety and the efficacy of the investigational product. Therefore, any subjects who want to withdraw from the study on a voluntary basis or due to the adverse events will be replaced with new subjects as long as the drug administration in the dosage group that the withdrawn subject was in is not complete. The study data obtained from such a subject until the point of drop out will be, where possible, included in the data pool for analysis at the final evaluation stage.

#### 9 Definition of Adverse Events

An adverse event (AE) is defined as any undesired clinical responses or complication experienced by a subject. All operative and postoperative adverse events, whether related or not, will be documented on the AE case report form (CRF).

# 9.1 Criteria for Safety Assessment

Vital sign monitoring, physical examination (swelling, tenderness, range of motion, and pain), and laboratory evaluations will be carried out to determine the safety of the investigational product. When an adverse event occurs, the type, the severity, dates of the onset and resolution of the adverse event, and the relationship between the investigational product and the adverse event will be investigated and documented on the case report form.

Causality of the adverse events will be determined according to the following criteria:

- ✓ Not related: the adverse experience is definitely not related to the investigational product
- ✓ Unlikely: there are other, more likely causes and the investigational product is not suspected as a cause
- Suspected, reasonable possibility: the direct cause and effect relationship between the drug and the adverse event has not been demonstrated but there is a reasonable possibility that the event was caused by the drug.
- ✓ Probable: there probably is a direct cause and effect relationship between the adverse event and the investigational product

CARTISTEM® 

Certainty of causal relationship between the adverse event and the investigational product (or any other reasons – progression of an underlying disease, concomitant therapy, etc.) will be determined on the basis of how well the adverse event could be explained in light of the following factors:

- ✓ Known pharmacological effect and mechanism of the investigational product
- ✓ Similar events previously reported for the investigational product or other substances of the same class
- ✓ Drug reactions frequently reported with similar medications
- ✓ Events that are temporally associated with the investigational product (events that are resolved once the drug is discontinued but reappear with the next administration)

The study will be under ongoing periodic reviews by an assigned Independent Data Monitoring Committee (IDMC). An IDMC will independently review data on a periodic basis as detailed in the IDMC charter. Serious AEs will be reported to the IDMC as outlined in the IDMC charter. The IDMC will make recommendations to the Sponsor as to whether the trial should be revised or closed.

# 10 Statistical Analysis

#### 10.1 Analysis Populations

#### 10.1.1 Safety Population

The safety analysis for all clinical and laboratory adverse experiences will be based on all enrolled patients who are administered the investigational product.

#### 10.1.2 Efficacy Population

The efficacy population will be defined as all patients who met the eligibility criteria and received at least one dose of the investigational product, and had been assessed at least once for at least one efficacy endpoint.

#### 10.2 Analysis of Safety Variables and Statistical Evaluation

# 10.2.1 Safety Variables

All adverse events will be coded according to the latest version of MedDRA and the classification according to the System Organ Class of MedDRA using preferred term.

All adverse events will be summarized and analyzed.

CARTISTEM® 

Serious adverse events and drop-out patients due to adverse events will be described in details.

Descriptive statistics including means, medians, SD (standard deviation), minimum and maximum will be used to present the other safety endpoints, laboratory tests including routine hematology and chemistry, thrombin generation (PT and aPTT), vital signs, autoimmune disease test (T-cell subset) and ECGs. For laboratory data, the number of subjects who deviated from the normal range will be presented for each analyte, by visit, and by dosage phase. The results will be also classified into normal, decreased, or increased in relation to the normal range.

## 10.2.2 Analysis of Safety Endpoints

Analysis of the adverse events, adverse drug reactions, and serious adverse events will be presented with number of case (# of subject who experienced), number of adverse events, and percentage.

Analysis of the adverse events will include the severity, the seriousness and the relationship with the study medication. It will be presented with number of event and percentage.

Incidence rates of the adverse events including adverse drug reactions and serious adverse events occurred in each dose group will be presented with frequency, percentage, and 95% confidence interval of the rates. Homogeneity between dose groups will be analyzed using person's chi-square test or Fisher's exact test.

Incidence rates of the adverse drug reaction by SOC between two dose groups will be analyzed for homogeneity using pearson's chi-square test or Fisher's exact test.

#### 10.3 Analysis of Efficacy Variables and Statistical Evaluation

#### 10.3.1 Efficacy Variables

Data such as subjective knee function of each category will presented using criteria for the IKDC, the Lysholm score and the KOOS assessment, and the improvement level of pain will be analyzed using the 100-mm VAS. Structural information will be gained through the use of high-resolution (1.5 or 3 Tesla) magnetic resonance imaging (MRI) with cartilage-specific sequences (T2-mapping).

✓ Primary efficacy endpoint: post-operative change in subjective knee function will be obtained from the IKDC score at the 12-month time point as the primary

CARTISTEM® 

efficacy endpoint.

- ✓ Secondary efficacy endpoint: the Lysholm Score and the KOOS score will be used as the secondary efficacy endpoint to measure post-operative change of the knee function.
- ✓ Improvement degree of joint pain will be measured using a 100-mm VAS (Visual Analogue Scale).
- ✓ Grade of the cartilage regeneration and morphological constitution of the cartilage repair area will be assessed using high-resolution (1.5 or 3 Tesla) magnetic resonance imaging (MRI).

#### 10.3.2 Analysis of Efficacy Endpoints

The descriptive statistics of the categorical variables will be presented with percentage and frequency and that of the continuous variables such as mean, median, standard deviation, and interquartile range. The primary efficacy endpoint will be analyzed using the t-test. As for the secondary efficacy endpoints, differences of the continuous variables and the categorical variables between the two groups will be analyzed using the t-test and Fisher's exact test, respectively.

CARTISTEM® 

# 11 Rehabilitation Protocol

All patients must participate in the following standardized rehabilitation program after receiving treatment. Rehabilitation program will vary according to the defect location of each subject.

Stage 1- Proliferative Phase (Week 1 to 6)

# **Femoral Condyle Defect**

#### **PRIMARY GOALS**

DO NOT OVERLOAD GRAFT
INCREASE TIBIOFEMORAL AND PATELLOFEMORAL MOBILITY
RESTORE QUADRICEPS CONTROL

| R | R | A | $\boldsymbol{C}$ | R |
|---|---|---|------------------|---|

• Knee immobilizer with ambulation, until good quads control/SLR (approximately Week 3 to 6)

#### **GAIT**

Heel-toe TDWB with crutches

#### **ROM**

- Full AROM and gentle AAROM.
- CPM ≥ 6 to 8 hours daily for 6 weeks. Start at 0-40 degrees, progress range as tolerated.
- Goal: minimum 90 degrees flexion for the first 2 weeks, 110 degrees for the next 4 weeks (the 6 week time point of post-op)

#### **THEREX**

- Quad sets, SLR in knee immobilizer as needed, leg curl/heel slides, hip abduction
- Stationary bicycle with no resistance once 90 degrees knee flexion obtained (~ 4 weeks).
- 90 degree leg dangle hourly to improve ROM

#### **THERAPY**

- Gentle multi-directional patella mobilization starts immediately after surgery.
- Cryotherapy and compression stockings/TEDS for swelling and pain control.
- E-stim for VMO/quadriceps muscle re-education/biofeedback encouraged early after surgery if needed.
- Gentle massage/deep friction to hamstring insertions, suprapatellar quadriceps, medial/lateral gutters, and infrapatellar fat pad region at 2-3 weeks post-op.
- Pool therapy recommended 2-3 weeks post-op to enhance motion.

CARTISTEM® 

# Femoral Condyle Defect

#### **PRIMARY GOALS**

# DO NOT OVERLOAD GRAFT INCREASE TIBIOFEMORAL AND PATELLOFEMORAL MOBILITY RESTORE QUADRICEPS CONTROL

| DD | A | | $\mathbf{F}$ |
|----|---|----|--------------|
| BR | A | v. | r |

• Knee brace may be discontinued once independent SLR achieved

#### **GAIT**

• Week 7 & 8: 50% weight-bearing, week 9+: full weight-bearing

#### **ROM**

- Full AROM and gentle PROM exercises
- Progress towards full ROM until the 12 week time point.

#### **THEREX**

- Low weight (max 10-20lbs.) open-chain leg extension and curl
- Stationary bicycle with gradual increased tension per level of comfort
- Continue quad sets, SLR in brace, leg curl and heel slides
- Strengthen quadriceps, hamstrings, and hip abductors/extensors using ankle weights and/or elastic band resistance through full ROM as tolerated
- Gentle closed-chain terminal knee extension 0 to 40 degrees (TKE) permitted starting from the nine or ten week time point as tolerated per weight bearing restriction

#### **THERAPY**

- Gentle multi-directional patella mobilization
- Cryotherapy and compression stockings/TEDS for swelling and pain control
- E-stim for VMO/quadriceps muscle re-education/biofeedback encouraged
- Gentle massage/deep friction to hamstring insertions, suprapatellar quadriceps, medial/lateral gutters, and infrapatellar fat pad region
- Pool therapy recommended to enhance motion

CARTISTEM® 

#### -- or for trochlear defects --

Stage 1- Proliferative Phase (Week 0 to 6)

# **Trochlear Defect**

#### PRIMARY GOALS

DO NOT OVERLOAD GRAFT INCREASE TIBIOFEMORAL AND PATELLOFEMORAL MOBILITY RESTORE QUADRICEPS CONTROL

#### **BRACE**

- Bledsoe Hinge knee brace for ambulation (locked) and at night
- Out of brace for CPM.
- No brace, but towel/pillow behind heel when lying down

#### **PRECAUTIONS**

Full weightbearing in full extension (locked brace)

#### **ROM**

- Gentle AROM flexion as tolerated 3x/day. Only PROM extension allowed.
- CPM  $\geq$  6 to 8 hours daily. Starting from 0 to 40 degrees, progress range as tolerated after the first 2 weeks.
- Minimum 90 degrees flexion for the first 2 weeks, 110 degrees for the next 4 weeks

#### **THEREX**

- Quad sets, SLR with brace locked, leg curl/heel slides, hip abduction
- Stationary bicycle with no resistance once 90 degrees knee flexion obtained (> 4wks).
- 90 Degree Leg dangle hourly to improve ROM

#### **THERAPY**

- Gentle multi-directional patella mobilization right after surgery
- Cryotherapy and compression stockings/TEDS for swelling and pain control.
- E-stim for VMO/quadriceps muscle re-education/biofeedback encourage early after surgery if necessary.
- Gentle massage/deep friction to hamstring insertions, suprapatellar quadriceps, medial/lateral gutters, and infrapatellar fat pad region at the two to three week time point post-op.
- Pool therapy recommended two to three weeks post-op to enhance motion.

CARTISTEM® 

# **Trochlear Defect**

# **PRIMARY GOALS**

# DO NOT OVERLOAD GRAFT INCREASE TIBIOFEMORAL AND PATELLOFEMORAL MOBILITY RESTORE QUADRICEPS CONTROL

**BRACE** 

• Hinged knee brace may be discontinued once independent SLR achieved

**GAIT** 

Full weight-bearing as tolerated

**ROM** 

- Gentle A/AAROM flexion and extension permitted
- Progress towards full ROM until week 12.

**THEREX** 

- Stationary bicycling without resistance at short intervals (5 min, 2-3x/day) as tolerated
- Strengthening of quadriceps, hamstrings, and hip abductors/extensors using elastic band isometrics and closed-chain terminal knee extension 0-40 degrees only
- Backward treadmill walking with safety bars recommended to reduce patellofemoral compressive forces
- Pool exercise using kickboard allowed. Flutter/straight leg scissor kick only (no whip kick)
- No open-chain strengthening permitted until 6 months after surgery.
- No closed-chain leg pressing or squatting

**THERAPY** 

- Gentle multi-directional patella mobilization
- Cryotherapy and compression stockings/TEDS for swelling and pain control
- E-stim for VMO/quadriceps muscle re-education/biofeedback encouraged
- Gentle massage/deep friction to hamstring insertions, suprapatellar quadriceps, medial/lateral gutters, and infrapatellar fat pad region
- Pool therapy recommended to enhance motion

CARTISTEM® 

# 12 References

Athanasiou KA, Shah AR, Hernandez RJ, LeBaron RG. Basic science of articular cartilage repair. Clin Sports Med. 2001 Apr;20(2):223-47.

Barry FP. Mesenchymal stem cell therapy in joint disease. Novartis Found Symp. 2003;249:86-96; discussion 96-102, 170-4, 239-41.

Browne JE, Anderson AF, Arciero R, Mandelbaum B, Moseley JB Jr, Micheli LJ, Fu F, Erggelet C. Clinical outcome of autologous chondrocyte implantation at 5 years in US subjects. Clin Orthop Relat Res. 2005 Jul;(436):237-45.

Caplan AI, Dennis JE. Mesenchymal stem cells as trophic mediators. J Cell Biochem. 2006 Aug 1;98(5):1076-84.

Chang CH, Kuo TF, Lin CC, Chou CH, Chen KH, Lin FH, Liu HC. Tissue engineering-based cartilage repair with allogenous chondrocytes and gelatin-chondroitin-hyaluronan tricopolymer scaffold: A porcine model assessed at 18, 24, and 36 weeks. Biomaterials. 2006 Mar;27(9):1876-88. Epub 2005 Nov 8.

Chuma H, Mizuta H, Kudo S, Takagi K, Hiraki Y. One day exposure to FGF-2 was sufficient for the regenerative repair of full-thickness defects of articular cartilage in rabbits. Osteoarthritis Cartilage. 2004 Oct;12(10):834-42.

Dragoo JL, Samimi B, Zhu M, Hame SL, Thomas BJ, Lieberman JR, Hedrick MH, Benhaim P. Tissue-engineered cartilage and bone using stem cells from human infrapatellar fat pads. J Bone Joint Surg Br. 2003 Jul;85(5):740-7.

Elisseeff J. Injectable cartilage tissue engineering. Expert Opin Biol Ther. 2004 Dec;4(12):1849-59.

Gelse K, Söder S, Eger W, Diemtar T, Aigner T. Osteophyte development--molecular characterization of differentiation stages. Osteoarthritis Cartilage. 2003 Feb;11(2):141-8.

Giannoni P, Pagano A, Maggi E, Arbicò R, Randazzo N, Grandizio M, Cancedda R, Dozin B. Autologous chondrocyte implantation (ACI) for aged patients: development of the proper cell expansion conditions for possible therapeutic applications. Osteoarthritis Cartilage. 2005 Jul;13(7):589-600.

Guo X, Wang C, Zhang Y, Xia R, Hu M, Duan C, Zhao Q, Dong L, Lu J, Qing Song Y. Repair of large articular cartilage defects with implants of autologous mesenchymal stem cells seeded into beta-tricalcium phosphate in a sheep model. Tissue Eng. 2004 Nov-Dec;10(11-12):1818-29.

Hedrick MH, Daniels EJ. The use of adult stem cells in regenerative medicine. Clin Plast Surg. 2003 Oct;30(4):499-505.

Kasahara Y, Iwasaki N, Yamane S, Igarashi T, Majima T, Nonaka S, Harada K, Nishimura S, Minami A. Development of mature cartilage constructs using novel three-dimensional porous

CARTISTEM® 

scaffolds for enhanced repair of osteochondral defects. J Biomed Mater Res A. 2008 Jul;86(1):127-36.

Katayama R, Wakitani S, Tsumaki N, Morita Y, Matsushita I, Gejo R, Kimura T. Repair of articular cartilage defects in rabbits using CDMP1 gene-transfected autologous mesenchymal cells derived from bone marrow. Rheumatology (Oxford). 2004 Aug;43(8):980-5. Epub 2004 Jun 8.

Lee YS, Heo EA, Jun HY, Kang SH, Kim HS, Lee MS, Byun SJ, Lee SH, Park SH, Yoon KH. Articular cartilage imaging by the use of phase-contrast tomography in a collagen-induced arthritis mouse model. Acad Radiol. 2010 Feb;17(2):244-50. Epub 2009 Dec 4.

Marcacci M, Berruto M, Brocchetta D, Delcogliano A, Ghinelli D, Gobbi A, Kon E, Pederzini L, Rosa D, Sacchetti GL, Stefani G, Zanasi S. Articular cartilage engineering with Hyalograft C: 3-year clinical results. Clin Orthop Relat Res. 2005 Jun;(435):96-105.

Mizuta H, Kudo S, Nakamura E, Otsuka Y, Takagi K, Hiraki Y. Active proliferation of mesenchymal cells prior to the chondrogenic repair response in rabbit full-thickness defects of articular cartilage. Osteoarthritis Cartilage. 2004 Jul;12(7):586-96.

Moore RA, Derry S, Makinson GT, McQuay HJ. Tolerability and adverse events in clinical trials of celecoxib in osteoarthritis and rheumatoid arthritis: systematic review and meta-analysis of information from company clinical trial reports. Arthritis Res Ther. 2005;7(3):R644-65. Epub 2005 Mar 24.

Otsuka Y, Mizuta H, Takagi K, Iyama K, Yoshitake Y, Nishikawa K, Suzuki F, Hiraki Y. Requirement of fibroblast growth factor signaling for regeneration of epiphyseal morphology in rabbit full-thickness defects of articular cartilage. Dev Growth Differ. 1997 Apr;39(2):143-56.

Risbud M, Ringe J, Bhonde R, Sittinger M. In vitro expression of cartilage-specific markers by chondrocytes on a biocompatible hydrogel: implications for engineering cartilage tissue. Cell Transplant. 2001;10(8):755-63.

Smith GD, Knutsen G, Richardson JB. A clinical review of cartialge repair techniques. J Bone Joint Surg[Br]. 2005;87-B:445-9

Wakitani S, Imoto K, Yamamoto T, Saito M, Murata N, Yoneda M. Human autologous culture expanded bone marrow mesenchymal cell transplantation for repair of cartilage defects in osteoarthritic knees. Osteoarthritis Cartilage. 2002 Mar;10(3):199-206.

Wakitani S, Okabe T, Horibe S, Mitsuoka T, Saito M, Koyama T, Nawata M, Tensho K, Kato H, Uematsu K, Kuroda R, Kurosaka M, Yoshiya S, Hattori K, Ohgushi H. Safety of autologous bone marrow-derived mesenchymal stem cell transplantation for cartilage repair in 41 patients with 45 joints followed for up to 11 years and 5 months. J Tissue Eng Regen Med. 2010 Jul 5 [Epub ahead of print]

Watterson JR, Esdaile JM. Viscosupplementation: Therapeutic mechnisms and clinical potential in osteoarthritis of the knee. J Am Acad Orthop Surg. 2000;8:277-284.

CARTISTEM® 

Yanai T, Ishii T, Chang F, Ochiai N. Repair of large full-thickness articular cartilage defects in the rabbit: the effects of joint distraction and autologous bone-marrow-derived mesenchymal cell transplantation. J Bone Joint Surg Br. 2005 May;87(5):721-9.

CARTISTEM® 

2000

**IKDC** 

**KNEE FORMS** 

CARTISTEM® 

# **IKDC PATIENT REPORTED**

#### **SYMPTOMS\*:**

\*Grade symptoms at the highest activity level at which you think you could function without significant symptoms, even if you are not actually performing activities at this level.

| 1. | Strenuc | renuous activitate activities l | activities l<br>ties like h<br>ties like m<br>like walkin | ike jumpi<br>eavy phys<br>oderate pl<br>ng, house | ng or pivo<br>sical work<br>hysical wo<br>work or ya | oting as ir<br>s, skiing o<br>ork, runni<br>ard work | n basketba<br>r tennis<br>ng or jogg | all or socce | - | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 2. ] | During the | past 4 we | eeks, or si | nce your i | njury, hov | w often ha | ave you h | ad pain? | | | | | |
| | Never | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Constant |
| | $\odot$ | | | | | | | | | | | | |
| 3. | If you have | e pain, h | ow severe | e is it? | | | | | | | | | |
| | Never | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Worst Pain<br>Imaginable |
| | During the Not a What is the Very st Strenuc Modera Light a | t all highest larenuous activitate activities l | level of ac<br>activities l<br>ties like h<br>ties like m<br>like walkin | Aildly tivity you ike jumpi eavy physoderate plang, housev | can performs can perform can perform can be | Moder<br>orm withouting as ir<br>s, skiing o<br>ork, runni | rately<br>out signific<br>n basketba<br>r tennis<br>ng or jogg | cant swell ill or socco | Very | ır knee? | Е | extremely | 7 |
| 6. ] | During the | past 4 we | eeks, or si | nce your i | njury, did | l your kne | e lock or | catch? | | | | | |
| 7. | What is the Very st Strenuc Modera Light a | renuous activitate activities l | activities l<br>ties like h<br>ties like m<br>like walkin | ike jumpi<br>eavy phys<br>oderate pl<br>ng, housev | ng or pivo<br>sical work<br>hysical wo<br>work or ya | oting as ir<br>, skiing o<br>ork, runni<br>ard work | n basketba<br>r tennis<br>ng or jogg | all or socco | er | your knee? | | | |

CARTISTEM® 

# IKDC Subjective Knee Evaluation Form cont.

#### SPORTS ACTIVITIES:

| | □V€ □Str □M€ □Lig | is the highest level of acery strenuous activities like headerate activities like might activities like walking hable to perform any of | ike jump<br>eavy phy<br>oderate j<br>ng, house<br>the abov | oing or<br>vsical<br>physic<br>ework<br>e activ | r pivoti<br>work, s<br>al work | ng as<br>skiing<br>k, run<br>d wor | in bas<br>or ten<br>ning o | ketball<br>nis | or so | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 9. | How d | loes your knee affect yo | ur ability | / to: | | N | ot diff<br>at a | | | nimal<br>fficult | | | erately<br>icult | | Extremely difficult | | nable<br>o do |
| | a. | Go up stairs | | | | | | | | | | | | | | | |
| | b. | Go down stairs | | | | | | | | | | | | | | | |
| | c. | Kneel on the front of | your kne | e | | | | | | | | | | | | | |
| | d. | Squat | | | | | | | | | | | | | | | |
| | e. | Sit with your knee be | nt | | | | | | | | | | | | | | |
| | f. | Rise from a chair | | | | | | | | | | | | | | | |
| | g. | Run straight ahead | | | | | | | | | | | | | | | |
| | h. | Jump and land on you | r involv | ed leg | | | | | | | | | | | | | |
| | i. | Stop and start quickly | | | | | | | | | | | | | | | |
| | | ION: would you rate the fundability to perform any o | - | | | | | | | | - | mal, ex | cellent | func | tion and 0 | being | |
| FU | J <b>NCT</b> | ION PRIOR TO YOU | R KNEI | E INJ | URY: | | | | | | | | | | | | |
| | | Cannot perform daily activities | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | No | limitatio | n |
| CI | J <b>RRE</b> | NT FUNCTION OF Y | OUR K | NEE: | | | | | | | | | | | | | |
| | | Cannot perform daily activities | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | N | No limita | tion |

CARTISTEM® 

# APPENDIX 2. LYSHOLM SCORE

# LYSHOLM KNEE SCORING SCALE

Instructions: Below are common complaints which people frequently have with their knee problems. Please check the statement which best describes your condition.

| I.<br> | LIMP: I have no limp when I walk. (5) I have a slight or periodical limp when I walk. (3) I have a severe and constant limp when I walk. (0) | v | PAIN: I have no pain in my knee. (25) I have intermittent or slight pain in my knee during vigorous activities. (20) |
|---|---|---|---|
| п. | USING CANE OR CRUTCHES I do not use a cane or crutches. (5) | _ | I have marked pain in my knee during vigorous activities. (15) I have marked pain in my knee during or after walking more than 1 mile. (10) |
| _ | I use a cane or crutches with some weight-bearing. (2) Putting weight on my hurt leg is impossible. (0) | _ | I have marked pain in my knee during or after<br>walking less than 1 mile. (5)<br>I have constant pain in my knee. (0) |
| III | LOCKING SENSATION IN THE KNEE I have no locking and no catching sensations in my knee. (15) I have catching sensation but no locking sensation in my knee. (10) My knee locks occasionally. (6) My knee locks frequently. (2) My knee feels locked at this moment. (0) GIVING WAY SENSATION FROM THE KNEE My knee never gives way. (25) My knee rarely gives way, only during athletics or other vigorous activities. (20) My knee frequently gives way during athletics or other vigorous activities, in turn I am unable to participate in these activities. (15) My knee occasionally gives way during daily activities. (10) My knee often gives way during daily activities. (5) My knee gives way every step I take. (0) | VI | SWELLING I have no swelling in my knee. (10) I have swelling in my knee only after vigorous activities. (6) I have swelling in my knee after ordinary activities. (2) I have swelling constantly in my knee. (0) CLIMBING STAIRS: I have no problems climbing stairs. (10) I have slight problems climbing stairs. (6) I can climb stairs only one at a time. (2) Climbing stairs is impossible for me. (0) SQUATTING I have no problems squatting. (5) I have slight problems squatting. (4) I can not squat beyond a 90 degree bend in my knee. (2) Squatting is impossible because of my knee. (0) |
| | ī | TOTAL | /100 |
| | RUCTIONS: Please place an X on the line to indicate the a anges from "no pain at all" to the "worst possible pain". | amount of | F pain you have had in your knee(s) the past 24 hours. Th |
| RIGHT | Γ KNEEno pain | | worst possible pain |
| LEFT | KNEE | | worst possible pain |

CARTISTEM® 

Knee injury and Osteoarthritis Outcome Score (KOOS), English version LK1.0

| Pain P1. How often do you Never | ou experience k<br>Monthly | nee pain?<br>Weekly | Daily | Always | |
|---|---|---|---|---|---|
| What amount of I following activities | | ve you experie | enced the last | week during the | |
| P2. Twisting/pivotin | g on your knee<br>Mild | Moderate | Severe | Extreme | |
| P3. Straightening kn | ee fully<br>Mild | Moderate | Severe | Extreme | |
| P4. Bending knee fu<br>None | lly<br>Mild<br>□ | Moderate | Severe | Extreme | |
| P5. Walking on flat None | surface<br>Mild | Moderate | Severe | Extreme | |
| P6. Going up or dow | vn stairs<br>Mild | Moderate | Severe | Extreme | |
| P7. At night while in None | n bed<br>Mild | Moderate | Severe | Extreme | |
| P8. Sitting or lying None | Mild | Moderate | Severe | Extreme | |
| P9. Standing upright None | Mild | Moderate | Severe | Extreme | |
| Function, daily live The following quest ability to move an activities please in last week due to y | stions concerr<br>ound and to<br>ndicate the de | look after you | irself. For each | of the following | ١ |
| A1. Descending stain None | rs<br>Mild | Moderate | Severe | Extreme | |
| A2. Ascending stairs | Mild | Moderate | Severe | Extreme | |

CARTISTEM® 

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your knee.

| A3. Rising from s None | sitting<br>Mild | Moderate | Severe | Extreme |
|---|---|---|---|---|
| A4. Standing None | Mild | Moderate | Severe | Extreme |
| A5. Bending to fl<br>None | oor/pick up an o<br>Mild | object<br>Moderate | Severe | Extreme |
| A6. Walking on f | lat surface<br>Mild | Moderate | Severe | Extreme |
| A7. Getting in/ou<br>None | t of car<br>Mild | Moderate | Severe | Extreme |
| A8. Going shoppi<br>None | ing<br>Mild | Moderate | Severe | Extreme |
| A9. Putting on so None | cks/stockings<br>Mild | Moderate | Severe | Extreme |
| A10. Rising from None | bed Mild | Moderate | Severe | Extreme |
| A11. Taking off s None | socks/stockings<br>Mild | Moderate | Severe | Extreme |
| A12. Lying in bed | d (turning over, Mild | maintaining knee p<br>Moderate<br>□ | oosition)<br>Severe | Extreme |
| A13. Getting in/o | ut of bath<br>Mild | Moderate | Severe | Extreme |
| A14. Sitting None | Mild | Moderate | Severe | Extreme |
| A15. Getting on/o | off toilet<br>Mild | Moderate | Severe | Extreme |

CARTISTEM® 

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your knee.

A16. Heavy domestic duties (moving heavy boxes, scrubbing floors, etc)

None Mild Moderate Severe Extreme

A17. Light domestic duties (cooking, dusting, etc) None Mild Moderate Severe Extreme 

#### Function, sports and recreational activities

The following questions concern your physical function when being active on a higher level. The questions should be answered thinking of what degree of difficulty you have experienced during the **last week** due to your knee.

| SP1. Squatting None | Mild | Moderate | Severe | Extreme |
|---|---|---|---|---|
| SP2. Running None | Mild | Moderate | Severe | Extreme |
| SP3. Jumping None | Mild | Moderate | Severe | Extreme |
| SP4. Twisting/piv | oting on your i<br>Mild | njured knee<br>Moderate | Severe | Extreme |
| SP5. Kneeling None | Mild | Moderate | Severe | Extreme |
| Quality of Life | | | | |
| Q1. How often are Never | e you aware of Monthly | your knee problem'<br>Weekly | ?<br>Daily<br><b>D</b> | Constantly |
| Q2. Have you mo | dified your life | style to avoid poter | ntially damagins | g activities |
| to your knee? Not at all | | Moderately | Severely | Totally |
| Q3. How much ar<br>Not at all | e you troubled<br>Mildly | with lack of confidence Moderately | ence in your kne<br>Severely | Extremely |
| Q4. In general, ho | w much diffict<br>Mild | ulty do you have wind Moderate | th your knee? Severe | Extreme |

Thank you very much for completing all the questions in this questionnaire.

CARTISTEM® 

# Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES
National Institutes of Health
National Cancer Institute

CARTISTEM® 

# Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

Publish Date: May 28, 2009

#### Quick Reference

The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term

#### Components and Organization

#### SOF

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### CTCAE Terms

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may <u>not</u> be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

#### Definitions

A brief definition is provided to clarify the meaning of each AE term.

#### Grades

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL\*\*.

Grade 4 Life-threatening consequences; urgent intervention indicated.

Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

#### Grade 5

Grade 5 (Death) is not appropriate for some AEs and therefore is not an option.

#### Activities of Dally Living (ADL)

"Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

""Self care ADL refer to bathing dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

CARTISTEM® 

<sup>1</sup> CTCAE v4.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.com).

| | В | lood and lymphatic syst | em disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | -2 | 3 | 4 | 5 |
| Anemia | Hemoglobin (Hgb) < LLN - 10.0<br>g/dL; < LLN - 6.2 mmol/L; < LLN -<br>100 g/L | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9<br>mmol/L; <100 - 80g/L | Hgb <8.0 - 6.5 g/dL; <4.9 - 4.0<br>mmol /L; <80 - 65 g/L;<br>transfusion indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| 1 15 15 UE SE U | zed by an reduction in the amount on, palpitations of the heart, soft syst | NE 74 2000 (COEPE | S-1054 | ay indude pallor of the skin and m | nucous |
| Bone marrow hypocellular | Mildly hypocellular or <= 25 % reduction from normal cellularity for age | Moderately hypocellular or >25 -<br><50 % reduction from normal<br>cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer<br>than 2 weeks | Death |
| Definition: A disorder characteri | zed by the inability of the bone man | row to produce hematopoletic ele | ments. | | |
| Disseminated intravascular<br>coagulation | 1 | Laboratory findings with no<br>bleeding | Laboratory findings and bleeding | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by systemic pathological activa | tion of blood clotting mechanisms | which results in dot formation thr | oughout the body. There is an incr | rease in the |
| risk of hemorrhage as the body | is depleted of platelets and coagula | ation factors. | | 03 80 | |
| Febrile neutropenia | | | Present | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a decrease in neutrophils as | sociated with fever. | 5 | | 28 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and >=2<br>gm decrease in hemoglobin , no<br>transfusion | Transfusion or medical<br>intervention indicated (e.g.,<br>steroids) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by laboratory test results that in | Idioate widespread erythrocyte œ | II membrane destruction. | , | 9 |
| Hemolytic uremic syndrome | Evidence of RBC destruction<br>(schistocytosis) without dinical<br>consequences | | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder characteri | zed by a form of thrombotic microar | giopathy with renal failure, hemo | lytic anemia, and severe thromboo | cytopenia. | 00<br>20 |
| Leukocytosis | ( <b>*</b> 27 | • | >100 ,000 /mm3 | Clinical manifestations of<br>leucostasis; urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | ,<br>zed by laboratory test results that in | Idicate an increased number of w | nite blood cells in the blood. | | 4 |
| Lymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 3 | 5 |
| Definition: A disorder characteri | zed by a sensation of marked disco | mfort in a lymph node. | 7 | Tananan anna | Towns and |
| Spleen disorder | Incidental findings (e.g., Howell-<br>Jolly bodies); mild degree of<br>thrombocytosis and<br>leukocytosis | Prophylactic antibiotics indicated | | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder of the sple | en. | ¥0 | 30<br>20 | 7 | 00 I |
| Thrombotic thrombocytopenic<br>purpura | Evidence of RBC destruction<br>(schistocytosis) without dinical<br>consequences | - | Laboratory indings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-thre atening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | zed by the presence of microangiop<br>sual disturbances. It is an acute or s | | cytopenic purpura, fever, renal abr | normalities and neurological abnor | malities such |
| Blood and lymphatic system<br>disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization in dicated;<br>disabling; limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : 8 bod and tym phatb system disorde  $\sigma$ 

CARTISTEM® 

| | | Cardiac disorde | rs | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1: | -2 | 3 | 4 | 5 |
| Acute coronary syndrome | 28 | Sympto matic, progressive<br>angina; cardiac enz ymes<br>normal; hemodynamically stable | Symptomatic, unstable angina and/or acute myocardial infarction, cardiac enzymes abnormal, hemodynamically stable | Symptomatic, unstable angina<br>and/or acute myo cardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>unstable | Death |
| | ed by signs and symptoms related<br>unstable angina to myocardial infa | | lium secondary to coronary artery | disease. The clinical presentation | co vers a |
| Aortic valve disease | Asymptomatic valvular | Asymptomatic; moderate | Symptomatic; severe | Life-threatening consequences; | Death |
| volue disease | thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | regurgitation or stenosis by imaging | regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteria | red by a defect in a ortic valve funct | ion or structure. | 7 | | |
| Asystole | Periods of asystole; non-urgent medical management indicated | | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | ed by a dysrhythmia without cardi:<br>T | ac electrical activity. Typically, this<br>T | is accompanied by cessation of th | ne pumping function of the heart. | riy<br>Formovony |
| Atrial fibrillation | Asymptomatic, intervention not<br>indicated | Non-urgent medical intervention<br>indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ed by a dysrhythmia without disce | rnible P waves and an irregular ve | entricular response due to multiple | reentry circuits. The rhythm distur | bance |
| originates above the ventrides. | 10 00 A | Te- | 100 (c) | 00 00 | |
| Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria<br>atria. | ,<br>red by a dysrhythmia with organize | ,<br>d rhythmic atrial contractions with | a rate of 200-300 beats per minut | ,<br>e . The rhythm disturbance origina: | tes in the |
| Atrioventricular block complete | 50 | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | ed by a dysrhythmia with complete | e failure of atrial electrical impulse | conduction through the AV node t | othe ventrides. | 8 |
| Atrioventricular block first<br>degree | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | - | | - |
| | ed by a dysrhythmia with a delay i<br>interval greater than 200 milliseco | 기가 있는 것이 없는 것이 없는 아무리 가장 없는 것이 없는 것이 없다고 있다. | tion of an electrical impulse throug | the atrioventricular (AV) node bo | eyond D.2 |
| Cardia c arrest | Intervargreater than 200 miniseco | 0 | | FIZ. de como cita de como como como como como como como com | Death |
| | red by cessation of the pumping fu | notion of the heart | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting instrumental ADL | Pain at rest; limiting self care<br>ADL | 8 | 5 |
| Definition: A disorder characteria | ed by substemal discomfort due to | insufficient myocardial oxygenati | on. | | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disord er characteriz | ed by pathological irregularities in | the cardiac conduction system. | | | |
| Constrictive pericarditis | | | Symptomatic heart failure or<br>other cardiac symptoms,<br>responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| Definition: A disorder characteriz | ed by a thickened and fibrotic peri | cardial sac; these fibrotic changes | impe de normal myocardial functio | on by restricting myocardial musde | e action. |
| Heart failure | Asymptomatic with laboratory<br>(e.g., BNP (B- Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or<br>with minimal activity or exertion;<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic<br>support) | Death |
| Definition: A disorder characteriz<br>in the filling pressure. | ed by the inability of the heart to p | ump blood at an adequate volume | to me et tissue metabolic requiren | nents, or, the ability to do so only a | at an elevatio |

CTCAE 4.0 - May 28, 2009 : Cardiac disorders

CARTISTEM® 

| 9:<br>S | | Cardiac disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1: | -2 | 3 | 4 | 5 |
| Le t ventricular systolic<br>dysfunction | \$ | | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | zed by failure of the left ventride to<br>nea, orthopnea, and other signs ar | \$10 ACC \$10 ACC \$10 | e an increase in distending pressur<br>estion and edema. | e and in end-diastolic volume. Clin | ical |
| Mitral valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe<br>regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteri | zed by a defect in mitral valve func | tion or structure. | The second secon | Tourist | |
| Mobitz (type) II atrioventricular<br>block | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely<br>controlled medically, or<br>controlled with device (e.g.,<br>pacemaker) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | zed by a dysrhythmia with relativel<br>atrioventricular (AV) node to the ve | [전문] [1] [1] [1] [2] [2 | block of an atrial impulse. This is t | he result of intermittent failure of a | trial electrical |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | zed by a dysrhythmia with a progre<br>on through the atrioventricular (AV | 그는 이 시민은 사람들은 내가 많아서 있다면 있다. | rior to the blocking of an atrial impu | ,<br>Ilse. This is the result of intermitter | nt failure of |
| Myocardial infarction | i esi | Asymptomatic and cardiac<br>enzyme's minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences;<br>hemodynamically un stable | Death |
| Definition: A disorder characteri | zed by gross ne crosis of the myoca | ardium; this is due to an interrupti | on of blood supply to the area. | | |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic<br>support) | Death |
| Definition: A disorder characteri | zed by inflammation of the muscle | tissue of the heart. | - | | |
| Palpitations | Mild symptoms; intervention not indicated | Intervention indicated | ** | 8 | |
| Definition: A disorder characteri | zed by an unpleasant sensation of | irregular and/or force ful be ating o | fthe heart. | | |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical management indicated | M medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically, cardioversion<br>indicated | Death |
| Definition: A disorder characteri<br>originates in the atria. | zed by a dysrhythmia with abrupt o | nset and sudden termination of a | trial contractions with a rate of 150- | 250 beats per minute. The rhythm | n disturbance |
| Pericardial effusion | - | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by fluid collection within the pe | ricardial salo, usually due to inflan | nmation. | Incore es | - S |
| Pericardial tamponade | 5 | - | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an increase in intrapericardi | ial pressure due to the collection | of blood or fluid in the pericardium. | | |
| Pericarditis | Asymptomatic, ECG or physical findings (e.g., rub) consistent with pericarditis | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic<br>consequences (e.g., pericardial<br>constriction) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | ed by imitation to the layers of the | pericardium (the protective sac a | round the heart). | | |

CTCAE 4.0 - May 28, 2009 : Candiac disords is

CARTISTEM® 

| 5 | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1: | -2 | 3 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder character | ized by a defect in pulmonary valve | function or structure. | | | |
| Restrictive cardiomyopathy | To the properties as the properties | Think organization sensets | Symptomatic heart failure or<br>other cardiac symptoms,<br>responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| Definition: A disorder character | ized by an inability of the ventricles | to fill with blood because the myo | ardium (heart musde) stiffens an | d loses its flexibility. | |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated<br>with hypoxemia, right heart<br>failure; oxygen indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., ventricular assist device);<br>heart transplant indicated | Death |
| 2012/1972 | ized by impairment of right ventricul: | (C.28) (C.2) (28) | 100 000 000 100 000 000 000 000 000 000 | 0100000 700 | 122 22 |
| Sick sinus syndrome | Asymptomatic, intervention not<br>indicated | Non-urgent intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ized by a dysrhythmia with alternation | | | | T. |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, medical<br>intervention indicated | Severe, medically significant,<br>medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia with a heart r | ate less than 60 beats per minute | that originates in the sinus node. | | T. |
| Sinus tachycardia | Asymptomatic, intervention not indicated | Symptomatic; non-urgent medical intervention indicated | Urgent medical intervention indicated | | |
| Definition: A disorder character | ized by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates in the sinus no | ode. | 991 |
| Supraventricular tachycardia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Me dical intervention in dicate d | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates above the ven | tricles. | |
| Tricuspid valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| | ized by a defect in tricuspid valve fu | | | | Stronger |
| Ventricular amhythmia | Asymptomatic, intervention not<br>indicated | Non-urgent medical intervention<br>indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia that originate | s in the ventricles. | 0.5 | | 001 |
| Ventricular fibrillation Definition: A disorder character | ized by a dysrhythmia without disce | rnible QRS complexes due to rapi | -<br>d repetitive excitation of myocardi | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated<br>ial fibers without coordinated contr | Death action of |
| ventricles. | | | | | |
| Ventri cular tach y cardia | 140 | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia with a heart n | ate greater than 100 be ats per mi | nute that originates distal to the bu | undle of His. | (V) |
| Wolff Parkinson-White<br>syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically or controlled with procedure | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder obacted | I<br>ized by the presence of an accessor | I<br>or conducting nathway between th | | J<br>ses niremature sentricular activation | L<br>D |
| PERSONAL PROPERTY AND PROPERTY. | 1 - 3 - | Marine Carrier | The purpose of the control of the purpose of the state of the control of the cont | a Christian Comment of the Comment o | Daniel Control |
| Cardiae disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or nonin vasive intervention indicated; limiting ageappropriate instrumental ADL | Severe or me dically significant<br>but not imme diately life-<br>thre attening; hospitalization or<br>prolongation of existing<br>hospitalization in dicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Cand lacid to ride is  $6\,$ 

CARTISTEM® 

| | Congenital, familial and genetic disorders | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Congenital, familial and<br>genetic disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations<br>only; intervention not<br>indicated | Moderate; minimal, local<br>or noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately life-<br>threatening, hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Congenital, familial and genetic disorders 7

CARTISTEM® 

| Ear and labyrinth disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Earpain<br>Definition: A disorder character | Mild pain | Moderate pain; limiting instrumental ADL moort in the ear. | Severe pain; limiting self care<br>ADL | | 25 |
| External ear inflammation | External otitis with erytherna or dry desquarmation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis;<br>stenosis or osteomyelitis;<br>necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by inflammation , swelling and n | edness to the outer ear and ear o | anal. | | |
| External ear pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain ; limiting self care<br>ADL | ā | - |
| Definition: A disord er character | ized by a sensation of marked disco | mfort in the external ear region. | 7. O | | - |
| Hearing impaired | Adults enrolled on a monitoring program (a 1, 2, 3, 4, 6 and 8 kHz audiogram): threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear or subjective change in the absence of a Grade 1 threshold shift Pediatrics (a 1, 2, 3, 4, 6 and 8 kHz audiogram): >20 dB at any frequency tested and does not meet criteria for > Grade 2 | Adults enrolled in monitoring program (a 1, 2, 3, 4, 6 and 8 kHz audiogram): threshold shift of >25 d B a veraged at 2 contiguous test frequencies in at least one ear Adult not enrolled in monitoring program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL Pediatrics (a 1, 2, 3, 4, 6 and 8 kHz audiogram): >20 dB at >4 kHz | Adults enrolled in monitoring program (a 1, 2, 3, 4, 6 and 8 kHz audiogram): threshold shift of >25 d B averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated Adults not enrolled in monitoring program: hearing loss with hearing aid or intervention indicated; limiting self care ADL Pediatrics (a 1, 2, 3, 4, 6 and 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing aids; >20 d B at 3 kHz and above in one ear; additional speech-language related services indicated | Adults: profound bilateral hearing loss (>80 dB at 2 kHz and above); non-serviceable hearing Pediatric: audiologic indication for cochlear implant and additional speech-language related services indicated | - |
| Definition: A disorder character | ized by partial or complete loss of th | e ability to detect or understand s | ounds resulting from damage to e | ar structures. | 2 |
| Middle ear in fammation | Serous otitis | Serous otitis, medical intervention indicated | Mastoiditis; necrosis of canal softissue or bone | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character<br>Tinnitus | ized by inflammation (physiologic re:<br>Mild symptoms; intervention not<br>indicated | No. | Severe symptoms; limiting self care ADL | | |
| Definition: A disorder character | ized by noise in the ears, such as rir | nging, buzzing, roaring or clicking. | | | T. |
| √entigo | Mild symptoms | Moderate symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | ٥ | - |
| Definition: A disord er character<br>vertigo). | ized by a sensation as if the externa | I world were revolving around the | patient (objective vertigo) or as if | he himselfwere revolving in spac | e (subjed |
| Æ stibular disorder | 120 | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | 3 | - |
| Definition: A disorder character | ized by dizziness, imbalance, nause | a, and vision problems. | | | ę. |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or me dically significant<br>but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting selfcare ADL | Life-threatening consequences; urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Ear and labyrin to disorders

CARTISTEM® 

| Endocrine disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Adrenal insufficiency | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rs when the adrenal cortex does not<br>ison's disease or primary adrenal in: | V. C. 120. | cortisol and in some cases, the ho | ormone aldosterone. It may be due | to a disor |
| Cushingoid | Mild symptoms; intervention not indicated | [2: | Severe symptoms, medical intervention or hospitalization indicated | ē | - |
| Definition: A disorder character<br>osteoporosis, usually due to ex | ized by signs and symptoms that re<br>togenous corticosteroids. | semble Cushing's disease or syno | drome: buffalo hump obesity, stria | tions , adip osity , hypertension , diab | etes, and |
| Delayed puberty | | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age<br>14 yrs for females; no increase<br>in testes volume or no Tanner<br>Stage 2 by age 16 yrs for<br>males; hormone replacement<br>indicated | | 12 |
| Definition: A disorder character | ized by unusually late sexual maturi | ty. | | | |
| Growth accelerated | -1 | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | | | |
| Definition: A disorder character | ized by greater growth than expecte | d forage. | | | |
| Hyperparath yroidism | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | | 8 | - |
| Definition: A disorder character<br>the blood). | ized by an increase in production of | r<br>parath yroid hormone by the para | thyroid glands. This results in hyp | ercaloemia (abnormally high levels | of calcium |
| Hyperthyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid<br>suppression therapy indicated;<br>limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by excessive levels of thyroid h | normone in the body. Common ca | uses include an overactive thyroid | gland orthyroid hormone overdos | e. |
| Hypoparathyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; medical<br>intervention or hospitalization<br>indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder character | ized by a decrease in production of | parathyroid hormone by the parat | hyroid glands. | 1 | |
| Hypothyroidism | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; thyroid replacement indicated; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; hospitalization<br>indicated | Life-threatening consequences;<br>urgent intervention indicated; | Death |
| Definition: A disorder character | ized by a decrease in production of | thyroid hormone by the thyroid gla | and. | | |
| Pre∞cious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical<br>markers of puberty for females<br><8 years and males <9 years | - | | |
| Definition: A disorder character<br>9 for boys. | ized by unusually early developmen | t of secondary sexual features; th | e onset of sexual maturation begi | ns usually before age 8 for girls an | d before a |
| Mrilization . | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | 100 | 9 | 2 |
| Definition: A disorder character | ized by inappropriate masculinizatio | n occurring in a female or prepub | erta I male . | 3 | 50 |
| Endocrine disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization in dicated;<br>disabling; limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Endocribe disorde s

CARTISTEM® 

| | Eye disorders | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | -2 | 3 | 4 | - 5 |
| Blumed vision | Intervention not indicated | Symptomatic; limiting instrumental ADL | Limiting self care ADL | | - |
| Definition: A disorder charact | terized by visual perception of unclear | or fuzz y images. | Ť a | · | ř |
| Cataract | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; moderate<br>decrease in visual acuity (20/40<br>or better) | Symptomatic with marked decrease in visual acuity (worse than 20/40 but better than 20/200); operative intervention indicated (e.g., cataract surgery) | Blindness (20/200 or worse) in<br>the affected eye | 5 |
| Definition: A disorder charact<br>untreated. | terized by partial or complete opacity o | of the crystalline lens of one or bot | h e yes. This results in a decrease | in visual acuity and eventual blind | ness if |
| Conjunctivitis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; topical intervention indicated (e.g., antibiotics); limiting in strumental ADL | Limiting self care ADL | | 5 |
| Definition: A disorder charact | terized by inflammation, swelling and r | redness to the conjunctiva of the e | ye. | | 0 |
| Come al ulœr | 130 | Symptomatic; medical<br>intervention indicated (e.g.,<br>topical agents); limiting<br>instrumental ADL | Umiting self care ADL; declining<br>vision (worse than 20/40 but<br>better than 20/200) | Perforation or blindness (20/200<br>or worse) in the affected eye | 5 |
| Definition: A disorder charact | terized by an area of epithelial tissue l | oss on the surface of the comea. | t is associated with in tammatory o | ells in the comea and anterior cha | mber. |
| Dryeye | Asymptomatic; clinical or<br>diagnostic observations only;<br>mild symptoms relieved by<br>lubricants | Symptomatio; multiple agents indicated; limiting instrumental ADL | Decrease in visual acuity<br>(<20 A0); limiting self care ADL | | |
| Definition: A disorder charact | terized by dryness of the comea and c | onjunctiva. | | | |
| Extraocular musde paresis | Asymptomatic; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL; disabling | ē | - |
| Definition: A disorder charact | terized by incomplete paralysis of an e | otraocular musdle. | Z | | |
| Eye pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | - |
| Definition: A disorder charact | terized by a sensation of marked disco | omfort in the eye. | ¥ | | 0 |
| Eyelid function disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; non operative<br>intervention indicated; limiting<br>instrumental ADL | Limiting self care ADL;<br>operative intervention indicated | 20 | • |
| Definition: A disorder charact | terized by impaired eyelid function. | É | To a second | | r |
| Flashing lights | Symptomatic but not limiting<br>ADL | Limiting instrumental ADL | Limiting self care ADL | 2 | 5 |
| Definition: A disorder charact | terized by a sudden or briefburst oflig | ht. | Torono or was | | ř |
| Floaters | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | | ē<br>2 |
| | terized by an individual seeing spots b | 6: | | | |
| Glaucoma | Bevated intraocular pressure<br>(EIOP) with single topical agent<br>for intervention; no visual field<br>deficit | EIOP causing early visual field<br>deficits; multiple topical or oral<br>agents indicated; limiting<br>instrumental ADL | EIOP causing marked visual<br>feld defoits (e.g., involving both<br>superior and inferior visual<br>felds); operative intervention<br>indicated; limiting self care ADL | Blindness (20/200 or worse) in<br>the affected eye | - |
| Definition: A disorder charact | terized by an increase in pressure in th | ne eyeball due to obstruction of the | aqueous humo routflow. | | |
| Keratitis | 30 | Symptomatic; medical<br>intervention indicated (e.g.,<br>topical agents); limiting<br>instrumental ADL | Dedine in vision (worse than<br>20/40 but better than 20/200);<br>limiting self care ADL | Perforation or blindness (20/200<br>orworse) in the affected eye | - |
| Definition: A disorder charact | erized by inflammation to the comea | of the eye. | T | | |

CTCAE 4.0 - May 28, 2009 : Eye disorde  $\ensuremath{\mathbf{g}}$ 

CARTISTEM® 

| | | Eye disorders | S | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only | Limiting vision of the affected eye (20/40 or better); | Limiting vision in the affected<br>eye (worse than 20/40 but<br>better than 20/200) | Blindness (20/200 or worse) in<br>the affected eye | - |
| Definition: A disorder characteri | zed by involvement of the optic ner | ve (second cranial nerve). | 6 | | 1 |
| Papilledema | Asymptomatic; no visual field defects zed by swelling around the optic dis | Symptomatic decline in vision;<br>visual field defect present<br>sparing the central 20 degrees | Marked visual field defect<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in<br>the affected eye | • |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | | |
| Definition: A disorder characteri | zed by fear and avoidance of light. | 18 | di S | ! | |
| Retinal detachment | Asymptomatic zed by the separation of the inner n | Exudative and visual acuity 20/40 or better | Rhegmatogenous or exudative detachment; operative intervention indicated; de dine in vision (worse than 20/40 but better than 20/200) | Blindness (20/200 or worse) in<br>the affected eye | |
| Retinal tear | - | Laser therapy or p neumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in<br>the affected eye | |
| Definition: A disorder characteri | ा<br>zed by a small laceration of the reti | 7 <sub>7</sub> 1 | 57 | | |
| Retinal vascular disorder | | Topical medication indicated | Intravitreal medication;<br>operative intervention indicated | | |
| Definition: A disorder characteri | zed by pathological retinal blood ve | ssels that adversely affects vision | t. | 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked<br>decrease in visual acuity (worse<br>than 20/40); disabling; limiting<br>selfcare ADL | Blindness (20/200 or worse) in<br>the affected eye | |
| Definition: A disorder involving t | he retina. | 161<br> | (5) (5) | | |
| Soleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20 40 or better) | Symptomatio, limiting self care<br>ADL; marked decrease in visual<br>acuity (worse than 20/40) | Blindness (20/200 or worse) in<br>the affected eye | |
| Definition: A disorder characteri | zed by involvement of the sclera of | the eye. | , | , | |
| Uveitis | Asymptomatic; clinical or diagnostic observations only | Anterior uveitis; medical<br>intervention indicated | Posterior or pan-uveitis | Blindness (20/200 or worse) in<br>the affected eye | |
| | zed by inflammation to the uvea off | On the second record records | La accompanion de la companion | www.moreover. | |
| treo us hemorrhage | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL;<br>vitrectomy indicated | Blindness (20/200 or worse) in<br>the affected eye | - |
| Definition: A disorder characteri | zed by blood extravasation into the | vitreou's humor. | 5 | E | |
| Vatering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | 3 | |
| Definition: A disorder of excessi | ve tearing in the eyes; it can be cau | ised by overproduction oftears or | impaired drainage of the tear duo | 100 | |
| Eye disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately sight-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Sight-threatening consequences; urgent intervention indicated; blindness (20/200 or worse) in the affected eye | 7 |

CTCAE 4.0 - May 28, 2009 : Eye disorde &

CARTISTEM® 

| | 16 | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | : |
| % dominal distension | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self<br>care ADL | | |
| Definition: A disorder chara | acterized by swelling of the abdomen. | T- | T | | T |
| % dominal pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain ; limiting self care<br>ADL | | - |
| Definition: A disorder chara | acterized by a sensation of marked disc | omfort in the abdominal region. | ¥ | | - |
| Anal 1stula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tuble feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | Mild; intervention not indicated | 1/2. | | Life throatening conceasions of | Death |
| An al hemorrhage | acterized by bleeding from the anal region | Moderate symptoms; medical<br>intervention or minor<br>cauterization in dicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| An al mucositis | | 16 | C | 1 14 14 11 | Donah |
| ÷n al mucosπis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | acterized by inflammation of the mucous | membrane of the anus. | | | |
| Anal necrosis | | | TP N or hospitalization indicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder chara | acterized by a necrotic process occurring | g in the anal region. | 1 | | |
| ≏n al pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 8 | - |
| Definition: A disorder chara | acterized by a sensation of marked disc | omfort in the anal region . | N . | | (i) |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicate d | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated; TPN or hospitalization<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder chara | ,<br>acterized by a narrowing of the lumen of | the anal canal. | \$2007000740 B | , | (1)<br>(c) |
| An al ulœr | Asymptomatic; clinical or diagnostic observations only; intervention not indicate d | Symptomatic; altered GI function | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder chara | acterized by a circumscribed, in fammato | ory and necrotic erosive lesion on t | he mucosal surface of the analica | nal. | (2) |
| Ascites | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; invasive<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder chara | acterized by accumulation of serous or h | emorrhagic fluid in the periton eal | cavity. | 7 | - C |
| Hoating | No change in bowel function or oral intake | Symptomatic, decreased oral intake; change in bowel function | *) | 3 | 5 |
| Definition: A disorder chara | acterized by subject-reported feeling of u | un comfortable fullness of the abdo | men. | | 200 |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization in dicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| efinition: A disorder chara | acterized by bleeding from the cecum. | 5 | 2 | | |
| Cheilitis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | | · · |

CTCAE 4.0 - May 28, 2009 : Glastrola testical disorde s

CARTISTEM® 

| <u> </u> | | Gastrointestinal dis | oi dei S | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | ं |
| Colitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood<br>in stool | Severe abdominal pain; change<br>in bowel habits; medical<br>intervention indicated;<br>peritoneal signs | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | sterized by inflammation of the colon. | | | | |
| Colonic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an abnormal communication | between the large intestine and a | an other organ or anatomic site. | | Transaction |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | sterized by bleeding from the colon. | No. | at a second | | Terring |
| Colonic obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Ho spitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | sterized by blockage of the normal flow | of the intestinal contents in the co | lon. | | Perment |
| Colonic perforation | | Symptomatic; medical<br>intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by a rupture in the colonic wall. | S 60 for 55305 | \$257 (160 No.) \$253,000 (100 H) | (a20)0 yo | 120 00 |
| Colonic stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a narrowing of the lumen of t | the colon. | | | 100 |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | sterized by a circumscribed, in fammato | ry and necrotic erosive lesion on t | the mucosal surface of the colon. | | 2 |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with<br>regular use of laxatives or<br>enemas; limiting instrumental<br>ADL | Obstipation with manual<br>evalouation indicated; limiting<br>self care ADL | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder charac | terized by irregular and infrequent or di | flicult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis<br>or periapical abscess or<br>resulting in tooth loss | 2 | - |
| Definition: A disorder charac | sterized by the decay of a tooth, in which | h it becomes softened, discolored | and/orporous. | | |
| Diarrh ea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | In ore ase of 4-8 stools per day<br>over baseline; moderate<br>increase in ostomy output<br>compared to baseline | horease of >=7 stools per day<br>over baseline; in continence;<br>hospitalization in dicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by frequent and watery bowel n | novements. | To the state of th | | 7 |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake<br>alterations (e.g., copious water,<br>other lubricants, diet limited to<br>purees and or soft, moist foods);<br>unstimulated saliva 0.1 to 0.2<br>ml/min | hability to ad equately aliment<br>orally; tube feeding or TPN<br>indicated; unstimulated saliva<br><0.1 ml/min | | 1 |

CTCAE 4.0 - May 28, 2009 : Gastroli testical disorde s

CARTISTEM® 

| | | Gastrointestinal dis | sorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely attered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | terized by an abnormal communicatio | 128(07 St St St St St | Two sales seems a | District was | 05000040 |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the duoden u | m. | | | |
| Duodenal obstruction | Asymptomatic; clinical or<br>diagnostic observations only,<br>intervention not indicated | Symptomatic; altered GI function | Ho spitalization or elective<br>operative intervention indicated;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by blockage of the normal 10 w | of stomach contents through the | duodenum. | | |
| Duodenal perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a rupture in the duodenal w | all. | T-00 00 00 001000 00 | Transit et | Paris 100 |
| Duodenal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; ho spitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a narrowing of the lumen of | the duodenum. | 101 101 | 5.<br>U | 01<br>01 |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical<br>intervention indicated; limiting<br>instrumental ADL | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a circumscribed, in fammate | ory and necrotic erosive lesion on | the mucosal surface of the duoder | nal wall. | r |
| Dyspepsia | Mild symptoms; intervention not<br>indicated<br>terized by an uncomfortable, often pai | intervention indicated | Severe symptoms; surgical intervention indicated | home include huming stomach, blo | - |
| neartbum, nausea and vomi | NO 18 NO 10 | *** | | i | 53 |
| Dysph agia | Symptomatic, able to eat regular diet | Symptomatic and altered eating/swallowing | Severely aftered<br>eating/swallowing; tube feeding<br>or TPN or hospitalization<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by difficulty in swallowing. | | | | |
| Enterocolitis | Asymptomatic; clinical or<br>diagnostic observations only,<br>intervention not indicated | Abdominal pain; mucus or blood<br>in stool | d Severe or persistent abdominal<br>pain; fever; ileus; peritoneal<br>signs | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by inflammation of the small a | nd large intestines. | 100 00 00 00 00 00 00 0 | 10000 10 | PHO 80 |
| Entero ve sical fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; non invasive<br>intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an abnormal communicatio | n between the urinary bladder an | d the intestine . | - | |
| Esoph ageal fistula | Asymptomatic; dinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| | .1 | 10-<br>10-1 | (2) | | |
| Definition: A disorder charac | terized by an abnormal communicatio | n between the esophagus and an | other organ or an atomic site. | iz. | · · |

CTCAE 4.0 - May 28, 2009 : Glastroli testical disorde s

CARTISTEM® 

| | | Gastrointestinal di | suruers | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | -2 | 3 | 4 | |
| Esophageal ne <i>c</i> ro <i>s</i> is | | Secretary and the sec | hability to a liment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | eterized by a necrotic process occurring | in the esophageal wall. | 1 | 1 | |
| Esophageal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | sterized by blockage of the normal flow | V. 55 (2) (3) (3) | 155 1575555 7570 | I | |
| Esophageal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | • | * |
| Definition: A disorder charac | eterized by a sensation of marked disco | omfort in the esophageal region. | 1 | 1 | |
| Esophageal perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | sterized by a rupture in the wall of the e | sophagus. | | | |
| Esophageal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; ho spitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a narrowing of the lumen of | the esophagus. | | | |
| Esophageal uloer | Asymptomatic; clinical or<br>diagnostic observations only,<br>intervention not indicated | Symptomatic; altered GI<br>function; limiting in strumental<br>ADL | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | sterized by a circumscribled, in fammato | Burney or any and a second | 1/32 | Et en | Ť |
| Esophageal varices<br>hemorrhage | | Self-limited; intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | sterized by bleeding from esophageal v | 25 | 1 | I | Ī |
| Esophagitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered<br>eating/swallowing; oral<br>supplements indicated | Severely altered eating/swallowing; tube feeding, TPN or hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| TAN HONO CHOILE CHOCKENGAR | sterized by inflammation of the esopha | Alexander and an area and an area and an area | Tauxinama wantana ana ana an | 50 | ř. |
| Fecal incontinence | Occasional use of pads required | Daily use of pads required | Severe symptoms; elective operative intervention indicated | • | - |
| | sterized by inability to control the escap | | 10° = 27 | I | T |
| Flatulence | Mild symptoms; intervention not<br>indicated | psychosocial sequelae | | | |
| A STATE OF | sterized by a state of excessive gas in t | N N N N N N N N N N N N N N N N N N N | 187 18 30 SOUTH OF | 1575 G | - W |
| Gastrio fistula | Asymptomatic; dinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest; tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | sterized by an abnormal communication | n between the stornach and anoth | ner organ or anatomic site. | | r - |
| Ga stric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the gastric wa | all. | 1 | I | |
| Ga stric necro sis | | | hability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

CTCAE 4.0 - May 28, 2009 : Glastroli testical disorde s 15

**CARTISTEM®** 
| | | Gastrointestinal dis | surders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Gastric perforation Definition: A disorder charact | erized by a rupture in the stomach wa | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Gastrio stenosis | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening consequences; | Death |
| od stille stellosis | diagnostic observations only;<br>intervention not indicated | function | tube feeding; ho spitalization<br>indicated; elective operative<br>intervention indicated | urgent operative intervention indicated | Death |
| Definition: A disorder charact | erized by a narrowing of the lumen of | the stomach. | STATE AND ADDRESS OF A STATE OF THE STATE OF | | • |
| Ga stric ulcer | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening consequences; | Death |
| | diagnostic observations only,<br>intervention not indicated | function; medical intervention<br>indicated; limiting instrumental<br>ADL | TP N indicated; elective operative or endoscopic intervention indicated; limiting self care ADL; disabling | urgent operative intervention<br>indicated | |
| | erized by a circumscribed, in fammato | CARLES CONTROL OF LAND CONTROL OF | | If however, the state of the st | en<br>Percesse |
| Gastritis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated | Severely aftered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | erized by inflammation of the stornach | | Termonium managan ma | | in I |
| Gastroesophageal reflux<br>disease | Mild symptoms; intervention not<br>indicated | Moderate symptoms; medical<br>intervention indicated | Severe symptoms; surgical intervention indicated | | ŀ |
| | erized by reflux of the gastric and/or d | | 경기 회사 가장 아니는 아이들이 살아 있다면 하는데 그렇게 하는데 모르게 되었다. | nd usually caused by incompetenc | e ofthe l |
| | ay result in injury to the esophageal m | Co. C. | Control of the Contro | Y 11/2 (17/2 | Downer |
| Gastrointestinal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely aftered GI function;<br>tuble feeding, TPN or<br>hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | between any part of the gastroin | testinal system and another organ | or a natomic site. | 001 |
| Ga strointestinal pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | |
| Definition: A disorder charact | erized by a sensation of marked disco | mfort in the gastrointestinal regio | n. | | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to<br>maintain nutrition with dietary<br>and lifestyle modifications; may<br>need pharmacologic<br>intervention | Weight loss; refractory to<br>medical intervention; unable to<br>maintain nutrition orally | 8 | T |
| Definition: A disorder charact | erized by an incomplete paralysis ofth | '<br>he musdes ofthe stomach wall re | sulting in delayed emptying of the | ,<br>gastric contents into the small inte | stine. |
| Bingival pain | Mild pain | Moderate pain interfering with<br>oral intake | Severe pain; inability to aliment orally | - | 2 |
| Definition: A disorder charact | erized by a sensation of marked disco | omfort in the gingival region . | 101 109 10 | | 00 F |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization in dicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder charact | erized by bleeding from the hemorrhoi | ids. | 100 ST | | 001<br>T: |
| Hemorrhoids | Asymptomatic; dinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | 0 | |
| Definition: A disorder charact | erized by the presence of dilated vein: | s in the recturn and surrounding a | irea. | | 001 |
| leal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | between the ileum and another | organ or anatomic site. | | eri<br>P |
| leal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>caute rization in dicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Glastroln test hall disorde s

CARTISTEM® 

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | |
| eal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self-care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal 1 ou | of the intestinal contents in the il | eum. | | |
| leal perforation | | Symptomatic; medical<br>intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | erized by a rupture in the ileal wall. | P. | 1 | | r |
| leal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function | Severely aftered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen o | f the ileum. | F-0 | Towner et | |
| leal ulcer | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, in fammat | ory and necrotic erosive lesion or | the mucosal surface of the ileum. | · | 001 |
| leus | ŀ | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TP N indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| 1010 10 00 00 | erized by failure of the ileum to trans | V 55 125 125 125 125 | 10 10 101 1010 | 7772 0 | 12 7 |
| ntra-abdominal hemorrha ge | | Medical intervention or minor<br>cauterization in dicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding in the abdominal o | ca vity. | The state of the s | , | |
| Jejun al fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely aftered GI function;<br>TP N or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | erized by an abnormal communicatio | n between the jejunum and anoth | er organ or anatomic site. | V PROBLEMS SERVICE SERVICE STATES AND | or<br>Percenso |
| lejuna I h emorrhag e | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization in dicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the jejunal w | all. | (8) (8) (8) (9) (9 | | (8)<br>(0) |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting in strumental<br>ADL | Ho spitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal 10 w | of the intestinal contents in the j | ejunum. | | 7 |
| lejunal perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a rupture in the jejunal wall | F1 | m S | | 2 |
| Jejunal stenosis | Asymptomatic; dinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tuble feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen o | fthe jejunum. | | · | |
| lejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a circumscribed, inflammat | ory and necrotic erosive lesion or | the mucosal surface of the jejunum | n. | |
| Lip pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 8 | |

CTCAE 4.0 - May 28, 2009 : Glastroli testical disorde s

CARTISTEM® 

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | : |
| Lower ga strointestinal<br>hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by bleeding from the lower gas | strointestinal tract (small intestine, | large intestine, and anus). | | ř. |
| Malab sorption | Ī | Altered diet; oral intervention<br>indicated | hability to a liment adequately;<br>TP N indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | rerized by inadequate absorption of n | utrients in the small intestine. Sym | ptoms include abdominal marked o | discomfort, bloating and diamhea. | Tanana |
| Mucositis oral | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Moderate pain; not interfering<br>with oral intake; modified diet<br>indicated | Severe pain ; interfering with oral intake | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | rerized by inflammation of the oral mu | cosal. | interessed in the second secon | | 001<br>Tr |
| Nausea | Loss of appetite without alteration in eating habits | Oral intake decreased without<br>significant weight loss,<br>dehydration or malnutrition | ha dequate oral caloric or fluid<br>intake; tube feeding, TPN, or<br>hospitalization indicated | 50 | |
| | erized by a queasy sensation and/or | | | 110000000000000000000000000000000000000 | Dogwe |
| Obstruction gastric | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; limiting in strumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by blockage of the normal 10 w | of the contents in the stomach. | (A) | | (2)<br>(2) |
| Oral cavity fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal communicatio | n between the oral cavity and ano | ther organ or anatomic site. | | |
| Oral dysesthesia | Mild discomfort; not interfering with oral intake | Moderate pain; interfering with<br>oral intake | Disabling pain; tube feeding or TP N indicated | | |
| Definition: A disorder charact | rerized by a burning or tingling sensat | ion on the lips, to ngue or entire m | outh. | | r |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | rerized by bleeding from the mouth. | TS. | Ť · | | T |
| Oral pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | ľ |
| Definition: A disorder charact | erized by a sensation of marked disc | omfort in the mouth, tongue or lips | 1 | | ini. |
| Pancreatic duct stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a narrowing of the lumen of | fthe pancreatic duct. | 1 | | |
| Pancreatic 1 stula | Asymptomatic; dinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tuble feeding or TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by an abnormal communicatio | n between the pancreas and a not | her organ or anatomic site. | | |
| Pancreatic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by bleeding from the pancreas | <u> </u> | | La constitución de la constituci | |
| Pancreatic necrosis | | • | Tuble feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-thre atening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a necrotic process occurring | g in the pancreas. | 200 800 MOVED 100000 | OSOFO YO | |
| Pancreatitis | | Enzyme elevation or radiologic<br>in dings only | Severe pain; vomiting; medical intervention indicated (e.g., analgesia, nutritional support) | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : G as trols test hall disorde  $\sigma$ 

CARTISTEM® 

| | | Gastrointestinal disorders | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | - 5 |
| Definition: A disorder charac | terized by inflammation of the pancrea | ıs. | 10% | | 01 |
| Periodontal disease | Gingival recession or gingivitis;<br>limited bleeding on probing; mild<br>local bone loss | Moderate ging ival recession or<br>ging ivitis; multiple sites of<br>bleeding on probing; moderate<br>bone loss | Spontaneous bleeding; severe<br>bone loss with or without tooth<br>loss; o steonecrosis of maxilla or<br>mandible | 8 | 5 |
| Definition: A disorder in the | ging ival tissue around the teeth. | 10 | 16) 6 | 1 | 2 |
| Peritoneal necrosis | | | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | nterized by a necrotic process occurring | ; in the peritoneum. | Tanana and a same | | Ď |
| Proctitis | Rectal discomfort, intervention<br>not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | sterized by inflammation of the rectum. | ő | | | |
| Rectal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TP N or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an abnormal communication | between the rectum and anothe | r organ or an atomic site. | | 01 |
| Rectal he morrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization in dicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the rectal wal | l and discharged from the anus. | 10% | | ni. |
| Rectal mucositis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by inflammation of the mucous | membrane of the rectum. | 100 | | 01 |
| Rectal ne crosis | | - | Tube feeding or TPN indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a necrotic process occurring | in the rectal wall. | 100 | | ni- |
| Rectal ob struction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function; limiting in strumental<br>ADL | Ho spitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | sterized by blockage of the normal flow | of the intestinal contents in the re | ectum. | | 201 |
| Rectal pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 3 | 1 |
| | terized by a sensation of marked disco | | T second security of the second secon | | ni<br>Shrichan |
| Rectal perforation | | Symptomatic; medical<br>intervention indicated | Severe symptoms; elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a rupture in the rectal wall. | 50<br>703 | 181 III | | 51<br>(0) |
| Rectal stenosis | Asymptomatic; dinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a narrowing of the lumen of | the rectum. | T . | | r |
| Rectal ulcer | Asymptomatic; dinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function (e.g. altered dietary<br>habits, vomiting, diarrhea) | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

CTCAE 4.0 - May 28, 2009 : Gastroli testical disorde s

CARTISTEM® 

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | Grade 1 2 3 4 5 | | | |
| Adverse Event | 1 | 2 | 3 | 4 | ÷ |
| Retroperitoneal hemorrhage | isad bu blasding to make potencial | Self-limited; intervention indicated | Transfusion, medical, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rized by bleeding from the retroperit | 15 | I consider the contract of the | V 44/2 4 (10/2004) 1 4/2000 (4/2004) 1 (1/2004) 1 (1/2004) | L |
| Salivery duct in fammation | Slightly thickened saliva; slightly<br>altered taste (e.g., metallic) | Thick, ropy, sticky saliva;<br>markedly aftered taste;<br>afteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | Acute salivary gland necrosis; severe secretion-induced symptoms (e.g., thick saliva/oral secretions or gagging); tube feeding or TPN indicated; limiting self care ADL; disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the salivary | duct. | 0 | | 001 |
| Salivery gland fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatio; altered GI function; tube feeding indicated | Severely altered GI function;<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by an abnormal communicatio | n between a salivary gland and an | other organ or anatomic site. | | (2)<br>(2) |
| Small intestinal mu∞sitis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatio; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe pain; interfering with oral<br>intake; tube feeding, TPN or<br>hospitalization indicated; limiting<br>self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting in strumental<br>ADL | Ho spitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by blockage ofthe normal fow | of the intestinal contents. | 211111111111111111111111111111111111111 | | ~ |
| Small intestinal perforation | 184 | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a rupture in the small intest | ine wall. | | | |
| Small intestinal stenosis | Asymptomatic; clinical or diagnostic observations on ly; intervention not indicate d | Symptomatic; altered GI function | Symptomatic and severely altered GI function; tube feeding, TPN or hospitalization indicated; non-emergent operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a narrowing of the lumen of | the small intestine. | • | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicate d | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Severely altered GI function;<br>TP N indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a circumscribed, in fammat | ory and necrotic erosive lesion on | the mucosal surface of the small in | testine. | |
| Stomach pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | • | ŧ |
| Definition: A disorder character | ized by a sensation ofmarked disc | omfort in the stomach. | | | |
| Footh development disorder | Asymptomatic; hypoplasia of tooth or enamel | Impairment correctable with oral surgery | Maldevelopment with<br>impairment not surgically<br>correctable; disabling | | - |
| Definition: A disorder character | ized by a pathological process of th | e teeth occurring during tooth dev | elopment. | | |
| Footh discoloration | Surface stains | - | 159 | 20 | ŀ |
| Definition: A disorder character | ized by a change in tooth hue or tin | t. | 0. 2. 2. | | 001 |
| Foothache | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | E . | |

CTCAE 4.0 - May 28, 2009 : Glastrolytes thial disorde is

CARTISTEM® 

| | | Gastrointestinal dis | sorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Typhlitis | | | Symptomatic (e.g., abdominal<br>pain, fever, change in bowel<br>habits with ileus); peritoneal<br>signs | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by inflammation of the decum. | 1 | | | _ |
| Upper ga strointestinal<br>hernorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the upper gas | strointestinal tract (oral cavity, pha | arynx, esophagus, and stomach). | - | |
| Vorniting | 1 - 2 episodes (separated by 5<br>minutes) in 24hrs | 3 - 5 episodes (separated by 5<br>minutes) in 24 hrs | >=6 episodes (separated by 5<br>minutes) in 24 hrs; tube feeding,<br>TPN or hospitalization indicated | • | Death |
| Definition: A disorder characte | erized by the reflexive act of ejecting t | the contents of the stomach throu | gh the mouth. | | |
| Gastrointestinal disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Gastrointestinal disorders 21

CARTISTEM® 

| | General | disorders and administra | | | |
|---|---|---|---|---|---|
| 1 | | Grade | | | |
| Adverse Event | 1: | 2 | 3 | 4 | - 5 |
| Chills | Mild sensation of cold;<br>shivering; chattering of teeth | Moderate tremor of the entire body; narcotics in dicated | Severe or prolonged, not responsive to narcotics | S | ŀ |
| Definition: A disorder chara | acterized by a sensation of cold that ofte | n marks a physiologic response to | sweating after a fever. | | - |
| Death neon atal<br>Definition: A disorder chara | -<br>acterized by cessation of life occurring di | -<br>uring the first 28 days of life. | <b>5</b> | | Death |
| Death NOS | 1 | | | 16 | Death |
| Definition: A cessation of li | fe that cannot be attributed to a CTCAE | term a ssociated with Grade 5. | | , | 2 |
| Edema face | Localized facial edema | Moderate localized facial<br>edema; limiting in strumental<br>ADL | Severe swelling; limiting self care ADL | 3 | 7 |
| Definition: A disorder chara | acterized by swelling due to excessive 10 | uid a coumulation in facial tissues. | 00 00 | 2 | (X)<br>(X) |
| Edema limb s | 5 - 10 % inter-limb discrepancy<br>in volume or circumference at<br>point of greatest visible<br>difference; swelling or<br>obscuration of anatomic<br>architecture on close inspection | >10 - 30 % inter-limb<br>discrepancy in volume or<br>circumference at point of<br>greatest visible difference;<br>readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | >30 % inter-limb discrepancy in<br>volume; gross deviation from<br>normal anatomic contour;<br>limiting self care ADL | | 5 |
| Definition: A disorder chara | acterized by swelling due to excessive 10 | uid a coumulation in the upper or lo | wer extremities. | | |
| Edema trunk | Swelling or obscuration of<br>anatomic architecture on close<br>inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | anatomic contour; limiting self | 8 | i. |
| Definition: A disorder chara | acterized by swelling due to excessive 10 | uid a coumulation in the trunk area | | | |
| acial pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 8 | |
| Definition: A disorder chara | acterized by a sensation of marked disco | omfort in the face. | % V | 5 | (6) |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest;<br>limiting instrumental ADL | Fatigue not relieved by rest, limiting self care ADL | omplich daily activities | |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39 D - 40.0 degrees C (102.3 - 104.0 degrees F) | >40.0 degrees C (>1040<br>degrees F) for <=24 hrs | >40.0 degrees C (>104.0<br>degrees F) for >24 hrs | Death |
| Definition: A disorder chara | acterized by elevation of the body's temp | erature above the upper limit of n | ormal. | | |
| Flu like symptoms | Mild fu-like symptoms present. | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | | - |
| Definition: A disorder chara<br>cough. | acterized by a group of symptoms similar | r to those observed in patients with | hthe flu. It includes fever, chills, b | ody a ches, malaise, loss of appeti | te and d |
| Gait disturbance | Mild change in gait (e.g., wide-<br>based, limping or hobbling) | Moderate change in gait (e.g.,<br>wide-based, limping or<br>hobbling); assistive device<br>indicated; limiting instrumental<br>ADL | Disabling; limiting self care ADL | 5 | |
| Definition: A disorder chara | acterized by walking difficulties. | <b>3</b> 0 | X | 7 | 2 |
| Hypothermia | • 8 | 35 - >32 degrees C; 95 - >89.6<br>degrees F | 32 - >28 degrees C; 89.6 -<br>>82.4 degrees F | <=28 degrees C;82 4 degrees<br>F; life-threatening<br>consequences (e.g., coma,<br>h ypotension, pulmonary edema, | Death |

CTCAE 4.0 – May 28 , 2009 : General disorders and admin light rations the conditions

CARTISTEM® 

| 3 | General | disorders and administra | | | |
|---|---|---|---|---|---|
| | | E | Grade | 1 | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Infusion related reaction | Mild transient reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV1uids); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic me dication and/or brief interruption of in fusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by adverse reaction to the infu: | sion of pharmacological or biologic | al substances. | | |
| Infusion site extravasation | | Erythema with associated<br>symptoms (e.g., edema, pain,<br>induration, phlebitis) | Uceration or necrosis; severe<br>tissue damage; operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ized by leakage of a pharmacologic<br>reation and marked discomfort at th | | nfusion site into the surrounding ti | ssue. Signs and symptoms includ | e indurati |
| Injection site reaction | Tendemess with or without associated symptoms (e.g., warmth, erythema, itching) | Pain ; lipodystrophy; edema ;<br>phlebitis | Uceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an intense adverse reaction | (usually immunologic) developing | at the site of an injection. | 1 | |
| Imitability | Mild; e asil y consolable | Moderate; limiting instrumental<br>ADL; increased attention<br>indicated | Severe abnormal or excessive<br>response; limiting self care ADL;<br>inconsolable | | |
| Definition: A disorder character<br>condition . | ized by an abnormal responsivenes | s to stimuli or physiological arousa | al; may be in response to pain, frig | ht, a drug, an emotional situation | or a medi |
| Lo calized edema | Localized to dependent areas,<br>no disability or functional<br>impairment. | Moderate localized edema and<br>intervention indicated; limiting<br>instrumental ADL | Severe localized edema and<br>intervention indicated; limiting<br>self care ADL | | |
| Definition: A disorder character | ized by swelling due to excessive to | uid a coumulation at a specific anat | tomic site. | | ni<br>T |
| Malai se | Uneasiness or lack of well being | Uneasiness or lack of well being; limiting instrumental ADL | | 72 | |
| Definition: A disorder character | ized by a feeling of general discomf | ort or uneasiness, an out-of-sorts | feeling. | | |
| Multi-organ failure | | | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities | Life-threatening consequences<br>(e.g., vasopressor dependent<br>and oliguric or anuric or<br>ischemic colitis or lactic<br>acidosis) | Death |
| Definition: A disorder character | ized by progressive deterioration of | the lungs, liver, kidney and dotting | g mechanisms. | t. | · |
| Neck ederna | Asymptomatic localized neck<br>edema | Moderate neck edema; slight<br>obliteration of a natomic<br>landmarks; limiting instrumental<br>ADL | Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | 2 | 1 |
| Definition: A disorder character | ized by swelling due to an accumula | ation of excessive fluid in the neck | ž | | r |
| Non-cardiac chest pain | Mild pain | Moderate pain ; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 23 | - |
| Definition: A disorder character | ized by discomfort in the chest unre | lated to a heart disorder. | w G | is . | en en |
| Pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 2 | 1 |
| | ized by the sensation of marked dis | comfort, distress or agony. | 75<br>70<br>1 | I | tol<br>Tentesso |
| Sudden death NOS | 20 20200 00 2000 0 | 10 1 | # (50 9590) | 10 | Death |
| Definition: An unexpected cess | ation of life that cannot be attributed | to a CTCAE term associated with | Grade 5. | | |
| General disorders and<br>administration site conditions -<br>Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCA E 4.0 - May 28 , 2009 : General disorders and admin light ration site conditions

CARTISTEM® 

| | 10 | Hepatobiliary diso | rders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | |
| Bile duct stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Severely altered GI function;<br>radiologic, endo scopic or<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | terized by a narrowing of the lumen o | f the bile duct. | | | |
| Biliary fistula | | Symptomatic and intervention not indicated | Severely altered GI function;<br>TP N indicated; endoscopic<br>intervention indicated; elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | terized by an abnormal communication | n between the bile ducts and a not | ner organ or an atomic site. | Parking appe | Constant |
| Chole cystitis | 6 ts | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | terized by inflammation involving the | gallbladder. It may be associated w | ith the presence of gallstones. | *************************************** | 20 |
| Gallbladder istula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Symptomatic or severely altered<br>GI function; TPN indicated;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | terized by an abnormal communication | in between the galibladder and and | ther organ or anatomic site. | riz a constitution of the | D |
| Gallbladder necrosis | | | | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder charact | terized by a necrotic process occurrin | g in the gallbladder. | N. V. | | (i) |
| Gallbladder obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Symptomatic and severely altered GI function; tube feeding, TPN or hospitalization indicated; non-emergent operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | terized by blockage of the normal flow | ofthe contents ofthe gallbladder | The second of the | | |
| Gallbladder pain | Mild pain | Moderate pain ; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | es . | ž |
| Definition: A disorder charact | terized by a sensation of marked disc | omfort in the gallbladder region. | | | |
| Gallbladder perforation | 1 | | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by a rupture in the gallbladder | wall. | X V | | (4) |
| Hepatic failure | | 20 | Asterixis; mild encephalopathy;<br>limiting selfcare ADL | Moderate to severe<br>encephalopathy; coma; life-<br>threatening consequences | Death |
| | terized by the inability of the liver to m | netabolize chemicals in the body. L | ab oratory test results reveal abnor | mal plasma levels of ammonia , bi | lirubin, l |
| de hydrogen ase , and alkaline<br>Hepatic hemorrhage | Mild; intervention not indicated | Symptomatic; medical intervention indicated | Transfusion indicated | Life-threatening consequences; | Death |
| Definition: A disorder charact | I<br>terized by bleeding from the liver. | gyreche namenaou nambiétada Aus<br>197 | ž. | | |
| Hepatic necrosis | | | -38 | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder charact | <br>terized by a necrotic process occurrin | ι<br>σ in the henatic narenchuma | ž. | verravir in divale d | Ī |
| Hepatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | i i | |
| Definition: A disorder charact | ।<br>terized by a sensation of marked disc | K = | | | 25 |
| Perforation bile duct | 1.53 | | Radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

CTCAE 4.0 - May 28 , 2009 : Hepatobillary disorders

CARTISTEM® 

| 4 | | Hepatobiliary disc | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1. | 2 | 3 | 4 | 5 |
| Portal hypertension | | Decreased portal vein flow | Reversal/fetrograde portal vein<br>flow; associated with varices<br>and/or ascites | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | ed by an increase in blood pressu | re in the portal venous system. | · | | - |
| Portal vein thrombosis | | Intervention not indicated | Me dical intervention in dicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | ed by the formation of a thrombus | (blood clot) in the portal vein. | 27 S | 5 08 | T. |
| Hepatobiliary disorders - Other,<br>specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Hepatobiliary disorders 25 CTCAE 4.0 - May 28, 2009 : Immune system disorders 26

CARTISTEM® 

| | AV. | Immune system dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Allergic reaction | Transient flushing or rash, drug<br>fever <38 degrees C (<100.4<br>degrees F); intervention not<br>indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophyla ctic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic me dication and/or brief interruption of in fusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rized by an adverse local or general | response from exposure to an alle<br>T | rgen.<br>T | | É |
| An aphylaxis | | | Symptomatic bronchospasm, with or without urticaria; parenteral intervention indicated; allergy-related edema/angio edema; hypotension | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ized by an acute inflammatory react<br>presents with breathing difficulty, dia | 경영 : 10 (2.11) : 1 | | . () (~11.74) (~14.8) () ( ) ( ) ( ( ) ( ) ( ) ( ) ( ) ( ) | ypersensitiv |
| Autoimmune disorder | Asymptomatic; serologic or | Evidence of autoimmune | Autoimmune reactions involving | Life-threatening consequences; | Death |
| | other evidence of autoimmune<br>reaction, with normal organ<br>function; intervention not<br>indicated | reaction involving a non-<br>essential organ or function (e.g.,<br>hypothyroidism) | major organ (e.g., colitis,<br>anemia, myocarditis, kidney) | urgent intervention indicated | |
| Definition: A disorder resulting | from loss of function or tissue destru | Iction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses ofthe individ | ual to his ow |
| Cytokine release syndrome | Mild reaction; infusion interruption n ot indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NS AIDS, narcotics, IV fluids); prophylactic medications indicated for <= 24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic me dication and/or brief interruption of in fusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences;<br>pressor or ventilatory support<br>indicated | Death |
| Definition: A disorder character | ized by nausea, headache , tachyca | rdia , hypotension, ra <i>s</i> h , and shorti | ness of breath; it is caused by the | release of cytokines from the cells | ,<br>s. |
| Serum siokness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate arthralgia; fever, rash,<br>urticaria, antihistamines<br>indicated | Severe arthralgia or arthritis;<br>extensive rash; steroids or IV<br>fuids indicated | Life-threatening consequences;<br>pressor or ventilatory support<br>indicated | b., |
| | i zed by a delayed-type hypersensiti<br>he foreign antigen. Symptoms includ | | | 그런 경우 하나 아니다 아니라 이 유민들은 사람이 되었다. | |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninva sive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | 10000-20 |

CARTISTEM® 

**CONFIDENTIAL:** These all contents herein are the sole property of MEDIPOST Co., Ltd. Any reproduction or distribution of this document without the written consent of MEDIPOST Co., Ltd is prohibited. Copyright © 2017 MEDIPOST Co., Lt

| | Ţ. | Infections and infes | aations | | |
|---|---|---|---|---|---|
| | | - | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ab dominal infection | | | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara- | cterized by an infectious process invo | olving the abdominal cavity. | 1 | | |
| An orectal in fection | Localized ; local intervention indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | antiviral intervention in dicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | cterized by an infectious process invo | olving the anal area and the rectum. | THE PASSAGES AND THE | Todovo enss | SS<br>Descrease |
| Appendicitis | | 5)<br> | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara- | cterized by acute inflammation to the | vermiform appendix caused by a p | athogenic agent. | T | ř. |
| | cterized by acute inflammation to the | | 요즘 그렇게 하는 것이 되면 있었다. 그는 이번 그렇게 하지만 하게 되었다. | | Death<br>the |
| appendicearwan, me appe<br>Anteritis infective | | | Mantibiotic, antifungal, or | Life-threatening consequences; | Death |
| A lenus in e une | | | antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | urgent intervention indicated | Death |
| Definition: A disorder chara | cterized by an infectious process invo | olving an artery. | (6) V | ii | (i) |
| Biliary tract infection | 2 | (S) (N) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | terized by an infectious process invo | olving the biliary tract. | URPER CONCOUNTER OF CHEROCOLUMN AS | or . | |
| Bladder infection | | Oral intervention indicated (e.g., antibiotic, antifungal, antibiral) | Mantibiotic, antifungal, or antiviral intervention in dicated; radiologic, endo scopic, or operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder chara- | cterized by an infectious process invo | olving the bladder. | TERRESONAL PROPERTY CONTRACTOR AND AND CONTRACTOR A | | 2 |
| Bone infection | | -<br>-<br>- | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder chara- | cterized by an infectious process invo | olving the bones. | Ÿ. | | - |
| Breast infection | 100<br>8 | Local infection with moderate<br>symptoms; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral) | Severe infection; axillary<br>adenitis; f/ antibacterial,<br>antifungal, or antiviral<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | oterized by an infectious process invo | · · | T | | F |
| Bronchial infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | cterized by an intectious process invo | olving the bronchi. | 1. No temperation and the control of | | |
| Catheter related infection | | Localized; local intervention<br>indicated; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder chara | cterized by an infectious process that | t arises secon dany to catheter use. | The second of the | C AND | 1 |
| Cecal infection | 75 | ti e | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28 , 2009 : Intections and intestations

CARTISTEM® 

| 5 | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | - 5 |
| Definition: A disorder characte | rized by an infectious process | involving the œcum. | 103 | ı <sub>l</sub> | 001 |
| Cervicitis infection | rized by an infectious process | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | Tiecd by an inicatods process | Localized: local intervention | N/metiblishis metiblished on | Life-threatening consequences; | Death |
| Conjunctivitis infective | 100 20 | indicated (e.g., to pical a ntibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving the conjunctiva. Clinical manif | estations include pink or red color | in the eyes. | |
| Come al infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antifural) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving the cornea. | DV 10100 C4 100 to: | D13040 F3 | 1000 000 |
| Cranial nerve in fection | | 8) | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving a cranial nerve. | | | |
| Device related infection | | Ťo | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving the use of a medical device. | | | |
| Duodenal infection | The second second | Moderate symptoms; medical<br>intervention indicated (e.g., oral<br>antibiotics) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving the duodenum. | | | |
| En cephalitis infection | | | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>severe changes in mental<br>status; self-limited seizure<br>activity; focal neurologic<br>abnormalities | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving the brain tissue. | 1 | | |
| En cep halomyelitis infection | 1 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving the brain and spinal cord tissu | es. | | |
| Endocarditis infective | | | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process | involving the endocardial layer of the he | art. | | |
| En dophthalmitis | ) <b>9</b> 4 | Local intervention indicated | Systemic intervention or hospitalization in dicated | Blindness (20/200 or worse) | |

CTCAE 4.0 - May 28 , 2009 : Intections and intestations

CARTISTEM® 

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1: | 2 | 3 | 4 | |
| Enterocolitis infectious | -<br>acterized by an infectious process invol | Passage of >3 unformed stools<br>per 24 hrs or duration of illness<br>>48 hrs; moderate abdominal<br>pain | Mantibiotic, antifungal, or antiviral intervention in dicated; radiologic, endo scopic, or operative intervention indicated; profuse watery diarrhea with signs of hypovolemia; bloody diarrhea; fever; severe abdominal pain; ho spitalization indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | l l | TO THESE STORE AND THE | K245:-4441 | 1:6 4 - 4::- | Death |
| Esophageal infection | 100 | Local intervention indicated<br>(e.g., oral antibiotic, antifungal,<br>antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | acterized by an infectious process invol | ving the esophagus. | Q* = 24 | | ni<br>Evenesia |
| Eye infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated;<br>enucleation | Death |
| Jefinition: A disorder chara | acterized by an infectious process invol | ving the eye. | Ť | | i . |
| Gallbladder infection | | | M antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | acterized by an infectious process invol | ving the gallbladder. | | | |
| Gum infection | Local therapy indicated (Swish and swallow) | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | acterized by an infectious process invol | ving the gums. | Meta-control meta-control participation (Control participation (Cont | , | |
| Hepatic infection | | | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | acterized by an infectious process invol | ving the liver. | 0 | | ni. |
| Hepatitis viral | Asymptomatic, treatment not<br>indicated | | Symptomatic liver dysfunction;<br>fbrosis by biopsy; compensated<br>cirrhosis, reactivation of chronic<br>hepatitis | Decompen sated liver function<br>(e.g., a soites, coagulopathy,<br>encephalopathy, coma) | Death |
| Definition: A disorder chara | acterized by a viral pathologic process i | nvolving the liver parenchyma. | 1 | | |
| infective myositis | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder chara | acterized by an infectious process invol | ving the skeletal muscles. | | | |
| Joint in fection | | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); needle aspiration indicated (single or multiple) | Arthroscopic intervention indicated (e.g., drainage) or arthrotomy (e.g., open surgical drainage) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| AND THE DESIGNATION OF THE | acterized by an infectious process invol | ving a joint. | and the second second | Liz and the second | 6 |
| √idney in fection | | | M antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Intections and intestations

CARTISTEM® 

| 5 | | Infections and infes | Infections and infestations | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | - 5 |
| aryngitis | 28 | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | cterized by an inflammatory process i | involving the larynx. | | | |
| Lip in fection | Localized , local intervention indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | | - |
| | cterized by an infectious process invo | T 1000 | | 1886 G | 122 W |
| Lung infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | M antibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | cterized by an infectious process invo | FIGURE SERVICE CONTRACTOR AND ASSESSED. | | | 12ssae |
| Lymph gland in fection | | Localized; local intervention<br>indicated (e.g., to pical antibiotic,<br>antifungal, or antiviral) | M antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | cterized by an infectious process invo | olving the lymph nodes. | 1 | | - |
| Media stinal infection | | | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | oterized by an infectious process invo | olving the mediastinum. | | 1 | r |
| Meningitis | | | M antibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | cterized by acute inflammation of the | meninges of the brain and/or spinal | cord. | 2 | (a) |
| Mucosal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | oterized by an infectious process invo | olving a muco sal surface. | T . | | r |
| Nail infection | Localized, local intervention<br>indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | M antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | | |
| Definition: A disorder chara | oterized by an infectious process invo | olving the nail. | | | |
| Otitis externa | 200 | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | cterized by an infectious process invo | | | ive water exposure (swimmer's ea | rinfectio |
| ALCOHOLOGICA DE COMPANION DE CO | ymptoms include fullness, itching, sw | WEST CANDIDATES OF THE PROPERTY OF THE PROPERT | UNICESSALE STATE SALES AND ASSAULT | | in the same |
| Dtitis media | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | M antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder chara | cterized by an infectious process invo | olving the middle ear. | 1 | - | ř. |
| Ovarian in fection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Intections and intestation

CARTISTEM® 

| 8 | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | -2 | 3 | 4 | 5 |
| Pancreas in fection | La Company | | M antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involvi | ing the pancreas. | , | | |
| Papulopustular rash | Papules and/orpustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30 % BSA, which may or may not be associated with symptoms of pruritus or tendemess; associated with psychosocial impact; limiting instrumental ADL | Papules and for pustules covering >30% BSA, which may or may not be a ssociated with symptoms of pruritus or tendemess; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tendemess and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | rized by an eruption consisting of pa | | | | , and up |
| | his rash does not present with whiteh | | | sions. | T T |
| Paronychia | Nail fold edema or erythema;<br>disruption of the cuticle | Localized intervention indicated;<br>oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral;<br>nail fold edema or erythema<br>with pain; associated with<br>discharge or nail plate<br>separation; limiting instrumental<br>ADL | Surgical intervention or IV<br>antibiotics indicated; limiting self<br>care ADL | | |
| Definition: A disorder characte | rized by an infectious process involvi | ing the soft tissues around the nai | li . | | 2 |
| Pelvic infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involvi | ing the pelvic cavity. | 1 | | r - |
| Penile infection | - | Localized; local intervention<br>indicated (e.g., to pical antibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involvi | ing the penis. | <b>F</b> 44000940040040400000000000000000000000 | , | |
| Periorbital infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involved | ing the orbit of the eye. | ali eti | Windows Company College Colleg | ni<br>Perusus |
| Peripheral nerve in fection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | M antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involvi | ing the peripheral nerves. | 1 | | 7 |
| Peritoneal infection | | | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | rized by an infectious process involvi | ing the peritoneum. | | | |
| Pharyngitis | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | rized by inflammation of the throat. | | T | - | |
| Phlebitis infective | - Hel | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 25 , 2009 : Intections and intestations 31

CARTISTEM® 

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characte<br>of the infected vein. | rized by an infectious process invo | living the vein. Clinical manifestation | s include erythema, marked disco | mfort, swelling, and induration alo | ng the course |
| Pleural infection | | Localized; local intervention indicated (e.g., to pical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | lving the pleura . | 1 | | |
| Prostate infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | lving the prostate gland. | W 11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | |
| Rash pustular | | Localized; local intervention indicated (e.g., to pical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | | |
| Definition: A disorder characte | rized by a circumscribed and eleva | ated skin lesion filled with pus. | | | <u> </u> |
| Rhinitis infective | | Localized; local intervention<br>indicated (e.g., to pical antibiotic,<br>antifungal, or antiviral) | | | į |
| Definition: A disorder characte | rized by an infectious process invo | lving the nasal mucosal. | ali pondominacione de la compania del compania de la compania del compania de la compania del la compania de la compania del la compania de la compania de la compania del la compania del la compania del compania del la compania del la compania del la compania del la compania | | ni sa |
| Salivary gland infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | M antibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| C very consistent was all const | rized by an infectious process invo | State of the second sec | Transport of the second | IZ TO CATTO A COLONIA MASSAN INCOMENTA | Laconomic Contraction of the Con |
| Scrotal infection | 100 ISS 6000001 ISS 60 A | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rized by an infectious process invo | lving the scrotum. | 1 | | r |
| Sepsis | 1 | • | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| - Company of the Comp | rized by the presence of pathogen | ic microorganisms in the blood strea | | 1458 | Contraction 1 |
| Sinusitis | 100 TO 500 SERVICE TO FIRST | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | | lving the mucous membranes of the | | | 1 |
| Skin infection | Localized, local intervention indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | lving the skin. | Low yours on one or | Incorp 20 | Page 10 2 |
| Small intestine infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | lving the small intestine. | 90 St | T I | 01<br>01 E3 |
| Soft issue in fection | 978 | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | lving so <b>t</b> tissues. | 6<br>- | E . | (h) |
| Splenic in fection | • | | f√antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Intections and intestations

CARTISTEM® 

| | Infections and infestations | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disord er characteri | zed by an infectious process involvi | ng the spleen. | Q | | 001 |
| Stoma site infection | Localized , local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ng a stoma (surgically created op | ening on the surface of the body). | | T. |
| Tooth infection | -<br>zed by an infectious process involvi | Localized; local intervention indicated (e.g., to pical antibiotic, antifungal, or anti viral) | M antibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Fracheitis | Lea by an intections process involvi | Moderate symptoms; oral | Mantibiotic, antifungal, or | Life-threatening consequences; | Death |
| racrieus | | intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | antiblotic, antiblogar, of<br>antibral intervention indicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ng the trachea. | | | |
| Upper respiratory infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antifural intervention indicated;<br>radiologic, endo scopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ng the upper respiratory tract (no: | se, paranasal sinuses, pharynx, la | rynx, or trachea). | 001 |
| Urethral infection | ana | Localized; local intervention indicated (e.g., to pical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ng the urethra. | 6 | | (2)<br>(1) |
| Urinarytract infection | 425 | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ng the urinary tract, most commo | nly the bladder and the urethra. | | |
| Uterine infection | | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ng the endometrium. It may exten | d to the myometrium and parame | trial tissues. | |
| √a ginal infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disord er cha racteri | zed by an infectious process involvi | ng the vagina. | at a | | 001 |
| vUlval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characteri | zed by an infectious process involvi | ng the vulva. | 6 | ¥. | (%) |
| Wound in fection | da" " | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | Mantibiotic, antifungal, or<br>antiviral intervention in dicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri: | ा<br>zed by an infectious process involvi | ng the wound. | encredadentilitation (1707) | 1 | 1 |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or me dically significant but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization in dicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 25 , 2009 : Intections and line stations 33

CARTISTEM® 

| | Injury | , poisoning and procedu | 100000000000000000000000000000000000000 | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| nikle fracture | Mild; non-surgical intervention<br>indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective<br>surgery indicated | • | · |
| Definition: A finding of damage to<br>offected leg and foot. | o the ankle joint characterized by: | a break in the continuity of the ank | le bone. Symptoms include marke | d discomfort, swelling and difficult | y moving 1 |
| Aortic injury | | į. | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| Province accepted which the | | 12 | care ADL; disabling; repair or<br>revision indicated | e vidence of end organ damage;<br>urgent operative intervention<br>indicated | |
| Definition: A finding of damage t | o the aorta. | 16 | 1 | | |
| Arterial injury | Asymptomatic diagnostic<br>finding ; intervention not<br>indicated | Sympto matic (e.g., claudication); repair or revision not in dicated | Severe symptoms; limiting self-<br>care ADL; disabling; repair or<br>revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage t | o an artery. | 20 | 7 | | 20 |
| Biliary an astomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage o | f bile due to breakdown of a biliar, | / anastomosis (surgical connection | oftwo separate anatomic structu | res). | 2 |
| Bladder ana stomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage o | furine due to breakdown of a blad | der anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | 2 |
| Bruising | Localized or in a dependent area | Generalized | 50 | 5 | |
| Definition: A finding of injury ofth | ne soft tissues or bone characteriz | ed by leakage of blood into surrou | nding tissues. | | |
| Bum | Minimal symptoms; intervention not indicated | Medical intervention; minimal debridement indicated | Moderate to major debridement or reconstruction indicated | Life-threatening consequences | Death |
| | ntegrity to the anatomic site of an<br>depends on the length and intensi | | | nicals, direct heat, electricity, flam | es and |
| Dermatitis radiation | Faint enythema or dry | Moderate to brisk erythema; | Moist desquamation in areas | Life-threatening consequences; | Death |
| | desquarmation | patch y moist desquamation ,<br>mostly confined to skin folds<br>and creases; moderate edema | other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | |
| Definition: A finding of outaneou: | s in fammatory reaction occurring: | as a result of exposure to biologica | ally effective levels of ionizing radia | ation. | )C1 |
| Esophageal ana stomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an esophagea | Il an astomosis (surgical connection | n oftwo separate a natomic structu | res). | ž) |
| Fall : | Minor with no resultant injuries; intervention not indicated | Symptomatic; noninvasive intervention indicated | Ho spitalization indicated | Ī. | 5 |
| Definition: A finding of sudden m | ovement downward , usually result | ting in injury. | | | |
| Fallopian tub e anastomotic leak | Asymptomatic; dinical or diagnostic observations only; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of lankage d | . <b></b> | | | No. of the second secon | Ŀ |
| 기용되다 어디 전기사람 | ue to breakdown of a fallopian tub | S. 50 (CE) VAN (CE) | | SANT GES | D |
| Fallopian tube perforation | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms; elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A finding of rupture of | the fallopian tube wall. | 50 | Z = 2 | A CONTRACTOR OF THE PROPERTY OF THE STATE OF THE SECTION OF THE SE | SC |
| Fracture | Asymptomatic; dinical or diagnostic observations only; intervention not indicated | Symptomatic but non-displaced;<br>immobilization indicated | Severe symptoms; displaced or<br>open wound with bone<br>exposure; disabling; operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009: Injury, polsoning and procedural complications

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | - 5 |
| Gastric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated ue to breakdown of a gastric anas | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Ga strointestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a gastrointesti | n al anastomosis (surgical connec | tion of two separate anatomic struc | ctures). | 20 |
| Ga strointestinal stoma necrosis | | Superficial necrosis;<br>intervention not indicated | Severe symptoms;<br>hospitalization or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of a necrotic | process occurring in the gastroint | te stinal tract stoma. | 1 | | r |
| Hip fracture | | Hairline fracture; mild pain;<br>limiting instrumental ADL; non-<br>surgical intervention indicated | Severe pain; hospitalization or<br>intervention indicated for pain<br>control (e.g., traction); operative<br>intervention indicated | Life-threatening consequences;<br>symptoms associated with<br>neurovascular compromise | |
| Definition: A finding of traumatic | injury to the hip in which the contin | nuity of either the femoral head, fe | moral neck, intertrochanteric or su | btrochanteric regions is broken. | |
| Injury to carotid artery | - | • | Severe symptoms; limiting self<br>care ADL (e.g., transient<br>cerebral ischemia); repair or<br>revision indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the carotid artery. | | | | |
| Injury to inferior vena cava | 83<br>mrs - 1946 | • | • es | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the inferior vena cava. | | - | | |
| Injury to jugular vein | 200 | | Symptomatic limiting self care<br>ADL; disabling; repair or<br>revision indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the jugular vein. | | | | |
| Injury to superior vena cava | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; repair or revision<br>not indicated | Severe symptoms; limiting self<br>care ADL; disabling; repair or<br>revision in dicate d | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | the superior vena cava. | | * | x overnormorm | |
| Intestinal storna leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| E 2000 E 20 | ficontents from an intestinal stoma<br>T | POSITION OF THE POSITION AND THE POSITIO | | D8890 /0 | 1233 98 |
| Intestinal stoma obstruction | - | Self-limited; intervention not indicated | Severe symptoms; IV fluids,<br>tuble feeding, or TPN indicated<br>>= 24 hrs; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of blockage | ofthe normal flow ofthe contents | of the intestinal stoma. | | | 00 |
| Intestinal storna site bleeding | Minimal bleeding identified on<br>clinical exam; intervention not<br>indicated | Moderate bleeding; medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A finding of blood leak | age from the intestinal stoma. | F(2) | 6 | | (%)<br>(%) |
| Intraoperative arterial injury | Primary repair of injured organ/structure in dicate d | Partial resection of injured<br>organ /structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A finding of damage to | an artery during a surgical proce | dure. | | | |
| Intraoperative breast injury | Primary repair of injured<br>organ/structure in dicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 25, 2009 : In(417, poleoning and procedural complications  $36\,$ 

CARTISTEM® 

| | Injury, poisoning and procedural complications Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1: | -2 | 3 | 4 | - 5 |
| Definition: A finding of damage to | the breast parenchyma during | a surgical procedure. | 105 | en e | 101 |
| Intraoperative cardiac injury | | | Primary repair of injured organ /structure indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | o the heart during a surgical pro | cedure. | Tab As 30 9998 UV | TERRORS ONES | Lossocae |
| Intraoperative ear injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injure d<br>organ/structure indicated | Complete resection of injured<br>organ structure indicated;<br>disabling (e.g., impaired<br>hearing; impaired balance) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | othe ear during a surgical proo | e'dure. | The national engineering | Elj | Percesso |
| Intraoperative endocrine injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the endocrine gland during a : | surgical procedure. | 197 | Est. | 177 |
| Intraoperative gastrointestinal<br>injury | Primary repair of injure d<br>organ/structure indicate d | Partial resection of injured<br>organ/structure in dicated | Complete resection or<br>reconstruction of injured<br>organ structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the gastrointestinal system du | iring a surgical procedure. | | | |
| Intraoperative head and neck<br>injury | Primary repair of injure d<br>organ/structure indicate d | Partial resection of injured<br>organ/structure in dicated | Complete resection or<br>reconstruction of injured<br>organ structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the head and neck during a s | urgical procedure. | | | |
| Intraoperative hemorrhage | - | | Posto perative ra diologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of uncontroll | ed bleeding during a surgical pr | roce dure. | | | |
| Intraoperative hepatobiliary<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ /structure indicated | Complete resection or<br>reconstruction of injured<br>organ structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the hepatic parenchyma and/ | or biliarytract during a surgical pro | cedure. | 51 <u>)</u> | 001 |
| Intraoperative musculoskeletal<br>injury | Primary repair of injured<br>organ/structure in dicate d | Partial resection of injured<br>organ istructure indicated | Complete resection or<br>reconstruction of injured<br>organ /structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | 1 22 | 6: 386 0: | 1 | | T |
| Intraoperative neurological<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ /structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the nervous system during a s | surgical procedure. | | | |
| Intraoperative ocular injury | Primary repair of injured<br>organ/structure in dicate d | Partial resection of injured<br>organ /structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the eye during a surgical proc | edure. | 2 4 4 4 TO SECOND STATE OF THE SECOND STATE OF | | |
| Intraoperative renal injury | Primary repair of injured<br>organ/structure in dicated | Partial resection of injured organ structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the kidney during a surgical p | rocedure. | 101 SVRVG | 965<br>51) | 101<br>501 |
| Intraoperative reproductive tractinjury | | Partial resection of injured organ Istructure indicated | Complete resection or reconstruction of injured organ/structure indicated; | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Injury, poisoning and procedural complications

36

CARTISTEM® 

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | - 5 |
| | the reproductive organs during a | All and the second second | | | |
| Intraoperative respiratory injury | Primary repair of injure d<br>organ/structure indicate d | Partial resection of injured<br>organ/structure indicated | Complete resection or reconstruction of injured organ /structure indicated; disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | o the respirator y system during a s | urgical procedure. | © Di | | 20 |
| Intraoperative skin injury | Primar y repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | othe skin during a surgical proced | ure. | | | |
| Intraoperative splenic injury | | Primary repair of injured<br>organ/structure in dicated | Resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | othe spleen during a surgical prod<br>T | 7.5 | 1 | | |
| Intraoperative urin ary injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ &tructure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | o the urinary system during a surg | ical procedure . | 1550 454 500 m | 10000 PO | PHIS 100 |
| Intraoperative venous injury | Primary repair of injure d<br>organ/structure indicate d | Partial resection of injured<br>organ/structure in dicated | Complete resection or<br>reconstruction of injured<br>organ /structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | o a vein during a surgical procedu | re, | 61 D.845 15<br>At | | 01 |
| Kidney anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage o | furine due to breakdown of a kidn | ey anastomosis (surgical connecti | on of two separate anatomic struc | tures). | ni |
| Large intestinal an astomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatio; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an anastomos | is (surgical connection of two sep: | arate anatomic structures) in the la | rge intestine. | 01 |
| Pancreatic anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a pancreatic a | nastomosis (surgical connection o | ftwo separate anatomic structure | s). | <u> </u> |
| Pharyngeal ana stomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatio; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | in dicate d | Death |
| Definition: A finding of leakage d | ue to breakdown of a pharyn geal :<br>T | anastomosis (surgical connection :<br>T | PRODUCT SECURITION SECRETARIES | es),<br>T | ni<br>Pomerano |
| Postoperative hemorrhage | Minimal bleeding identified on<br>olinical exam; intervention not<br>indicated | Moderate bleeding; radiologic,<br>endo scopic, or operative<br>intervention indicated | Transfusion indicated of >=2 units (10 co/kg for pediatrics) pRBCs beyond protocol specification; urgent radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A finding of bleeding | occurring after a surgical procedur | Prince technical accompany | Teg 02 20 1040 | T0 2022 72 101 | PS10 230 |
| Postoperative thoracic<br>procedure complication | • | Extubated within 24 - 72 hrs<br>postoperatively | Extubated >72 hrs<br>postoperatively, but before<br>tracheostomy indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A finding of a previous | ,<br>sly undocumented problem that oc | curs after a thora dic procedure . | 00 GE | 5.59 | or<br>or |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent a ter manual<br>reduction; local imitation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental<br>ADL | Severe symptoms; elective operative intervention indicated; limiting self-care ADL | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

CTCAE 4.0 - May 28, 2009 : hijkny, polsoning and proceds rail complications

CARTISTEM® 

| | injary | , poisoning and procedu | 0.00 | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| | on of the intestinal stoma (surgically | | | Market and the control of the contro | Departure |
| rolapse of urostomy | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Local care or maintenance;<br>minor revision indicated | Dysfunctional stoma; elective<br>operative intervention or major<br>stomal revision indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of displace | ment of the urostomy. | 102 | 61 VC | | 01 |
| Radiation recall reaction<br>(dermatologic) | Faint erythema or dry<br>desquarmation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | Death |
| Definition: A finding of acute sk | in in fammatory reaction caused by | drugs, especially chemotherapeut | ic agents, forweeks ormonths foll | owing radiotherapy. The in famma | tory read |
| s confined to the previously im | adiated skin and the symptoms disa | ppear after the removal of the pha | rmaceutical agent. | Incodes es | I see see |
| Rectal an astomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of a rectal anasto | omo sis (surgical connection of two | separate anatomic structures). | | |
| Seroma | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; simple aspiration indicated | Symptomatic, elective radiologic<br>or operative intervention<br>indicated | * | |
| Definition: A finding of tumor-lik | te collection of serum in the tissues. | To 20 200 20 | T-007 - 00000 - 00 | Ingovo yo | DEC 10 |
| Small intestinal anastomotic<br>eak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the si | mall bowel. | |
| Spermatic cord anastomotic<br>eak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of a spermatic co | ord ana stomosis (surgical connecti | on oftwo separate anatomic struc | tures). | |
| Spinal facture | analgesics indicated | prescription analgesics<br>indicated; limiting instrumental<br>ADL | Severe back pain;<br>hospitalization or intervention<br>indicated for pain control (e.g.,<br>vertebroplasty); limiting self care<br>ADL; disability | Life-threatening consequences;<br>symptoms associated with<br>neurovascular compromise | Death |
| | c injury to the spine in which the con | 5.3 | Tarana and a second | | Leon |
| Stenosis of gastrointestinal<br>storna | | Symptomatic; IV fluids indicated<br><24 hrs; manual dilatation at<br>bedside | Severely altered GI function;<br>tuble feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of narrowin | g of the gastrointestinal stoma (surg | gically created opening on the surt | ace ofthe body). | | |
| Stomal ulcer | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; elective<br>operative intervention indicated | • | |
| | ized by a circumscribed, in tammato | ory and necrotic erosive lesion on t | he jejunal mucosal surface close t | to the anastomosis site following a | Ę |
| ga stroentero storny pro ce dure. | Пр.<br>У противлитест и путуровным известники имеля и | iki<br>Manuputan menangan menangan sa | ati. Tenyappa saanja ya ommyoo oo a | | ni<br>Protesta |
| racheal hemorrhage | Minimal bleeding identified on<br>clinical or diagnostic exam;<br>intervention not indicated | Moderate bleeding; medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A finding of bleeding | from the trachea. | 1/21 | 6 B | ( | 94<br>0- |
| Fracheal obstruction | Partial asymptomatic<br>obstruction on examination<br>(e.g., visual, radiologic or<br>end oscopic) | Symptomatic (e.g., noisy airway breathing), no respiratory distress; medical intervention indicated (e.g., steroids); limiting instrumental ADL | Stridor; radiologic or endo scopic<br>intervention indicated (e.g.,<br>stent, laser); limiting self care<br>ADL | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |

CTCAE 4.0 - May 28, 2009 : Injury, polsoning and procedural complications

CARTISTEM® 

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1: | 2 | 3 | 4 | : |
| racheostomy site bleeding | Minimal bleeding identified on<br>clinical exam; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of blood lea | kage from the tracheo storny site. | | | • | |
| Jreteric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage ( | due to breakdown of a ureteral ana | stomosis (surgical connection of to | o separate anatomic structures). | | |
| Jrethral ana stomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | due to breakdown of a urethral ana<br>T | T.E. | | | E |
| Jrostomy leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | of contents from a urostomy. | | , | | |
| Jrostomy obstruction | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; dilation or<br>endo scopic repair or stent<br>placement indicated | Attered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences;<br>organ failure; urgent operative<br>intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | | And the control of the second | , | |
| Jrostomy site bleeding | Minimal bleeding identified on<br>olinical exam; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of bleeding | from the urostomy site. | 13 | | | li . |
| Jrostorny stenosis | - g of the opening of a urostomy. | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endo scopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Jterine anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage ( | due to breakdown of a uterine an a | l<br>tomosis (sumical connection oftw | 100 C 000000000000000000000000000000000 | Interest of | 1 |
| the rine perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disord er cha racteri | zed by a rupture in the uterine wall | | | | |
| /aginal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | due to breakdown of a vaginal ana: | 1.5 | | | |
| /as deferens anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage ( | due to breakdown of a vas de feren | s an astomosis (surgical connection | n oftwo separate anatomic structu | res). | |
| /ascular access complication | - | De vice dislodgement, blockage,<br>leak, or malposition; device<br>replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including<br>pulmonary embolism or life-<br>threatening thrombus | Death |

CTCAE 4.0 - May 28, 2009 : Injury, poleoning and procedual complications  $39\,$ 

CARTISTEM® 

| <u> </u> | nijui y | , poisoning and procedu | rai complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1. | 2 | 3 | 4 | 5 |
| Wenous injury | Asymptomatic diagnostic finding; intervention not indicated | Sympto matic (e.g.,<br>claudication); repair or revision<br>not indicated | Severe symptoms; limiting self<br>care ADL; repair or revision<br>indicated; disabling | Life-threatening consequences;<br>e vidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage t | o a vein. | | | | |
| Wound complication | Incisional separation of <=25 % of wound, no deeper than superficial fascia | Incisional separation >25% of<br>wound; local care indicated | Hemia without evidence of<br>strangulation; fascial<br>disruption/dehiscence; primary<br>wound closure or revision by<br>operative intervention indicated | Hernia with evidence of strangulation; major reconstruction fap, graiting, resection, or amputation indicated | Death |
| | ent of a new problem at the site of<br>T | Mariante de la companya del la companya de la compa | To the second second | | n<br>Dominia |
| Wound dehiscence | Incisional separation of <=25 % of wound, no deeper than superficial fascia | Incisional separation >25% of<br>wound with local care;<br>asymptomatic hernia or<br>symptomatic hernia without<br>evidence of strangulation | Fascial disruption or dehiscence without evisceration; primary wound closure or revision by operative intervention indicated | Life-threatening consequences;<br>symptomatic hemia with<br>evidence of strangulation;<br>fascial disruption with<br>evisceration; major<br>reconstruction fap, graiting,<br>resection, or amputation<br>indicated | Death |
| Constant makes | n of the approximated margins of a<br>T | (77.535 | Tarress and the same of the sa | ra- | ĺ |
| Wrist fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective<br>surgery indicated | | |
| Definition: A finding of traumatio | injury to the wrist joint in which the | continuity of a wrist bone is brok | en. | | ×. |
| Injury, poisoning and procedural<br>complications - Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Injury, poisoning and procedural complications 40

CARTISTEM® 

| | (5 | Investigations | š | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| ctivated partial thromboplastin<br>me prolonged | >1 - 1.5 x ULN | >1.5 - 2.5 X ULN | > 2.5 x ULN; hemorrhage | 5 | |
| | ry test result in which the partial th<br>) may occur in a variety of disease | | reater than the control value. As a related to treatment. | possible indicator of coag | ulopathy, a prolon |
| Manine aminotran sferase<br>norea se d | >ULN -3D x ULN | Asymptomatic with ALT >3.0 - 5.0 x ULN; >3 x ULN with the appearance of worsening of fatigue, nausea, vomiting, right upper quadrant pain or tendemess, fever, rash, or eosinophilia | >5.0 - 20.0 x ULN; >5 x ULN for<br>>2 weeks | >20.0 x ULN | - |
| Definition: A finding based on lat | oratory test results that indicate a | n increase in the level of alanine a | minotransferase (ALT or SGPT) in | the blood specimen. | 100 |
| Akaline phosphatase increased<br>Definition: A finding based on lal | >ULN - 2.5 x ULN<br>poratorytest results that indicate a | >2.5 - 5.0 x ULN<br>n in crease in the level of alkaline i | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Aspartate aminotransferase<br>increased | >ULN-30×ULN | Asymptomatic with AST >3.0 - 5.0 x ULN; >3 x ULN with the appearance of worsening of fatigue, nausea, vomiting, right upper quadrant pain or tendemess, fever, rash, or eosinophilia | >5.0 - 20.0 x ULN; >5 x ULN for<br>>2 weeks | >20.0 x ULN | ō |
| Definition: A finding based on lat | ooratory test results that indicate a | n in crease in the level of aspartate | aminotransferase (AST or SGOT | ) in a blood specimen. | |
| Blood antidiuretic hormone<br>abnormal | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | 8 | |
| Definition: A finding based on lat | ooratory test results that indicate a | bnormal levels of antidiuretic hom | none in the blood specimen. | | 30 |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN<br>in the blood. Excess bilirubin is as | > 10.0 x ULN | ŀ |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Ho spitalization indicated | | - |
| Definition: A finding based on lat | ooratory test results that indicate a | n decrease in levels of corticotrop | hin in a blood specimen. | | 100 mm |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | E . | - |
| Definition: A finding based on lat | ooratory test results that in dicate a | b normal levels of gonadotrophin h | ormone in a blood specimen. | | 200 |
| Blood prolactin abnormal | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicate d | Moderate symptoms; limiting<br>instrumental ADL | 28 | 2 | - |
| Definition: A finding based on lat | oratory test results that in dicate a | bnormal levels of prolactin hormor | ne in a blood specimen. | | 22/ |
| Carbon mon oxide diffusing<br>capacity decreased | 3 - 5 units below LLN; for follow-<br>up, a decrease of 3 - 5 units<br>(ml/sec/mm Hg) below the<br>baseline value | 6 - 8 units below LLN; for follow-<br>up, an asymptomatic decrease<br>of > 5 - 8 units (ml/sec/mm Hg)<br>below the baseline value | Asymptomatic decrease of >8 units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., > Grade 2 hypoxia or > Grade 2 or higher dyspnea) | | - |
| Definition: A finding based on lur | ng function test results that indicate | a decrease in the lung capacity | to absorb carbon monoxide. | , | 001 |
| Cardia o troponin linoreased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | | Levels consistent with<br>myocardial in farction as defined<br>by the manufacturer | | • |
| Definition: A laboratory test resul | t which indicates in creased levels | of cardiac tropon in I in a biologica | l specimen. | | (6)<br>(1) |
| Cardia o troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myo cardial infarction as defined<br>by the manufacturer | | Levels consistent with<br>myocardial infarction as defined<br>by the manufacturer | ii. | - |

CTCAE 4.0 - May 28, 2009 : Investigations

CARTISTEM® 

| | | Investigations | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| CD4 lympho cytes decrea sed | <lln -="" 0.5="" 500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | |
| | oratory test results that indicate ar<br>T | | | | 201 |
| Chole sterol high | >ULN - 300 mg/dL; >ULN - 7.75<br>mmol/L | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | 12.92 mmol/L | >500 mg/dL; >12.92 mmol/L | 1 |
| 20-4-01 | oratory test results that indicate hi | CONTRACTOR SUPPLIES SERVICES | FOR CHANGE STATE | D. 651.7 V.C. 7699 | _ |
| CPK increased<br>Definition : A finding based on lab | >ULN - 2.5 x ULN<br>oratory test results that indicate ar | >2.5 x ULN - 5 x ULN<br>n in crease in levels of creatine pho | >5 x ULN - 10 x ULN<br>osphokinase in a blood specimen. | > 10 x ULN | ŀ |
| Creatinine in creased | >1 - 1.5 x baseline ; >ULN - 1.5 | >1.5 - 3.0 x baseline; >1.5 - 3.0 | >3.0 baseline; > 3.0 - 6.0 x ULN | >8,0 x ULN | |
| | x ULN | x ULN | 9 | - Announcement | Į. |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of creatinine in a b | iological specimen . | | -001<br>-001 |
| Ejection fraction decreased | 5 | Resting ejection fraction (EF) 50<br>- 40%; 10 - 19% drop from<br>baseline | Resting ejection fraction (EF) 39<br>-20%; > 20% drop from<br>baseline | Resting ejection fraction (EF)<br><20% | 5.0 |
| Definition: The percentage comp<br>contraction. | uted when the amount of blood eje | ected during a ventricular contracti | on of the heart is compared to the | amount that was present prior to | the |
| Bectrocardiogram QT corrected<br>interval prolonged | QTc 450 - 480 ms | QTc 481 - 500 ms | QTc >= 501 ms on at least two<br>separate ECGs | QTc >= 50 1 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventrioular tachycardia or<br>sign s/symptoms of serious<br>arrhythmia | 2 |
| Definition: A finding of a cardiac | dysrhythmia characterized by an a | bnormally long corrected QT inter | val. | | 187<br>201 |
| Fibrin ogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 - 0.25 x LLN or 50 - <75 % decrease from baseline | <0.25 x LLN or 75 % decrease<br>from baseline or absolute value<br><50 mg/d L | |
| Definition: A finding based on lab | oratory test results that indicate ar | ı<br>n decrease in levels of fibrinogen i | n a blood specimen. | 1 180 | 101 |
| Forced expiratory volume<br>decreased | FEVI % (percentages of observed FEVI and FVC related to their respective predicted values) 99 - 70 % predicted | FEV1 60 - 69 % | 50 - 59% | <= 49 % | Ī |
| Definition: A finding based on tes | t results that in dicate a relative de | crease in the fraction of the forced | vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | 1 |
| | oratory test results that in dicate hi | | | | nma- |
| Growth hormone abnormal | ne transfer of a gamma glutamyl g<br>Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | arinino acid | s of water. | 2 |
| Definition: A finding based on lab | ,<br>oratory test results that in dicate al | :<br>onormal levels of growth hormone | in a biological specimen. | | 8 |
| Haptoglobin decreased | <lln< td=""><td></td><td></td><td>2</td><td>1</td></lln<> | | | 2 | 1 |
| Definition: A finding based on lab | ,<br>oratory test results that in dicate ar | n decrease in levels of haptoglobir | n in a blood specimen. | , | |
| Hernoglobin increased | Increase in >0 - 2 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | In crease in >2 - 4 gm/d Labove<br>ULN or above baseline if<br>baseline is above ULN | horease in >4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | 8 | ŧ |
| Definition: A finding based on lab | oratory test results that in dicate in | creased levels of hemoglobin in a | biological specimen. | | |
| NR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5<br>times above baseline if on<br>antico agulation | >2.5 x ULN; >2.5 times above<br>baseline if on anticoagulation | - | |
| Definition: A finding based on lab | oratory test results that in dicate ar | n increase in the ratio of the patier | nt's prothrombin time to a control s | ample in the blood. | |
| ipase in creased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | |
| Definition: A finding based on lab | ,<br>oratory test results that in dicate ar | n increase in the level of lipase in | a biological specimen. | | (S) |
| ymphocyte count decreased | <lln -="" -<br="" .8="" 0="" 800="" <lln="" mm3;="" x="">10e9 /L</lln> | <800 - 500 /mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200 mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10 e9 /L | 2 |
| Definition: A finding based on lab | oratory test results that in dicate a | decrease in number of lymphocyt | es in a blood specimen. | | -001 |
| Lymphocyte count increased | | >4000/mm3 - 20,000/mm3 | >20000/mm3 | | 1. |

CTCAE 4.0 - May 28, 2009 : Investigations 42

CARTISTEM® 

| | X. | Investigations | : | | |
|---|---|---|---|---|---|
| Adverse Event | | | Grade | | |
| | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding based on lab | oratory test results that indicate ar | abnormal increase in the numbe | roflymphocytes in the blood, effu | sions or bone marrow. | X. |
| Neutrophil count decreased | 10e9 /L | <1500 - 1000/mm3 ; <1.5 - 1.0 x<br>10e9 /L | 10e9 /L | <500 /mm3; <0.5 x 10e9 /L | |
| 1 10 10 10 | oratory test results that indicate a | decrease in number of neutrophil:<br>I | F81 " 2: 1/1227 " W | | ř |
| Pancreatic enz ymes decreased | <lln a="" and="" p="" symptomatic<=""></lln> | horease in stool frequency,<br>bulk, or odor; steatorrhea | Sequelae of absorption deficiency | | t e |
| Definition: A finding based on lab | oratory test results that indicate ar | de crease in levels of pancreatio | enzymes in a biological specimen | | |
| Platelet count decreased | <lln -="" -<br="" 75,000.mm3;="" <lln="">75.0 x 10e9 /L</lln> | <75,000 - 50,000/mm3; <75.0 -<br>50.0 x 10e9 /L | <50 000 - 25,000 /mm3; <50.0 -<br>25.0 x 10e9 /L | <25,000 /mm3; <25.0 x 10e9 /L | |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | 98<br> |
| Serum armylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5 D x ULN | >5.0 x ULN | ž |
| Definition: A finding based on lab | oratory test results that indicate ar | n increase in the levels of amylase | in a serum specimen. | r underendation : | 8: |
| Urine output decreased | | | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | |
| | rt results that in dicate urin e produc<br>T | | Í | | E |
| vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value;<br>limiting instrumental ADL | <50% of predicted value;<br>limiting self care ADL | | |
| Definition: A finding based on pu<br>value. | Imonary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | um inhalation) when compared to | the predicte |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >= 20 % from baseline | | į. |
| Definition: A finding characterize | d by an increase in overall body w | eight; for pediatrics, greater than t | he baseline growth ourve. | , | |
| Weight loss | 5 to < 10 % from baseline;<br>intervention not indicated | 10 - <20% from baseline;<br>nutritional support indicated | >= 20 % from baseline; tube<br>feeding or TPN indicated | | |
| Definition: A finding characterize | d by a decrease in overall body we | ight; for pediatrics, less than the b | paseline growth curve. | | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <3000 - 2000/mm3; <3.0 - 2.0 x<br>10e9 /L | <2000 - 1000/mm3; <2.0 - 1.0 x:<br>10e9 /L | <1000.mm3; <1.0 x 10e9 /L | |
| Definition: A finding based on lab | ।<br>oratory test results that in dicate ar | i<br>n decrease in number of white blo | od cells in a blood specimen. | | h |
| Investigations - Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or me dically significant<br>but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization in dicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Investigations 43

CARTISTEM® 

| | * | Metabolism and nutrition | n alsoraers | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | -2 | 3 | 4 | 5 |
| Acido sis | pH <normal, but="">7.3</normal,> | | pH <7.3 | Life-threatening consequences | Death |
| Definition: A disorder charact | terized by abnormally high acidity (high | hydrogen-ion concentration) of t | he blood and other body tissues. | | 2 |
| Alcohol into lerance | | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact<br>vorniting, indigestion and hea | terized by an increase in sensitivity to to<br>adaches. | the adverse effects of alcohol, wh | ich can include nasal congestion, | skin fushes, heart dysrhythmias, i | nausea, |
| Alkalosis | pH >normal, but <=7.5 | - | pH > 7.5 | Life-threatening consequences | Death |
| Definition: A disorder charact | terized by abnormally high alkalinity (lo | ow hydrogen-ion concentration) of | fthe blood and other body tissues | | 25) |
| An orexia | Loss of appetite without alteration in eating habits | Oral intake altered without<br>significant weight loss or<br>malnutrition; oral nutritional<br>supplements in dicated | Associated with significant weight loss or malnutrition (e.g., inade quate oral caloric and/or fuid intake); tube feeding or TPN indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by a loss of appetite. | 02 | ************************************** | 2 | |
| Dehydration | Increased oral fuids indicated;<br>dry mucous membranes;<br>diminished skin turgor | M fluids indicated <24 hrs | M fluids or hospitalization indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by excessive loss of water from | the body. It is usually caused by | severe diarrheal, vomiting or diap | horesis. | 37 |
| Gluco se intolerance | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an inability to properly metal | bolize glucose. | regional personal assemble ass | Torrena orangona masa | Toward and |
| Hypercalcemia | >ULN - 115 mg/dL; >ULN - 2.9<br>mmol/L; lonized calcium >ULN<br>- 15 mmol/L | >11.5 - 12.5 mg/dL; >2.9 - 3.1<br>mmol/L; lonized calcium >1.5 -<br>1.6 mmol/L; symptomatic | >12.5 - 13.5 mg/dL ;>3.1 - 3.4<br>mmol/L; lonized calcium >1.6 -<br>1.8 mmol/L; hospitalization<br>indicated | >13.5 mg/dL; >3.4 mmol/L;<br>lonized calcium >1.8 mmol/L;<br>life-threatening consequences | Death |
| Definition: A disorder charact | terized by laboratory test results that in | ndicate an elevation in the concer | tration of calcium in blood. | | |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8.9 mmol/L | Fasting glucose value >160 -<br>250 mg/dL; Fasting glucose<br>value >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-<br>thre attening consequences | Death |
| Definition: A disorder charact<br>intolerance. | terized by laboratory test results that in | ndicate an elevation in the concern | tration of blood sugar. It is usually | an indication of diabetes mellitus | or glucos |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charact<br>the use of diuretic drugs. | terized by laboratory test results that in | ndicate an elevation in the concern | tration of potassium in the blood; | associated with kidney failure or so | ometimes |
| Hypermagne se mia | >ULN - 3 D mg/dL; >ULN - 123<br>mmol/L | | >3.0 - 8.0 mg/dL; >1.23 - 3,30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charact | terized by laboratory test results that in | dicate an elevation in the concer | tration of magnesium in the blood | | |
| Hypematremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| 240 (M22) 2440 27 | terized by laboratory test results that in | PARTIES SENSO SENSO SENSO SENSOR | TORREST VENUE PROPERTY DIVING TORREST | Transaction to contract the | 0.000.00 |
| Hypertriglyœridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42mmol/L | >300 mg/dL - 500 mg/dL; >3.42<br>mmoI/L- 5.7 mmoI/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4mmol/L | > 1000 mg/dL; > 11.4 mmol/L;<br>life-threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate an elevation in the concern | tration of triglyceride concentratio | n in the blood. | |
| Hyperuricemia | >ULN - 10 mg/dL; <=0.59<br>mmol/L without physiologic<br>consequences | • | >ULN - 10 mg/dL; <=0.59<br>mmol/L with physiologic<br>consequences | > 10 mg/d L; >0.59 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate an elevation in the concen | tration of uric acid. | | |
| Hypoalbumin emia | <lln -="" 3="" 30="" dl;<lln="" g="" l<="" td=""><td>&lt;3 - 2 g /dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences;<br/>urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g /dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | erized by laboratory test results that in | 15 | | | |
| Hypocalcemia | <lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln<br>- 1.0 mmol/L</lln<br></lln> | <8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | <7.0 - 6.0 mg/d L; <1.75 - 1.5<br>mmol/L; lonized calcium <0.9 -<br>0.8 mmol/L; hospitalization<br>indicated | <6.0 mg/dL; <1.5 mmol/L;<br>lonized calcium <0.8 mmol/L;<br>life-threatening consequences | Death |

CTCAE 4.0 - May 28, 2009: Metabolism and nutrition disorders

CARTISTEM® 

| | - N | Metabolism and nutrition | on disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate a low concentration of ca | licium in the blood. | 9 | 000 |
| Hypoglycemia | <lln -="" 3.0<br="" 55="" <lln="" dl;="" mg="">mmol/L</lln> | | <40 - 30 mg/d L; <2.2 - 1.7<br>mmol /L | <30 mg/dL; <1.7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| | erized by laboratory test results that in | Zerovicznosta czasta wystaki w w w w w w w w w w w w w w w w w w w | | | Lange |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-thre atening consequences</td><td>Death</td></lln> | <lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-thre atening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate a low concentration of po | tassium in the blood. | 9 | 00:<br>00: |
| Hypomagne semia | <lln -="" 0.5<br="" 1.2="" <lln="" dl;="" mg="">mmol/L</lln> | <1.2 - 0.9 mg/dL ;<0.5 - 0.4<br>mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L | <0.7 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate a low concentration of m | agnesium in the blood. | | |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt; 120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | - | <130 - 120 mmol/L | < 120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate a low concentration of so | dium in the blood. | | |
| Hypopho sphatemia | <lln -="" 0.8<br="" 2.5="" <lln="" dl;="" mg="">mmol/L</lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6<br>mmol/L | <2.0 - 1.0 mg/dL; <0.6 - 0.3<br>mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | Idicate a low concentration of ph | osphantes in the blood. | | Ä |
| Iron overload | 1 | Moderate symptoms;<br>intervention not indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | erized by accumulation of iron in the ti | issues. | 85 B | 5 Mg | (E) |
| Ob esity | | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.99 kg/m2, or 1 or 2<br>decimals should be used<br>consistently over both grades | BMI >= 40 kg/m2 | |
| Definition: A disorder charact | erized by having a high amount of boo | lyfat. | | <i>5</i> | 75<br>20 |
| Tumor lysis syndrome | # <b>5</b> 00 | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | erized by metabolic abnormalities that | result from a spontaneous or th | erap y-related cytolysis of tumor cel | ls. | |
| Metabolism and nutrition<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization in dicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Metabolism and nutrition disorders 45

CARTISTEM® 

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | |
| Abdominal so <b>t</b> tissue necrosis | | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri: | zed by a necrotic process occurrin | g in the soft tissues of the abdomir | nal wall. | | |
| Arthralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | E . | - |
| | zed by a sensation of marked disc<br>T | [S | T | T <sub>n</sub> | T |
| Arthritis | Mild pain with inflammation,<br>erythema, or joint swelling | Moderate pain associated with<br>signs of inflammation ,<br>erythema, or joint swelling;<br>limiting instrumental ADL | Severe pain associated with<br>signs of infarrmation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling; limiting self care ADL | | |
| Definition: A disorder characteria | zed by inflammation involving a joi | nt. | To a meno w | Transmit and | Townson |
| Awascular necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL, elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | | ne tissue due to interruption of bloo | od supply. Most often affecting the | epiphysis of the long bones, the r | ecrotic |
| changes result in the collapse al<br>Back pain | nd the destruction of the bone stru<br>Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | 3 | 5 |
| Definition: A disorder characteri: | l<br>zed by marked discomfort sensatio | | 1702 | J | E |
| Bone pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | PK | 1. |
| | | instrumental ADL | ADL | | |
| | zed by marked discomfort sensatio | 1/2. | I | | 1 |
| Buttock pain | Mild pain | Moderate pain ; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | j* | ľ |
| Definition: A disorder characteri: | zed by marked discomfort sensatio | on in the buttocks. | 7 | | T |
| Chest wall pain | Mild pain | Moderate pain ; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 8 | ŀ |
| Definition: A disorder characteri: | zed by marked discomfort sensatio | on in the chest wall region. | ¥ | | - |
| Exostosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL, elective operative<br>intervention indicated | ž. | 5 |
| Definition: A disorder characteri: | zed by non-neoplastic overgrowth | ofbone. | <u> </u> | | - |
| Fibrosis deep connective tissue | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to slide or pinch skin; limiting joint or orifice movement (e.g., mouth, anus); limiting self care ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characteria | ed by fibrotic degeneration of the | deep connective tissues. | | | |
| Flank pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 8 | ŀ |
| Definition: A disorder characteria | ed by marked discomfort sensation | on on the lateral side of the body in | the region below the ribs and abo | ove the hip. | (6)<br>(1) |
| Generalized muscle weakne <i>s</i> s | Symptomatic; weakness<br>perceived by patient but not<br>evident on physical exam | Symptomatic; weakness evident<br>on physical exam; weakness<br>limiting in strumental ADL | Weakness limiting self care<br>ADL; disabling | | |
| Definition: A disorder characteria | ed by a reduction in the strength ( | of muscles in multiple an atomic site | es. | \$ | (8) |
| Growth suppression | Reduction in growth velocity by<br>10 - 29 % ideally measured over<br>the period of a year | Reduction in growth velocity by<br>30-49 % ideally measured over<br>the period of a year or 0 - 49 %<br>reduction in growth from the | Reduction in growth velocity of<br>>=50% ideally measured over<br>the period of a year | | - |

CTCAE 4.0 – May 28, 2009 : Missor bakeletal and connective that eldisorders

CARTISTEM® 

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Head soft tissue necrosis | | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by a necrotic process occurring | in the soft tissues of the head. | | | |
| Joint effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated; disabling | 8 | |
| | zed by excessive fluid in a joint, uso | T <sub>=</sub> | 1 31 | | T |
| Joint range of motion decreased | d <= 25 % loss of ROM (range of<br>motion); decreased ROM<br>limiting athletic activity | >25 - 50% decrease in ROM;<br>limiting instrumental ADL | >50 % decrease in ROM; limiting self care ADL; disabling | is . | |
| Definition: A disorder characteria | zed by a decrease in joint flexibility | ofanyjoint. | | • | |
| Joint range of motion decreased<br>cervical spine | | Rotation <60 degrees to right or | Ankylosed/fused over multiple<br>segments with no C-spine<br>rotation | | |
| Definition: A disorder characteria | zed by a decrease in flexibility of a | cervical spine joint: | | | |
| Joint range ofmotion decreased<br>umbar spine | the foorto pick up a very light<br>object but able to do athletic<br>activity | Pain with range of motion<br>(ROM) in lumb ar spine; requires<br>a reaching aid to pick up a very<br>light object from the floor | <50% lumbar spine flexion;<br>associated with symptoms of<br>ankylosis or fused over multiple<br>segments with no L-spine<br>flexion (e.g., unable to reach to<br>floorto pick up a very light<br>object) | -2 | • |
| | zed by a decrease in flexibility of a | 7.5 | | | T |
| Kypho sis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative<br>intervention indicated; limiting<br>self care ADL | | - |
| Definition: A disord er characteria | zed by an abnormal increase in the | curvature of the thoracic portion of | ofthe spine. | | |
| Lordosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | £ | - |
| Definition: A disorder characteria | zed by an abnormal increase in the | our vature of the lumbar portion of | fthe spine. | | |
| Muscle weakness lett-sided | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL; disabling | | G<br>F |
| Definition: A disorder characteria | zed by a reduction in the strength o | f the muscles on the left side of th | e body. | | |
| Musde weakness lowerlimb | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL; disabling | ea . | - |
| Definition: A disorder characteria | zed by a reduction in the strength o | f the lower limb musdes. | | | |
| vlus de weakness right-sided | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL; disabling | | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the right side of t | he body. | | |
| vfus de weakness trunk | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL; disabling | | + |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the trunk muscles. | | | |
| Muside weakness upper limb | Symptomatic; perceived by | Symptomatic; evident on | Limiting self care ADL; disabling | ® | - |

CTCAE 4.0 - May 28, 2009 : Misson bake leital and connective its see disorders

CARTISTEM® 

| 5 | Muscu | loskeletal and connectiv | re tissue disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Musculoske letal de formity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis (e.g.,<br>shoe insert) or covered by<br>clothing | Significant deformity,<br>hypoplasia, or a symmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>dothing; disabling | | |
| Definition: A disorder characte | rized by of a malformation of the mu: | sculoskeletal system. | D9 8///ASI38 D639 | T | |
| Myalgia | Mild pain | Moderate pain ; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 5 | ÷ |
| Definition: A disord er characte | rized by marked discomfort sensatio | n originating from a muscle or gro | up of muscles. | | |
| Ayositis | Mild pain | Moderate pain associated with<br>weakness; pain limiting<br>instrumental ADL | Pain associated with severe<br>weakness; limiting selfcare<br>ADL | ē | ÷ |
| Definition: A disorder characte | rized by inflammation involving the s | keletal musdes. | | | |
| Neck pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | |
| Definition: A disorder characte | rized by marked discomfort sensatio | n in the neck area. | 1 | | |
| Neck soft tissue necrosis | • | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings ortopical<br>medications) | Operative debridement or other<br>invasive intervention indicated<br>(e.g. tissue reconstruction, flap<br>or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | in the soft tissues of the neck. | - | | |
| Osteone crosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., to pical a gents); limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | in the bone of the mandible. | T24 32 0002 7234 | T | |
| Osteoporosis | Radiologic evidence of<br>osteoporosis or Bone Mineral<br>Density (BMD)t-score - 1 to -2.5<br>(osteopenia); no loss of height<br>or intervention indicated | BMD t-score <-2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >= 2 cm;<br>hospitalization indicated; limiting<br>self care ADL | | |
| Definition: A disorder characte<br>composition), resulting in incre | rized by reduced bone mass, with a | decrease in cortical thickness and | d in the number and size of the trail | peculae of cancellous bone (but no | omal cher |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | in the second | - |
| Definition: A disorder characte | rized by marked discomfort sensatio | n in the upper or lower extremities | 5. | ř. | 200 |
| Pelvic so <b>t</b> tissue necrosis | | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, tap or grafting) | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | in the soft tissues of the pelvis. | T | | r |
| Scolio sis | <20 degree s; clinically und ete ctable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward fexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | | <u>.</u> |
| Definition: A disorder characte | rized by a malformed, lateral curvatu | re of the spine. | | Toronto est | |
| So <b>t</b> tissue necrosis lower limb | i sed | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings ortopical<br>medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, tap or grafting) | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | in the soft tissues of the lower ex | dremity. | | (A) |
| So <b>1</b> tissue necrosis upper limb | ). · | Local wound care; medical intervention indicated (e.g., dressings ortopical medications) | Operative debridement or other invasive intervention indicated (e.g. ti ssue reconstruction, tap or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Muscu bakeletal and connective than eldisorders

CARTISTEM® 

| 2 | Muscu | loskeletal and connectiv | e ussue uisuruers | | |
|---|---|---|---|---|---|
| Adverse Event | Grade | | | | |
| | 1. | 2 | 3 | 4 | - 5 |
| Superficial soft tissue fibrosis | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicularto skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characteriz | ed by fibrotic degeneration of the s | superficial soft tissues. | | | |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring small bites, so t foods or purees | Decreased ROM with inability to<br>adequately aliment or hydrate<br>orally | | 10 |
| Definition: A disorder characteriz | ,<br>ed by lack of ability to open the mo | outh fully due to a decrease in the | range of motion of the muscles of | ma stication. | |
| Unequal limb length | Mild length discrepancy < 2 cm | Moderate length discrepancy 2 -<br>5 cm; shoe lift indicated; limiting<br>instrumental ADL | Severe length discrepancy > 5<br>cm; limiting self-care ADL;<br>disabling; operative intervention<br>indicated | | T. |
| Definition: A disorder characteriz | ed by of a discrepancy between th | e lengths ofthe lowerorupper ex | tremities. | | - T |
| Musculoskeletal and connective<br>tissue disorder - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Musculoskeletal and connective tissue disorders 49 CTCAE 4.0 - May 28, 2009 : Neoplasms benign, malignant and unspecified (incl cysts and polyps) 50

CARTISTEM® 

| | Neoplasms benig | ın, malignantand unspe | ecified (incl cysts and poly | /ps) | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 23 |
| Leukemia secondaryto<br>on cology chemotherapy | - | | | Present | Death |
| Definition: A disorder characteri: | zed by leukemia arising as a result | of the mutagenic effect of chemo | otherap y agents. | | |
| Myelodysplastic syndrome | 1 E2. | • | ************************************** | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by insufficiently he alth y hemata | spoietic cell production by the bo | пе татош. | | A: |
| Treatment related secondary<br>malignancy | | | Non life-threatening secondary<br>malignancy | Acute life-threatening secondary<br>malignancy; blast crisis in<br>leukemia | Death |
| Definition: A disorder characteria | ,<br>zed by development of a malignand | ,<br>cymost probably as a result oftr | eatment for a previously existing ma | alignancy. | te: |
| Tumor pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain ; limiting self care<br>ADL | 2 | ō |
| Definition: A disorder characteria | zed by marked discomfort from a n | eoplasm that may be pressing or | n a nierve, blocking blood vessels, ir | nflamed or fractured from metastas | is. |
| Neoplasms benign, malignant<br>and unspecified (incloysts and<br>polyps) - Other, specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically signi ficant<br>but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CARTISTEM® 

| | 30 | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | |
| b ducens nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | | - |
| | rized by involvement of the abducen | 15 | | 10 | |
| Accessory nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | |
| Definition: A disorder character | rized by involvement of the accessor | ry nerve (eleventh cranial nerve). | Y <sub>1</sub> | | (4) |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | | - |
| Definition: A disorder character | rized by involvement of the acoustic | nerve (eighth cranial nerve ). | T | | |
| 4kathisia | Mild restlessness or increased<br>motor activity | Moderate restlessness or<br>increased motor activity; limiting<br>instrumental ADL | Severe restlessness or<br>increased motor activity; limiting<br>self care ADL | | - |
| Definition: A disorder character | rized by an uncomfortable feeling of | inner restlessness and inability to | stay still; this is a side effect of so | me psychotropic drugs. | (1) |
| Amne sia | Mild; transient memory loss | Moderate; short term memory loss; limiting instrumental ADL | Severe; long term memory loss;<br>limiting self care ADL | | - |
| Jefinition: A disorder character | rized by systematic and extensive lo | ss of memory. | A: | | ř |
| iphonia P | ŀ | | Voicelessness; unable to speak | 8 | |
| Definition: A disord er character | rized by the inability to speak. It may | result from injuries to the vocal co | ords or may be functional (psycho | genic). | |
| rach noiditis | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | rized by inflammation of the arachno | oid membrane and adjacent subar:<br>T | achnoid space. | | |
| *taxia | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL; mechanical assistance indicated | | |
| Definition: A disorder character | rized by lack of coordination of musc | de movements resulting in the imp | airment or in ability to perform volu | intary activities. | 8) |
| Brachial plexopathy | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | (A) | - |
| Definition: A disorder character | ,<br>rized by regional paresthesia of the l | '<br>brachial plexus, marked discomfor | '<br>t and muscle weakness, and limite | '<br>ed movement in the arm or hand. | 8 |
| Central nervous system | Asymptomatic; clinical or | Moderate symptoms; | Severe symptoms; medical | Life-threatening consequences; | Death |
| earosis | diagnostic observations only;<br>intervention not indicated | corticosteroids indicated | intervention indicated | urgent intervention indicated | Death |
| Definition: A disord er character | rized by a necrotic process occurring | in the brain and/or spinal cord. | - N | | 01 |
| Cerebrospinal 1 uid leakage | Post-craniotomy:<br>asymptomatic; Post-lumbar<br>puncture: transient headache;<br>postural care indicated | Post-craniotomy: moderate<br>symptoms; medical intervention<br>indicated; Post- lumbar<br>puncture: persistent moderate<br>symptoms; blood patch<br>indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| Definition: A disorder character | rized by loss of cerebrospinal fluid in | nto the surrounding tissues. | | | ~· |
| Cognitive disturbance | Mild cognitive disability; not<br>interfering with work/school.life<br>performance; specialized<br>educational services/devices<br>not indicated | Moderate cognitive disability;<br>interfering with work/school/life<br>performance but capable of<br>independent living; specialized<br>resources on part time basis<br>indicated | Severe cognitive disability;<br>significant impairment of<br>work/school/life performance | | |
| Definition: A disorder character | rized by a conspicuous change in co | ognitive function. | 25 | | 80 |
| Concentration impairment | Mild inattention or decreased<br>level of concentration | Moderate impairment in<br>attention or decrea sed leivel of<br>concentration; limiting<br>instrumental ADL | Severe impairment in attention<br>or decreased level of<br>concentration; limiting self care<br>ADL | 8 | ÷ |

CTCAE 4.0 - May 28, 2009 : Ne mois system disorders

CARTISTEM® 
| 3 | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | |
| Depressed level of<br>consciousness | Decreased level of alertness | Sedation; slow response to<br>stimuli; limiting instrumental<br>ADL | Difficult to arouse | Life-threatening consequences | Death |
| | erized by a decrease in ability to pero | 18 | 1 | | i - |
| Dizziness | Mild unsteadiness or sensation<br>of movement | Moderate unsteadiness or<br>sensation of movement; limiting<br>instrumental ADL | Severe unsteadiness or<br>sensation of movement; limiting<br>self care ADL | - | - |
| Definition: A disorder charact | erized by a disturbing sensation of ligh | hthead edness , unsteadiness , gid d | iness, spinning or rocking. | i | 5 |
| Dysarthria | Mild slurred speech serized by slow and slurred speech res | Moderate impairment of articulation or sturred speech | Severe impairment of articulation or slurred speech | | - |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | r | |
| Definition: A disorder charact | erized by distortion of sensory percep | tion , resulting in an abnormal and | unpleasant sensation. | , | |
| Dysgeusia | Attered taste but no change in diet | Attered taste with change in diet<br>(e.g., oral supplements);<br>noxious or unpleasant taste;<br>loss oftaste | - | | ÷ |
| Definition: A disorder charact | erized by abnormal sensual experience | ·<br>ce with the taste of food stuffs ; it ca | n be related to a decrease in the : | sense of smell. | 101 |
| Dysph asia | Awareness of receptive or<br>expressive characteristics; not<br>impairing ability to communicate | Moderate receptive or<br>expressive characteristics;<br>impairing ability to communicate<br>spontaneously | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly | | |
| Definition: A disorder charact | erized by impairment of verbal comm | unication skills, often resulting from | n brain damage . | | (10)<br>(1) |
| Edema cerebral | | | | Life-threatening consequences;<br>urgent intervention indicated | 2 |
| Definition: A disorder charact | erized by swelling due to an excessiv | e accumulation of fluid in the brain<br>T | ig<br>Personal managan mengenasa salah sebagai | | Terressor |
| En œphalopath y | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| 125 37.5557337 37 | erized by a pathologic process involvi | 2.5550 SX XX | 18 6 N | 3836 G | 222 30 |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary<br>movements; limiting<br>instrumental ADL | Severe involuntary movements<br>or torticollis; limiting self care<br>ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by abnormal, repetitive, involur | itary muscle movements, frenzied | speech and extreme restlessnes: | | |
| Facial mu <i>s</i> cle weakness | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | | <del>1</del> |
| Definition: A disorder charact | erized by a reduction in the strength o | f the facial muscles. | Tax 220025 921 | T | |
| Facial nerve disorder | Asymptomatic; dinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | 8 | |
| Definition: A disorder charact | erized by involvement of the facial ne | rve (seventh cranial nerve). | 1000 popular | 0000 | |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; dinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by involvement of the glossoph | aryn geal nerve (ninth cranial nerv | e). | , | <i>x</i> : |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | ŧ |
| Definition : A disorder charact | erized by a sensation of marked disco | mfort in various parts of the head | , not confined to the area of distrib | ution of any nerve. | |
| Hydrocephalus | Asymptomatic; dinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms;<br>intervention not indicated | Severe symptoms or<br>neurological deficit; intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal increase of cer | e brospinal fluid in the ventricles o | fthe brain. | | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for sleep | Severe increased need for sleep | D | - |

CTCAE 4.0 - May 28, 2009 : Ne moits system disorders

CARTISTEM® 

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | |
| Hypoglossal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | 8 | |
| | rized by involvement of the hypoglos | (S | I | X 44/0 X 70/00/00 1 A 20/00/00/00 1 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | L |
| intracranial hemorrhage | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical<br>intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the cranium. | | | | |
| schemia cerebrovascular | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms | • | | |
| Definition: A disorder characte<br>damage. | rized by a decrease or absence of b | lood supplyto the brain caused by | obstruction (thrombosis or embol | ism) of an artery resulting in neuro | logical |
| l'vth nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | | <del>.</del> |
| Definition: A disorder characte | rized by involvement of the trochlear | nerve (fourth cranial nerve). | 1 | T | |
| Lethargy | Mild symptoms; reduced<br>alertness and awareness | Moderate symptoms; limiting instrumental ADL | *** | * | ŧ |
| Definition: A disorder characte | rized by a decrease in consciousnes | ss chara cterized by mental and ph | ysical inertness. | 1 | |
| Le uko encephal opathy | Asymptomatic; small focal<br>T2/FLAIR hyperintensities;<br>involving periventricular white<br>matter or <1.8 of susceptible<br>areas of cerebrum +4 mild<br>increase in subarachnoid space<br>(SAS) and/or mild<br>ventriculomegaly | Moderate symptoms; focal T2/FLAIR hyperintensities, involving periventricular white matter extending into centrum semiovale or involving 1/8 to 2/8 of susceptible areas of cerebrum +/- moderate increase in SAS and/or moderate ventriculomegaly | Severe symptoms; extensive<br>T2/FLAIR hyperintensities,<br>involving periventricular white<br>matter involving 2/3 or more of<br>susceptible areas of cerebrum<br>+/- moderate to severe increase<br>in SAS and/or moderate to<br>severe ventriculomegaly | Life-threatening consequences; extensive T2/FLAIR In yperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Death |
| Definition: A disorder characte | rized by diffuse reactive astrocytosis | with multiple areas of necrotic for | i without inflammation. | | 001 |
| Memory impairment | Mild memory impairment | Moderate memory impairment;<br>limiting instrumental ADL | Severe memory impairment;<br>limiting selfcare ADL | 2 | |
| Definition: A disorder characte | rized by a deterioration in memory for | unction. | T257 Y560-0C 5011 | (a.2070 yo | 120 00 |
| denin gismus | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by neck stiffness, headache, a | nd photophobia resulting from irrit: | ation of the cerebral meninges. | | |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | - |
| Definition: A disorder characte | rized by uncontrolled and purposele | ss movements. | W En | ı. | |
| Myelitis | Asymptomatic; mild signs (e.g.,<br>Babinski's reflex or Lhermitte's<br>sign) | Moderate weakness or sensory<br>loss; limiting instrumental ADL | Severe weakness or sensory<br>loss; limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation involving the s | pinal cord. Symptoms include wea | kness, paresthesia, sensory loss, | marked discomfort and incontiner | nce. |
| Neuralgia | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 30 | 2 |
| Definition: A disorder characte | rized by intense painful sensation al | ong a nerve or group of nerves. | Other Company of the | I | T. |
| Vystagmus | | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | T. | |
| Definition: A disorder characte | rized by involuntary movements of the | he eyeballs. | T-000 90Matrices (Matrice) | T | |
| Oculomotor nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | | |
| Definition: A disorder characte | rized by involvement of the oculomo | tor nerve (third cranial nerve). | | | |
| Olfactory nerve disorder | 184 | Moderate symptoms; limiting | Severe symptoms; limiting self | 8 | ŧ |

CTCAE 4.0 - May 28, 2009 : Ne moits system disorders

CARTISTEM® 

| 9 | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | -2 | 3 | 4 | 5 |
| Paresthe sia | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | ٥ | - |
| Definition: A disorder characteriz<br>are experienced in the absence ( | | ensory neurons resulting in abnor | mal cutaneous sensations of tingli | ng, numbness, pressure, cold, and | warmth that |
| Peripheral motor neuropathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; assistive device<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation or degeneratio | n of the peripheral motor nerves. | to to | t ( | 01 |
| Peripheral sensory neuro pathy | Asymptomatic; loss of deep<br>tendon reflexes or paresthesia | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| [22] (12] (12] (12] (13] (13] (13] (13] (13] (13] (13] (13 | ed by inflammation or degeneratio<br>1 | DESCRIPTION OF STREET | | | - 8 |
| Phantom pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | |
| Definition: A disorder characteriz | ed by marked discomfort related to<br>T | o a limb or an organ that is remove<br>T | ed from or is not physically part of<br>T | the body. | 98 |
| Presyncope | - | Present (e.g., near fainting) | - | je. | - |
| Definition: A disorder characteriz | ed by an episode oflightheadedne<br>T | ess and dizziness which may prec<br>T | ede an episo de of syncope. | | ř |
| Pyramidal tract syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| 47 100 100 1000 100000 NAS-2000000000 | ed by dysfunction of the corticospi<br>nd a decrease in fine motor coord | | ord. Symptoms include an incre | ease in the musde tone in the lowe | er extremities, |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL; medical<br>intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>connecting nerve root. | ed by inflammation involving a ner | ve root. Patients experience mark | ed discomfort radiating along a ne | erve path because of spinal pressu | re on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by paralysis of the recurrent lar | yngeal nerve. | | | - 5 |
| Reversible posterior<br>leukoencephalopathy syndrome | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; abnormal imaging studies; limiting instrumental ADL | Severe symptoms; very<br>abnormal imaging studies;<br>limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | 19 (14 PH) HING SANDERS (17 PH) HING SANDERS | | | ,<br>findings of posterior leukoencephal<br>s an acute or subacute reversible ( | |
| Seizure | Briefpartial seizure; no loss of consciousness | Brief generalized seizure | Multiple seizures despite<br>medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characteriz | ed by a sudden, in voluntary skelet | al muscular contractions of cereb | ral or brain stem origin. | | - 50 |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting selfcare<br>ADL | 2 | ŧ |
| Definition: A disorder characteriz | ed by marked discomfort in the fac | e, between the eyes, or uppertee | eth originating from the sinuses. | | |
| Somn olence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stup or | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by characterized by excessive: | sleepiness and drowsiness. | 9/ ti | | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle<br>tone and increase in resistance<br>through range ofmotion | Severe increase in muscle tone<br>and increase in resistance<br>through range of motion | Life-threatening; unable to move<br>active or passive range of<br>motion | Death |
| Definition: A disorder characteriz<br>disturbances. | ed by increased involuntary muscl | e tone that affects the regions inte | riering with voluntary movement. | t results in gait, movement, and s | peech |
| Stroke | Asymptomatic or mild<br>neurologic deficit; radiographic<br>findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a sudden loss of sensory fur | nction due to an intracranial vascu | lar event. | | |
| Syncope | <b>3</b> 3 | | Fainting; orthostatic collapse | 98 | |
| Definition: A disorder characteriz | ed by spontaneous loss of conscio | ousness caused by in sufficient blo | od supplyto the brain. | | 23 |

CTCAE 4.0 - May 25, 2009 ; Ne no to system disorders

CARTISTEM® 

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Transient ischemic attacks | Mild neurologic deficit with or without imaging confirmation | Moderate neurologic deficit with<br>or without imaging confirmation | - | £ | - |
| Definition: A disorder characte | rized by a brief attack (less than 24 h | nours) of cerebral dysfunction of v | ascular origin, with no persistent r | neurological deficit. | 00 |
| Tremor | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | <u> </u> | |
| Definition: A disorder characte | rized by the uncontrolled shaking mo | vernent of the whole body or indiv | idual parts. | | W. |
| Trigeminal nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | i <del>.</del> |
| Definition: A disorder characte | rized by involvement of the trigemina | I nerve (fifth cranial nerve). | | · | 2 |
| Valgus nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by involvement of the vagus ne | rve (tenth cranial nerve). | #: **<br> | er | |
| Va sovagal reaction | 3.5 | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte increase in the stimulation of the | rized by a sudden drop of the blood p<br>ne vagus nerve . | pressure, bradycardia, and periph | eral vasodilation that may lead to | loss of consciousness, It results fr | om an |
| Nervous system disorders -<br>Other , specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CARTISTEM® 

| | Pregna | ancy, puerperium and pe | erinatal conditions | | |
|---|---|---|---|---|---|
| Adverse Event | Grade | | | | |
| | 1 | 2 | 3 | 4 | 5 |
| Fetal death | | | | | Fetal loss at<br>any<br>gestational<br>age |
| Definition: A disorder character<br>expulsion from the uterus, with | ized by death in utero; failure of the<br>out possibility of resuscitation. | product of conception to show ev | vidence of respiration, heartbeat, o | r definite movement of a voluntary | /muscle a ter |
| Fetal growth retardation | | <10 % percentile of weight for gestational age | <5% percentile of weight for gestational age | <1% percentile of weight for gestational age | |
| Definition: A disorder character | ized by inhibition of fetal growth res | ulting in the inability of the fetus to | achieve its potential weight. | | |
| Premature delivery | Delivery of a liveborn infant at >34to 37 weeks gestation | Delivery of a liveborn infant at >28 to 34 weeks gestation | Delivery of a liveborn infant at 24 to 28 weeks gestation | Delivery of a liveborn in fant at 24 weeks of gestation or less | - |
| Definition: A disorder character<br>ge station. | ized by delivery of a viable infant be | fore the normal end of gestation. | Typically, viability is achievable be | Atween the twentieth and thirty-se | venth week of |
| Unintended pregnancy | - | 8 | Unintended pregnancy | NO. | ŀ |
| Definition: A disorder character | ized by an unexpected pregnancy a | t the time of conception. | 25 | | ***<br>*** |
| Pregnancy, puerperium and<br>perinatal ∞n ditions - Other,<br>specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, local or noninvasive<br>intervention indicated; limiting<br>instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Nervous system disorders 55 CTCAE 4.0 - May 28, 2009 : Pregnancy, puerperium and perinatal conditions 56

CARTISTEM® 

| | 1/4 | Psychiatric dison | ders | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | - 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | Severe agitation; hospitalization not indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by a state of restlessness asso | ciated with unpleasant feelings of | irritability and tension. | | ř |
| An orgasmia | Inability to achieve orgasm not<br>adversely affecting relationship | hability to achieve orgasm<br>adversely a ffecting relationship | . 159<br>10 | 3 | 5 |
| Definition: A disorder charac | terized by an inability to achieve orgas | m. | The same will | Transport and the superiores | Doggano |
| Anxiety | Mild symptoms; intervention not<br>indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; hospitalization not<br>indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder charac<br>stimulus. | terized by apprehension of danger and | d dread accompanied by restlessn | ess, tension , tachycardia , and dys | spinea unattached to a clearly ident | ifable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by a lack of clear and orderly t | hought and behavior. | 2 | | |
| Delayed orgasm | Delay in a chie ving orgasm not adversely affecting relationship | Delay in achieving orgasm<br>adversely a ffecting relationship | • | 9 | ē |
| | terized by sexual dysfunction characte | (c) | 1 | 1 | |
| Delirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional state; limiting self care ADL; hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization in dicated | Death |
| Definition: A disorder charac<br>eversible condition . | terized by the acute and sudden devel | opment of confusion , illusions , mo | vernent changes, inattentiveness | , agitation, and hallucinations. Usu | ally, it is |
| Delusion s | 5 <b>*</b> 25 | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac | terized by false personal beliefs held o | ,<br>ontrary to reality, de spite contradi | ,<br>ctorv evidence and common sens | | E |
| Depre ssion | Mild depressive symptoms | Moderate depressive<br>symptoms; limiting instrumental<br>ADL | Severe depressive symptoms;<br>limiting selfcare ADL;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac | terized by melancholic feelings of grie | Elizabeth Communication Commun | | | E) |
| Suphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g.,<br>hypomania) | E . | |
| Definition: A disorder charac | terized by an exaggerated feeling of w | ,<br>ell-being which is disproportionate | to events and stimuli. | | |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac | terized by a false sensory perception i | n the absence of an external stimu | ilus. | | |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling<br>asleep , staying asleep or<br>waking up early | Severe difficulty in falling<br>asleep, staying asleep or<br>waking up early | | |
| Definition: A disorder charac | terized by difficulty in falling asleep an | d <i>i</i> or remaining asleep. | | | |
| ibido decreased | Decrease in sexual interest not<br>adversely affecting relationship | Decrease in sexual interest adversely a ffecting relationship | - | 8 | - |
| Definition: A disorder charac | terized by a decrease in sexual desire | 727<br> | 15. S | 5 | (5) |
| ibido increased | Mild increase in sexual interest<br>not adversely affecting<br>relation ship | Moderate increase in sexual<br>interest adversely affecting<br>relationship | Severe increase in sexual interest leading to dan gerous behavior | | - |
| Definition: A disorder charac | terized by an increase in sexual desire | 4 | io. V | 5 | (6) |
| Mania | Mild manic symptoms (e.g.,<br>elevated mood, rapid thoughts,<br>rapid speech, decreased need<br>for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g.,<br>hypomania; major sexual or<br>financial indiscretions);<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac | terized by excitement of psychotic pro | portions manifested by mental and | l physical hyperacti vity, disorgania | ration of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |

CTCA E 4  $\rm II$  - May 28 , 2009 : Psych lattic disorders

CARTISTEM® 

| | | Psychiatric disord | ders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1. | 2 | 3 | 4 | - 5 |
| Definition: A disorder character | rized by a conspicuous change in a p | person's behavior and thinking. | 50 E | | 2 |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(e.g., disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(e.g., paranoid; extreme<br>disorganization); hospitalization<br>not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder character<br>turnor. | ized by personality change, impaire | d functioning, and loss oftouch wi | th reality. It may be a manife statio | n of schizophrenia, bipolar disorde | r or brain |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | × | |
| Definition: A disorder character | ized by an inabilityto rest, relax or b | e still. | 50 X | 8 | XI. |
| Suicidal ideation | no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require<br>hospitalization | Specific plan to commit suicide<br>with serious intent to die which<br>requires hospitalization | - |
| Definition: A disorder character | ized by thoughts of taking one's own | n life. | | | r |
| Suicide attempt | 120 | | Suicide attempt or gesture<br>without intent to die which may<br>not require hospitalization | Suicide attempt with intent to<br>die which requires<br>hospitalization | Death |
| Definition: A disorder character | ized by selfin licted harm in an atte | mpt to end one's own life. | | | |
| Psychiatric disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin vasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting<br>self care ADL | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Psychiatric disorders 58

CARTISTEM® 

| | 10 | Renal and urinary dis | sorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | - 5 |
| Acute kidney injury Definition: A disorder charac | Creatinine level increase of >0.3 mg/dL; creatinine 1.5 - 2.0 x above baseline terized by the acute loss of renal functions. | Creatinine 2 - 3x above baseline | Creatinine >3x baseline or >40 mg &L hospitalization indicated | Life-threatening consequences;<br>dialysis indicated | Death |
| auses (ureteral or bladder o | 48 STAR RE 60 | <i>k</i> | 9 | ( | |
| Bladder perforation | terized by a rupture in the bladder wall | Extra peritoneal perforation, indwelling catheter indicated | Intraperitoneal perforation;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences;<br>organ failure; urgent operative<br>intervention in dicated | Death |
| Bladder spasm | Intervention not indicated | Antispasmo dics indicated | Ho spitalization indicated | | Ī. |
| | terized by a sudden and involuntary co | 9 | The spitalization indicated | 10 | F. |
| | - II 3 | 15 | -CED C-Cl20 45 | - OFD C-Q / 15 IX-:- 8 70 | Deat |
| Chronio kidney disease | eGFR (estimated Glomerular<br>Filtration Rate) or CrCl<br>(creatinine clearance) < 60<br>ml/min /1.73 m2 or proteinuria<br>2+ present; urine<br>protein & reatinine > 0.5 | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 16<br>ml tmin/1.73 m2 | e GFR or CrCl < 15 ml/min/1.73<br>m2; dialysis or renal transplant<br>indicated | Death |
| Definition: A disorder charac | terized by gradual and usually perman | ent loss of kidne y function resultin | g in renal failure. | | |
| Cystitis noninfective | Microscopic hematuria; minimal<br>increase in frequency, urgency,<br>dysuria, or nocturia; new onset<br>of incontinence | Moderate hematuria; moderate increase in frequency, urgency, dysuria, no cturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV<br>medications or hospitalization<br>indicated; elective endoscopio,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| | terized by inflammation of the bladder | White the second second second second | | | Longe |
| Hematuria | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; urinary catheter<br>or bladder i migation indicated;<br>limiting instrumental ADL | Gross hematuria; transfusion, M<br>medications or hospitalization<br>indicated; elective endoscopic,<br>radiologic or operative<br>intervention indicated; limiting<br>self care ADL | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder charac | terized by laboratory test results that in | dicate blood in the urine. | 20 2 | | 20 |
| Hemoglo binuria | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | | | • | |
| Definition: A disorder charac | terized by laboratory test results that in | dicate the presence of free hemo | globin in the urine. | | 20 |
| Proteinuria | 1+ proteinuria; urinary protein<br><1.0 g/24 hrs | Adults: 2+ proteinuria; urinary<br>protein 1.0 | Adults: urinary protein >3.5 g/24<br>hrs;<br>Pediatric urine P/C<br>(Protein/Creatinine)>1.9 | | |
| Definition: A disorder charac | terized by laboratory test results that in | dicate the presence of excessive | protein in the urine . It is predomin | antly albumin, but also globulin. | ř |
| Renal calculi | Asymptomatic or mild<br>symptoms; occasional use of<br>non prescription a nalge sics<br>indicated | Symptomatic; oral antiemetics<br>indicated; around the clock<br>nonprescription analgesics or<br>any oral narcotic analgesics<br>indicated | Ho spitalization indicated; IV<br>intervention (e.g., analgesics,<br>antiemetics); elective<br>endoscopic or radiologic<br>intervention indicated | Life-threatening consequences;<br>urgent radiologic, endoscopic or<br>operative intervention in dicated | Death |
| Definition: A disorder charac | terized by the formation of crystals in th | he pelvis of the kidne y. | 1 | | |
| Renal colic | Mild pain not interfering with<br>activity; nonprescription<br>medication indicated | Moderate pain ; limiting<br>instrumental ADL; prescription<br>medication indicated | Hospitalization indicated;<br>limiting self care ADL | - | - |
| Definition: A disorder charac | terized by paroxysmal and severe fank | k marked discomfort radiating to th | ne inguinal area . Often , the cause | is the passage of kidney stones. | |
| Renal hernorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit<br>monitoring indicated | Transfusion, radiation, or<br>hospitalization indicated;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Renatland infinary disorders

CARTISTEM® 

| | W. | Renal and urinary di | sorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder character | rized by bleeding from the kidney. | 50 | 77 | | 00 |
| Urinary fistula | | Noninvasive intervention indicated; urinary or suprapublic cath eterpla cement indicated | Limiting self care ADL; elective<br>radiologic, endo scopic or<br>operative intervention indicated;<br>permanent urinary diversion<br>indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| (: | rized by an abnormal communication | 10 | system and another organ or an ato | omic site. | |
| Urinary frequency | Pre sent | Limiting instrumental ADL;<br>medical management indicated | 5.0 | •3 | 1 |
| Definition: A disorder character | rized by urination at short intervals. | | å. | | 8 |
| Urinary incontinence | Occasional (e.g., with coughing,<br>sneezing, etc.), pads not<br>indicated | Spontaneous; pads indicated;<br>limiting instrumental ADL | Intervention indicated (e.g., clamp, collagen injections); operative intervention indicated; limiting self care ADL | No. | |
| Definition: A disord er character | rized by inability to control the flow o | f urine from the bladder. | | • | |
| Urinary retention | Urinary, suprapubic or intermittent catheter placement not indicated; able to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Bective operative or radiologic<br>intervention indicated;<br>substantial loss of affected<br>kidney function or mass | Life-threatening consequences;<br>organ failure; urgent operative<br>intervention in dicated | Death |
| SAC WELL STREET | rized by accumulation of urine within | V NA TORRESON | St. No. 101 SECTION SEC. | lass is | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ function (e.g., hydronephrosis, or renal dysfunction); elective radiologic, endo scopic, or operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | rized by blockage of the normal 10 w | of contents of the urinary tract. | RC 20 | | (F) |
| Urinary tract pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 12 | |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the urinary tract. | | | * |
| Urinar y urgency | Pre sent | Limiting instrumental ADL;<br>medical management indicated | 50 | 7/2 | E . |
| Definition: A disorder character | rized by a sudden compelling urge to | urinate. | | | X.: |
| Urine discoloration | Pre sent | 5 | 58 | 55 | - |
| Definition: A disorder character | rized by a change in the color of the | urine. | B 0 | | <b>N</b> |
| Renal and urinary disorders -<br>Other , specify | Asymptomatic or mild<br>symptoms; dinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, Jocal or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Renal and urinary disorders 60

CARTISTEM® 

| | Rep | roductive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | 1- | Grade | | |
| Adverse Event | 1 | -2 | 3 | 4 | 5 |
| Azoo spermia | -8 | <br>[: | Absence of sperm in ejaculate | 2 | - |
| Definition: A disorder characte | erized by laboratory test results that in | dicate complete absence of spen | matozoa in the semen . | 1 | 2 |
| Breast atrophy | Minimal asymmetry; minimal atroph y | Moderate asymmetry; moderate atrophy | Asymmetry >1.8 of breast volume; severe atrophy | ≅<br>} | |
| Definition: A disorder characte | erized by underdevelopment ofthe br | east. | | | |
| Breast pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 8 | - |
| | erized by marked discomfort sensation | E | T | 1 | F |
| Dysmenorrhea | Mild symptoms; Intervention not<br>indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | Ì |
| Definition: A disorder characte | erized by abnormally painful abdomin | al cramps during menses. | | | |
| Dyspareunia | Mild discomfort or pain<br>associated with vaginal<br>penetration; discomfort relieved<br>with use of vaginal lubricants or<br>estrogen | Moderate discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>partially relieved with use of<br>vaginal lubricants or estrogen | Severe discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>unrelie ved by vaginal lubricants<br>or estrogen | 3 | 5 |
| Definition: A disorder characte | erized by painful or difficult coitus. | | | | |
| Eja culation disorder | Diminished ejaculation | Anejaculation or retrograde ejaculation | | 8 | |
| Definition: A disorder characte | erized by problems related to ejaculat | on. This category includes prema | ture, delayed, retrograde and pair | nful ejaculation. | 35 |
| Erectile dysfunction | Decrease in erectile function<br>(frequency or rigidity of<br>erections) but intervention not<br>indicated (e.g., medication or<br>use of mechanical device,<br>penile pump) | Decrease in erectile function<br>(frequency/rigidity of erections),<br>erectile intervention indicated,<br>(e.g., medication or mechanical<br>devices such as penile pump) | Decrease in erectile function<br>(frequency/figidity of erections)<br>but erectile intervention not<br>helpful (e.g., medication or<br>mechanical devices such as<br>penile pump); placement of a<br>permanent penile prosthesis<br>indicated (not previously<br>present) | | - |
| Definition: A disorder characte | ।<br>erized by the persistent or recurrent in | l<br>abilitysto achieve or to maintain as | | Į. | 15 |
| Fallopian tube obstruction | Diagno stic ob servation's only;<br>intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | | |
| Definition: A disorder characte | ।<br>erized by blockage ofthe normal <b>1</b> ow | | | 1 | I. |
| Fallopian tube stenosis | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A disorder characte | erized by a narrowing of the fallopiant | tube lumen . | | | |
| Fernale genital tract fistula | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between a female reproductive s | ystem organ and another organ o | r anatomic site . | |
| eminization acquired | Mild symptoms; Intervention not indicated | Moderate symptoms; medical<br>intervention indicated | | 8 | - |
| Definition: A disorder characte | erized by the development of seconda | ry female sex characteristics in m | ales due to extrinsic factors. | 5 | (5) |
| Genital edema | Mild swelling or obscuration of<br>anatomic architecture on close<br>inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent de viation from normal<br>anatomic contour | Lymphorrhea; gross de viation<br>from normal anatomic contour;<br>limiting self care ADL | ů. | - |
| Definition: A disorder characte | erized by swelling due to an excessive | e accumulation of fuid in the genit | als. | 9 | 30 |
| Gynecomastia | Asymptomatic breast enlargement | Symptomatic (e.g., pain or psychosocial impact) | Severe symptoms; elective operative intervention indicated | E . | |
| Definition: A disorder characte | erized by excessive development of the | | | | |
| Hematosalpinx | Minimal bleeding identified on<br>imaging study or laparoscopy;<br>intervention not in dicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

CTCA E 4.0 - May 28,2009 : Reproductive system and breast disorders 61

CARTISTEM® 

| 3 | Rep | productive system and br | east disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | ं |
| | terized by the presence of blood in a t | allopian tube. | | | 001 |
| megular menstruation | Intermittent menses with<br>skipped menses for no more<br>than 1 to 3 months | Intermittent menses with<br>skipped menses formore than 4<br>to 6 months | Persistent amenormea for more than 6 months | | 5 |
| Definition: A disorder charact | terized by irregular cycle or duration o | fmenses. | | | 001 |
| Lactation disorder | Mild changes in lactation, not<br>significantly affecting production<br>or expression of breast milk | Changes in lactation ,<br>significantly affecting breast<br>production or expression of<br>breast milk | ₹0 | | 5 |
| Definition: A disorder charact | terized by disturbances of milk secretion | on. It is not necessarily related to p | regnancythat is observed in fem | ales and can be observed in male | s. |
| Meno mhagia | Mild; iron supplements indicated | Moderate symptoms; medical intervention indicated (e.g., hormones) | Severe; transfusion indicated;<br>surgical intervention in dicated<br>(e.g., hysterectomy) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by abnormally heavy vaginal b | leeding during menses. | (i) | į. | 0 |
| Nipple de formity | Asymptomatic; asymmetry with<br>slight retraction and for<br>thickening of the nipple areolar<br>complex | Symptomatic; asymmetry of<br>nipple areolar complex with<br>moderate retraction and/or<br>thickening of the nipple areolar<br>complex | 20 | 2 | |
| Definition: A disorder charact | erized by a mal formation of the nipple | And the second s | | , | |
| Oligospermia | Sperm concentration >48<br>million/mL or motility >68% | Sperm concentration 13 - 48<br>million/mLormotility 32 - 68% | Sperm concentration <13<br>million/mL or motility <32% | ÷. | ŧ |
| Definition: A disorder charact | terized by a decrease in the number o | f spermatozoa in the semen. | | | |
| Ovarian hemorrhage | Minimal bleeding identified on<br>imaging study or laproscopy;<br>intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | terized by bleeding from the overy. | TS 50 50 50 50 70 | E10 9000 200000 | 9890 70 | 200 00 |
| Ovarian rupture | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by tearing or disruption of the o | ovarian tissue. | | - | |
| Ovulation pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | * |
| | terized by marked discomfort sensatio | n in one side of the abdomen betw | een menstrual cycles, around the | time of the discharge of the own | fomth |
| ovarian follicle. | - T | | \$ 6550 ST | WFG C. | |
| Pelvic floormuscle weaknes: | <ul> <li>Asymptomatic; clinical or<br/>diagnostic observations only;<br/>intervention not indicated</li> </ul> | Symptomatic, not interfering with bladder, bowel, or vaginal function; limiting in strumental ADL | Severe symptoms; limiting self<br>care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by a reduction in the strength o | f the muscles of the pelvic foor. | | | 001 |
| <sup>a</sup> elvic pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | ē. | - |
| Definition: A disorder charact | terized by marked discomfort sensatio | n in the pelvis. | Los Allianos Plan | | |
| <sup>p</sup> enile pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 2 | ŧ |
| Definition: A disorder charact | terized by marked discomfort sensatio | n in the penis. | | | |
| <sup>a</sup> erineal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | a | - |
| Definition: A disorder charact | erized by a sensation of marked disco | omfort in the area between the gen | ital organs and the anus. | is . | (V) |
| Premature menopause | - P | | Present | 2 | 2 |
| Definition: A disorder charact | erized by ovarian failure before the ag | ge of 40 . Symptoms include hot fla | shes, night sweats, mood swings | and a decrease in sex drive. | |
| Pro static hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

CTCA E 4.0 - May 28, 2009 : Reproductive system and breast disorders

CARTISTEM® 

| | | productive system and b | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | erized by bleeding from the prostate : | - | | | |
| Prostatic obstruction | Diagnostic observations only;<br>intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | 2 | 5 |
| Definition: A disorder characte<br>stream, and incomplete empty | erized by compression of the urethra<br>ying of the bladder). | secondary to enlargement of the p | prostate gland. This results in wold | ing difficulties (straining to void, sk | ow urine |
| Prostatic pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain ; limiting self care<br>ADL | 3 | 5 |
| Definition: A disorder characte | erized by a sensation of marked disc | omfort in the prostate gland. | | | |
| Scrotal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain ; limiting self care<br>ADL | 5 | |
| Definition: A disorder characte | erized by marked discomfort sensation | on in the scrotal area. | | | |
| Spermatic cord hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by bleeding from the spermation | cord. | To: 101 00 | T | |
| Spermatic cord obstruction | Diagnostic observations only;<br>intervention not indicated | Mild symptoms; elective<br>intervention indicated | Severe symptoms; elective operative intervention indicated | € | ŧ |
| Definition: A disorder characte | erized by blockage of the normal flow | of the contents of the spermatic o | ord. | 1 | r |
| Testicular disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicate d | Symptomatic but not interfering<br>with urination or sexual<br>activities; intervention not<br>indicated; limiting instrumental<br>ADL | Severe symptoms; interfering<br>with urination or sexual function;<br>limiting self care ADL;<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by involvement of the testis. | No. | 141 21 | 1 | 001 |
| Testicular hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by bleeding from the testis. | | | | |
| Testicular pain | Mild pain | Moderate pain ; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 30 | - |
| Definition: A disorder characte | erized by a sensation of marked disc | omfort in the testis. | Tale and the second street of | www.comerconarts.com | Tearmous |
| Uterine fistula | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communicatio | n between the uterus and another | organ or anatomic site. | | 001 |
| Uterine hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Source and a second second | erized by bleeding from the uterus. | Same and the same | Transportation of the second | 100 | r - |
| Uterine obstruction | Diagno stic observations only;<br>intervention not indicated | Mild symptoms; elective<br>intervention indicated | Severe symptoms; elective operative intervention indicated | | |
| Definition: A disorder characte | erized by blockage of the uterine outl | et. | | | T. |
| Iterine pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | S. | |
| Definition: A disorder characte | erized by a sensation of marked disc | omfort in the uterus. | | I | |
| ∕aginal discharge | Mild vaginal discharge (greater<br>than baseline for patient) | Moderate to heavy vaginal<br>discharge; use of perineal pad<br>or tampon indicated | | | |
| Definition: A disorder characte | erized by vaginal secretions. Mucus p | produced by the cervical glands is | discharged from the vagina natura | ally, especially during the childbear | ing years |
| | ALCOHOL WINGSON | Moderate vaginal dryness | Severe vaginal dryness | are. | L |

CTCA E 4.0 - May 28,2009 : Reproductive system and breast disorders

CARTISTEM® 

| | Grade | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| vaginal fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Vaginal hemorrhage | ed by an abnormal communication Minimal bleeding identified on clinical exam or imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characterizo | Mild discomfort or pain, edema,<br>or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal<br>ulceration; life-threatening<br>con sequences; urgent<br>intervention in dicated | Death |
| Definition: A disorder characterizo<br>Vaginal obstruction | Diagno stic ob servation's only; | Mild symptoms; elective | dness, edema, marked discomfort<br>Severe symptoms; elective | and an increase in vaginal dischar | rge. |
| Definition: A disorder characterize | intervention not indicated | intervention indicated | operative intervention indicated | | ŀ |
| Vaginal pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain ; limiting self care<br>ADL | - | |
| Definition: A disorder characterize | ed by a sen sation of marked disco<br>Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the vaginal wall | 20.<br> | % | | %<br>• |
| vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or<br>shortening not interfering with<br>physical examination | Vaginal narrowing and or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | | Death |
| Definition: A disorder characterize | ed by a narrowing ofthe vaginal c | anal. | | | |
| √a ginismus | Mild discomfort or pain<br>associated with vaginal spasm/<br>tightening; no impact upon<br>sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spasm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal spasm/<br>tightening; unable to tolerate<br>vaginal penetration or physical<br>examination | | |
| Definition: A disord er characterize<br>intercourse. | ed by involuntary spasms of the p | elvic floor muscles, resulting in pa | nthologic tightness of the vaginal w | all during penetration such as duri | ng sexua |
| Reproductive system and breast<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninva sive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization in dicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention in dicated | Death |

CARTISTEM® 

**CONFIDENTIAL:** These all contents herein are the sole property of MEDIPOST Co., Ltd. Any reproduction or distribution of this document without the written consent of MEDIPOST Co., Ltd is prohibited. Copyright © 2017 MEDIPOST Co., Lt

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | -2 | 3 | 4 | - 5 |
| Adult respiratory distress<br>syndrome | | | Present with radiologic findings;<br>intubation not indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac<br>surgeny. | cterized by progressive and life-th-reater | ning pulmonary distress in the abs | ence of an underlying pulmonary | condition, usually following major t | rauma o |
| Allergic rhinitis | Mild symptoms; intervention not indicated | intervention indicated | to the second second | 55 | |
| | cterized by an inflammation of the nasa<br>anes of the sinuses, eyes, middle ear, a | | | | ay also |
| Apnea | | | Present; medical intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by cessation of breathing. | en<br>Managone anno en | by Construction of the Science | | Errorran |
| Aspiration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Attered eating habits; coughing<br>or choking episodes after eating<br>or swallowing; medical<br>intervention indicated (e.g.,<br>suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); ho spitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by inhalation of solids or liquids | s into the lungs. | I. | | |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | oterized by the collapse of part or the el | DE SOLUTION DE LA COMPANIONE | | 1.2.4 | 40740 |
| Bronchial fstula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endo scopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder charac | cterized by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild wheezing); endoscopic evaluation indicated; radio graphic evidence of atelecta sis/lobar collapse; medical management indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor;<br>endoscopic intervention<br>indicated (e.g., laser, stent<br>placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by blockage of a bronchus pas | sage, most often by bronchial sec | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor;<br>endoscopic intervention<br>indicated (e.g., laser, stent<br>placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | cterized by a narrowing of the bronchial | tube. | T | T | C. |
| Bronchopleural fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endo scopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage ormultiple<br>thoracotomies indicated | Death |
| Definition: A disorder charac | cterized by an abnormal communication | between a bronchus and the ple | ural cavity. | | |
| Bro nchopulmon ary he mo mh | age Mild symptoms; intervention not indicated | Moderate symptoms; medical<br>intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g., | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention | Death |

CTCAE 4.0 - May 28, 2009 : Respiratory, the racid and medias thial disorders

CARTISTEM® 

| | Respii | atory, thoracic and med | 0.000 (0.000) | | |
|---|---|---|---|---|---|
| | | Grade 4 2 2 4 | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Pronchospasm | Mild symptoms; intervention not<br>indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | Limiting self care ADL; oxygen<br>saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | sterized by a sudden contraction of the | smooth muscles of the bronchial | wall. | | |
| Chylothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thoracentesis or<br>tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | eterized by milky pleural effusion (abnor | mal collection of fluid) resulting fi | om accumulation of lymph fuid in | the pleural cavity. | |
| Cough | Mild symptoms; nonprescription<br>intervention indicated | Moderate symptoms, medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | • | ŧ |
| Definition: A disorder charac | sterized by sudden, often repetitive, spa | smodic contraction of the thoraci | c cavity, resulting in violent release | e of air from the lungs and usually | accompa |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with minimal exertion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an uncomfortable sensation | of difficulty breathing. | ## S | | Si . |
| Epistaxis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated (e.g., nasal packing, cauterization; to pical vasoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | eterized by bleeding from the nose. | Tis | 1 | | r |
| Hiccups | Mild symptoms; intervention not indicated | Moderate symptoms; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; interfering<br>with sleep; limiting selfcare<br>ADL | | 2 |
| Definition: A disorder charac | eterized by repeated gulp sounds that re | sult from an involuntary opening | and closing of the glottis. This is a | rttributed to a spasm of the diaphra | igm. |
| Hoarsene ss | Mild or intermittent voice<br>change; fully understandable;<br>self-resolves | Moderate or persistent voice<br>changes; may require<br>occasional repetition but<br>understandable on telephone;<br>medical evaluation indicated | Severe voice changes including<br>predominantly whispered<br>speech | | 2 |
| Definition: A disorder charac | terized by harsh and raspy voice arisin | g from or spreading to the larynx | | Towns and the | |
| Hypoxia | - | Decreased oxygen saturation<br>with exercise (e.g., pulse<br>oximeter <88%); intermittent<br>supplemental oxygen | Decreased oxygen saturation at<br>rest (e.g., pulse oximeter <88 %<br>or Pa 02 <=55 mm Hg) | Life-threatening airway<br>compromise; urgent intervention<br>in dicated (e.g., tracheotomy or<br>intubation) | Death |
| | sterized by a decrease in the level of ox | CONTRACTOR CONTRACTOR | 10 2000 100 000 100 100 100 100 100 100 | TO THE PROPERTY AND ADDRESS OF THE PROPERTY OF | Discussion |
| La nyn geal edema | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | Stridor; respiratory distress;<br>hospitalization in dicate d | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charac | sterized by swelling due to an excessive | e accumulation of fluid in the lary | ix. | 1 | ř |
| Laryngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endo scopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thora coplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder charac | eterized by an abnormal communication | between the larynx and another | organ or anatomic site. | T0.00055 355 No. 1 | 2510 00 |
| Laryn geal hemorth age | Mild cough or trace hemoptysis;<br>laryngo scopic findings | Moderate symptoms; medical<br>intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charac | eterized by bleeding from the larynx. | No. | | | ni. |
| Laryngeal inflammation | Mild sore throat; raspy voice | Moderate sore throat; | Severe throat pain; endoscopic | 20 | ż |

CTCAE 4.0 - May 28, 2009 : Respiratory, the racid and medias that disorders

CARTISTEM® 

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | |
| aryngeal mucositis | Endoscopic findings only; mild discomfort with normal intake | Moderate discomfort; altered<br>oral intake | Severe pain; severely aftered<br>eating/su allowing; medical<br>intervention indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| | ed by an inflammation involving th | [= | T : | | r |
| Laryngeal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic (e.g., noisy airway<br>breathing), but causing no<br>respiratory distress; medical<br>management indicated (e.g.,<br>steroids); limiting instrumental<br>ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage ofthe laryngeal air | way. | 6<br>4 | | (1)<br>(1) |
| Laryngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway<br>breathing), but causing no<br>respiratory distress; medical<br>management indicated (e.g.,<br>steroids) | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the laryngeal | airway. | 100 100 10 | 0.5070 70 | PEID 60 |
| Laryngopharyngeal dysesthesia | Mild symptoms; no anxiety;<br>intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspnea and<br>swallowing difficulty; limiting self<br>care ADL | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by an uncomfortable persistent | sen sation in the area of the laryn | gopharynx. | | 2 |
| Laryngospasm | | Transient e pisode ; intervention<br>not indicate d | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngo scopy,<br>intubation, botox injection) | Death |
| Definition: A disorder characteriz | ,<br>ed by paroxysmal spasmodic mus | cular contraction of the vocal cord | S | • Note of the control | ķ: |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated<br>(e.g., hernostasis of bleeding<br>site) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the mediastin | um. | <b>5</b> | | Si<br>or |
| Nasal congestion | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Associated with bloody na sall<br>discharge or epistaxis | | 2 |
| Definition: A disorder characteriz | ed by obstruction of the nasal pas | sage due to mucosal edema. | N. S. | | gi<br>Perro-oco |
| Pharyngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endo scopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Character and person a street repaired | ed by an abnormal communication | Character and the Marian and the same | Tanada anamana and anamana and a | THE CONTRACTOR OF STREET | i.<br>Dominio |
| Pharyngeal hemorrhage | Mild symptoms; intervention not<br>indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the pharynx. | Diameter Control | | | |
| Pharyngeal muoositis | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics<br>indicated; altered oral intake;<br>limiting instrumental ADL | Severe pain; unable to<br>adequately aliment or hydrate<br>orally; limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an inflammation involving th | e mucous membrane of the phary | mx. | | Total Control |
| Pharyngeal necrosis | ======================================= | | hability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

CTCAE 4.0 – May 28, 2009 : Respirato  $y_{\rm c}$  tho racid and medias thall disorde is 67

CARTISTEM® 

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1: | 2 | 3 | 4 | : :: |
| Definition: A disorder charac | terized by a necrotic process occurring | in the pharynx. | as 20 | · | 01 |
| Pharyngeal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic (e.g., noisy airway<br>breathing), but causing no<br>respiratory distress; medical<br>management indicated (e.g.,<br>steroids); limiting instrumental<br>ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder charac | terized by a narrowing of the pharynge | al ainway. | | | |
| <sup>a</sup> haryngolar yng eal pain | Mild pain | Moderate pain ; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 5 | ÷ |
| Definition: A disorder charac | terized by marked discomfort sensation | n in the pharyngolaryngeal region | č | | |
| Pleural effusion | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; intervention<br>indicated (e.g., diuretics or<br>limited therapeutic<br>thoracentesis) | Symptomatic with respiratory distress and hypoxia; surgical intervention including chest tube or pleuro desis indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | terized by an increase in amounts of fl | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomfo | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage confirmed by thoracentesis | Symptomatic or a ssociated with<br>pneumothorax; chest tube<br>drain age indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charac | terized by bleeding from the pleural ca | vity. | 6)<br>() | £ ( | 21 |
| Pleuritic pain | Mild pain | Moderate pain ; limitin g<br>instrumental ADL | Severe pain ; limiting self care<br>ADL | - | - |
| Definition: A disorder charac | terized by marked discomfort sensation | n in the pleura. | 2 | | ni. |
| Pn eumonitis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; oxygen indicated | Life-threatening respiratory<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charac | terized by inflammation focally or diffus | sely affecting the lung parench ym: | 1. | | 20 |
| neumothorax | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; intervention indicated (e.g., tube placement without sclerosis) | Sclerosis and/or operative<br>intervention indicated;<br>hospitalization indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by abnormal presence of air in | the pleural cavity resulting in the | collapse of the lung. | | 51 |
| ostnasal drip | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | | | i<br>e |
| Definition: A disorder charac | terized by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | 01 |
| Productive cough | Occasional/minimal production of sputum with cough | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | | į. |
| Definition: A disorder charac | terized by expectorated secretions upo | D-8770 23 10 | T-22 52 50 10 11 | 1000000 72 50 50 | 200 00 |
| Pulmo nary e dema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspinea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspinea or dyspinea at<br>rest; o xygen indicated; limiting<br>self care ADL | Life-threatening respiratory<br>compromise; urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder charac | terized by accumulation of fuid in the I | ung tissues that causes a disturba | ance of the gas exchange that may | y lead to respiratory failure. | 01 |
| Pulmonary fibrosis | Mild hypoxemia; radiologic<br>pulmonary fibrosis < 25% of<br>lung volume | Moderate hypoxemia; evidence<br>of pulmonary hypertension;<br>radio graphic pulmona ry fibrosis<br>25-50 % | Severe hypoxemia; evidence of<br>right-sided heart failure;<br>radiographic pulmonary fbrosis<br>>50 - 75% | Life-threatening consequences<br>(e.g., hemodynamic/pulmonary<br>complications); intubation with<br>ventilatory support indicated;<br>radiographic pulmonary fibrosis<br>>75% with severe<br>honeycombing | Death |
| Definition: A disorder charac | terized by the replacement of the lung | tissue by connective tissue , leadir | ng to progressive dyspinea, reispira<br>I | tory failure or right heart failure. | ni<br>Persona |
| Pulmonary fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; tube<br>th oracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Umiting self care ADL;<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>in dicated | Death |

CTCAE 4.0 - May 28, 2009 : Respiratory, the racid and medias that disorders

CARTISTEM® 

| | Respii | ratory, thoracic and med | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | terized by an abnormal communication | | | STERNAD AND STREAM COLORS COLORS CO. | ni<br>Dogovos |
| Pulmonary hypertension | Minimal dyspnea; findings on physical exam or other evaluation terized by an increase in pressure with | Moderate dyspinea, cough;<br>requiring evaluation by cardiac<br>catheterization and medical<br>intervention | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening airway<br>consequences; urgent<br>internention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| | l some services and the services are services and the services and the services and the services are services and the services and the services are services are services and the services are services are services and the services are services are services are services are services and the services are services ar | I gamena y an earliant a con- | l and a second | I in the second | Domb |
| Respiratory failure | | | | Life-threatening consequences;<br>urgent intervention, intubation,<br>or ventilatory support indicated | Death |
| )efinition: A disorder charac<br>rith an increase in arterial le | terized by impaired gas exchange byt<br>wels of carbon dioxide: | he respiratory system resulting in | hypoxemia and a decrease in oxy | genation of the tissues that may b | e associa |
| Retinoic acid syndrome | Fluid retention; <3 kg of weight<br>gain; intervention with fluid<br>restriction and/or diuretics<br>indicated | Moderate signs or symptoms;<br>steroids indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences;<br>ventilatory support indicated | Death |
| Definition: A disorder charac<br>etino ic acid. | terized by weight gain, dyspnea, pleur | al and pericardial effusions, leukoc | cytosis and/or renal failure original | ly described in patients treated wit | h all-tran: |
| Sinus disorder | Asymptomatic mucosal crusting;<br>blood-tinged secretions | Symptomatic stenosis or edema/narrowing interfering with airflow; limiting instrumental ADL | Stenosis with significant nasal obstruction; limiting self care ADL | Necrosis of soft tissue or bone;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by involvement of the paranasa | al sinuses. | 5) b | | - |
| Gleep apnea | Snoring and noctumal sleep<br>arousal without apneic periods | Moderate apnea and oxygen<br>desaturation; excessive daytime<br>sleepiness; medical evaluation<br>indicated; limiting instrumental<br>ADL | Oxygen desaturation;<br>associated with hypertension;<br>medical intervention in dicated;<br>limiting self care ADL | Cardiovascular or<br>neurop sychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | ।<br>terized by cessation of breathing for sh | Landan Company of the | 1 | | Ŀ |
| on eezing | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | *1 | 8 | ŧ |
| | terized by the involuntary expulsion of | 7.5 | ALICE STATE OF THE SECOND | 0- | |
| ore throat | Mild pain | Moderate pain ; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to swallow | | |
| Definition: A disorder charac | terized by of marked discomfort in the | throat | 1 | | |
| Stridor | | | Respiratory distress limiting self<br>care ADL; medical intervention<br>indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charac | terized by a high pitched breathing sou | und due to laryngeal or upper airw | ay obstruction: | | |
| Fracheal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicate d | Symptomatic; tube<br>th oracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endo scopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder charac | terized by an abnormal communication | between the trachea and anothe | rorgan or anatomic site. | E 137 860 1 | ni<br>ni |
| racheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe pain; hemorrhage or respiratory symptoms; limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| lefinition: A disorder charac | terized by an inflammation involving th | e mucous membrane of the trache | 23. | 7 | n l |
| racheal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic (e.g., no isy airway<br>breathing), but causing no<br>respiratory distress; medical<br>management indicated (e.g., | Stridor or respiratory distress<br>limiting self care ADL;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |

CTCAE 4.0 – May 28, 2009 : Respirato  $y_{\rm c}$  tho racid and medias thal disorders 69

CARTISTEM® 

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Volice alteration Definition: A disorder character | Mild or intermittent change from normal voice | Moderate or persistent change from normal voice; still understandable | Severe voice changes including<br>predominantly whispered<br>speech; may require frequent<br>repetition or face-to-face contact<br>for understandability; may<br>require assistive technology | | • |
| Whee zing | Detectable airway noise with<br>minimal symptoms | Moderate symptoms; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe respiratory symptoms<br>limiting self-care ADL; oxygen<br>therapy or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | zed by a high-pitched, whistling sou | ,<br>and during breathing . It results fro | ,<br>m the narrowing or obstruction of t | he respiratory airways. | ida<br>C |
| Respiratory, thoracic and<br>mediastinal disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Respiratory, thoracic and mediastinal disorders 70

CARTISTEM® 

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Alopecia | for that individual that is not<br>obvious from a distance but only<br>on close inspection; a different<br>hair style may be required to<br>coverthe hair loss but it does | Hair loss of >50 % normal for<br>that individual that is readily<br>apparent to others; a wig or hair<br>piece is necessary if the patient<br>desires to completely<br>camouflage the hair loss;<br>associated with psychosocial<br>impact | 28 | | |
| Definition: A disorder charac | terized by a decrease in density of hair | 100 KN 100 10 | '<br>ndividual at a given age and body | location | 30 |
| Bo dy odor | Mild odor; physician intervention<br>not indicated; self care<br>interventions | Pronounced odor; psychosocial<br>impact; patient seeks medical<br>intervention | - | - | |
| Definition: A disorder charac | sterized by an abnormal body smell reso | ulting from the growth of bacteria : | on the body. | | 1 |
| Bullous dermatitis | Asymptomatic; blisters covering <10% BSA | Blisters covering 10-30 % BSA;<br>painful blisters; limiting<br>instrumental ADL | Blisters covering >30 % BSA;<br>limiting self care ADL | Blisters covering >30% BSA;<br>associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Dryskin | terized by inflammation of the skin cha<br>Covering <10% BSA and no<br>associated erythema or pruritus | Covering 10-30% BSA and associated with enythema or pruritus; limiting instrumental ADL | Covering >30 % B SA and associated with pruritus; limiting self care ADL | 5 | |
| Definition: A disorder charac | sterized by flaky and dull skin; the pores | are generally fine, the texture is: | a paperythin texture. | | Ť |
| Erythema multiforme | Target lesions covering <10%<br>BSA and not associated with<br>skin tenderness | Target le sions covering 10-30 %<br>BSA and associated with skin<br>tendemess | Target lesions covering >30 %<br>BSA and associated with oral or<br>genital erosions | Target lesions covering >30 %<br>B SA; associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder charac | terized by target lesions (a pink-red ring | g around a pale center). | 8 | | (8) |
| Erythroderma | | Erythema covering >90% BSA<br>without associated symptoms;<br>limiting instrumental ADL | Erytherna covering >90% BSA<br>with associated symptoms (e.g.,<br>pruritus ortendemess); limiting<br>selfcare ADL | Erythema covering >90% BSA<br>with associated fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder charac | terized by generalized inflammatory en | ytherna and exfoliation. The inflam | nmatory process involves > 90 % o | fthe body surface area. | |
| Fat atrophy | Covering <10% BSA and asymptomatic | Covering 10-30 % BSA and<br>associated with erythema or<br>tendemess; limiting instrumental<br>ADL | Covering >30 % B SA;<br>associated with erythema or<br>tendemess; limiting selfcare<br>ADL | | - |
| Definition: A disorder charac | sterized by shrinking of adipose tissue. | 20 | 2 | · | 22 |
| Hirsutism | | In women, increase in length,<br>thickness or density of hair in a<br>male distribution that requires<br>daily shawing or consistent<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial<br>impact | | 8 | |
| | terized by the presence of excess hair | growth in women in anatomic site | s where growth is considered to b | e a secondary male characteristic | and und |
| androgen control (beard, mo<br>Hyperhidrosis | Limited to one site (palms, soles, or axillae); self care interventions | h volving >1 site; patient seeks<br>medical intervention; associated<br>with psychosocial impact | Generalized involving sites other than palms, soles, or axillae; associated with electrolyte/hemodynamic imbalance | D | - |

CTCAE 4.0 - May 28, 2009 : Skill and subcutaneous tissue disorders

CARTISTEM® 

| | SK | in and subcutaneous tis | sue aisoraers | | |
|---|---|---|---|---|---|
| | | r | Grade | 1 | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or density of hair that the patient is either able to carnoufage by periodic shaving or removal of hairs or is not concerned enough about the overgrowth to use any form of hair removal | Increase in length, thickness or density of hair at least on the usual exposed areas of the body (face (not limited to beard/moustache area) plus/minus arms) that requires frequent shaving or use of destructive means of hair removal to camouflage; associated with psychosocial impact. | | | |
| Definition: A disorder characteri | ized by hair density or length beyon | d the accepted limits of normal in | a particular body region, for a part | icular age or race. | |
| Hypohidrosis | | Symptomatic; limiting instrumental ADL | horease in bodytemperature;<br>limiting self care ADL | Heat stroke | Death |
| Definition: A disorder characteri | zed by reduced sweating. | (E) | The second streams of the contract of the cont | | to: |
| ip ohypertroph y | Asymptomatic and covering <10% BSA | Covering 10-30% BSA and associated tenderness; limiting instrumental ADL | Covering >30% B SA and associated tendemess and narcotics or NS AIDs indicated; lipohypertrophy; limiting self care ADL | | Ī |
| Definition: A disorder characteri | zed by hypertrophy of the subcutan | eous a dipose tissue at the site of | multiple subcutaneous injections o | finsulin. | |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | | | + |
| | zed by a change in the color of the | 7.5 | T | | E |
| Nail loss | Asymptomatic separation of the<br>nail bed from the nail plate or<br>nail loss | Symptomatic separation of the<br>nail bed from the nail plate or<br>nail loss; limiting instrumental<br>ADL | | | |
| Definition: A disorder characteri | zed by loss of all or a portion of the | nail. | 2 | , | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | 6 | ed . | • | ŧ |
| Definition: A disorder characteri | zed by vertical or horizontal ridges | on the nails. | a × | , | |
| Pain ofskin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | P | |
| Definition: A disorder characteri | zed by marked discomfort sensation | n in the skin. | | | |
| <sup>p</sup> almar-plantar<br>erythrodysesthe <i>s</i> ia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>with out pain | Skin changes (e.g., peeling,<br>blisters, bleeding, edema, or<br>hyperkeratosis) with pain;<br>limiting instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>edema, or hyperkeratosis) with<br>pain; limiting self care ADL | ek | - |
| Definition: A disorder characteri | zed by redness, marked discomfort | , swelling, and tingling in the palm | s of the hands or the soles of the | feet. | |
| <sup>3</sup> eriorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual<br>disturbance; increased<br>intraocular pressure, glaucoma<br>or retinal hemorrhage; optio<br>neuritis; diuretios indicated;<br>operative intervention indicated | - | |
| Definition: A disorder characteri | zed by swelling due to an excessive | e accumulation of fuid around the | T . | | T |
| Photosen sitivity | Painless erythema and<br>erythema covering <10% BSA | Tender erythema covering 10-<br>30 % BSA | Erytherna covering >30% BSA<br>and erytherna with blistering;<br>photosensitivity; oral<br>conticosteroid therapy indicated;<br>pain control indicated (e.g.,<br>narcotics or NSAIDs) | Life-threatening consequences;<br>urgent intervention indicated | Death |

CTCAE 4.0 - May 28, 2009 : Skin and subcutaneous tasse disorders

CARTISTEM® 

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1: | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical<br>intervention indicated | Intense or widespread;<br>intermittent; skin changes from<br>scratching (e.g. edema,<br>papulation, excoriations,<br>lichenification, oozing.krusts);<br>oral intervention indicated;<br>limiting instrumental ADL | Intense or widespread;<br>constant; limiting self care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | | _ |
| lefinition: A disorder charact | terized by an intense itching sensation | | 6 | | 000 |
| urpura<br>Jefinition: A disorder charact | Combined area of lesions covering <10% BSA terior by hemorrhagic areas of the sk | Combined area of lesions covering 10-30 % BSA; bleeding with trauma in and mucous membrane. Newel | Combined area of lesions covering >30% BSA; spontaneous bleeding flesions appear reddish in color. ( | Older lesions are usually a darker j | purple col |
| nd e ventually become a bro | Fig. 10 | | (\$4) | \$5<br> | 700F |
| Rash acheiform | Papules and/orpustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30 % BSA, which may or may not be associated with symptoms of pruritus or tendemess; associated with psychosocial impact; limiting instrumental ADL | Papules and for pustules covering >30 % B SA, which may or may not be associated with symptoms of pruritus or tendemess; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tendemess and are associated with extensive superinfection with Martibiotics indicated; lifethreatening consequences | Death |
| efinition: A disorder charact | terized by an eruption of papules and p | oustules , typicall y appearing in fac<br>I | E12 12 10 10 10 10 | | |
| Rash ma culo-papular | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness) | Macules/papules covering 10-<br>30 % BS Awith or without<br>symptoms (e.g., pruritus,<br>burning, tightness); limiting<br>instrumental ADL | Macules/papules covering<br>>30 % B SA with or without<br>associated symptoms; limiting<br>self care ADL | | |
| | terized by the presence of macules (fla | | nown as morbillform rash, it is one | of the most common outaneous a | dverse |
| events, mequentry amecong tr<br>Scalp pain | he upper trunk, spreading centripetally<br>Mild pain | and associated with prumus. Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | S. | - |
| Definition: A disorder charact | terized by marked discomfort sensation | '<br>n in the skin covering the top and ' | the back of the head. | | |
| kin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10-30 % BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA;<br>associated with ulceration | | 2 |
| Definition: A disorder charact | terized by the degeneration and thinnin | ng ofthe epidermis and dermis. | 97 ts | | r e |
| kin hyperpigmentation | Hyperpigmentation covering<br><10% BSA; no psychosocial<br>impact | Hyperpigmentation colvering<br>>10 % BSA; associated<br>psychosocial impact | | | |
| Definition: A disorder charact | terized by darkening of the skin due to | excessive melanin deposition. | 57 th | | 7 |
| kin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering > 10 %<br>BSA; associated psychosocial<br>impact | | | 2 |
| lefinition: A disorder charact | terized by loss of skin pigment. | | | | |
| kin induration | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pin ching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration, unable to<br>slide or pinch skin; limiting joint<br>movement or orifice (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| lefinition: A disorder charact | terized by an area of hardness in the s | kin, | (5) | | (8)<br>(0) |
| kin ulceration | Combined area of ulcers <1 cm;<br>non blanchable erythema of<br>intact skin with a ssociated<br>warmth or edema | Combined area of ulcers 1 - 2<br>cm; partial thickness skin loss<br>involving skin or subcutaneous<br>fat | Combined area of ulcers >2 cm;<br>full-thickness skin loss involving<br>damage to ornecrosis of<br>sub outaneous tissue that may | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or supporting structures with or | Death |

CTCAE 4.0 - May 28, 2009 : Skin and subcutaneous tasse disorders

CARTISTEM® 

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome<br>Definition: A disorder characteri | -<br>zed by lessthan 10 % total body ski | In area separation of dermis. The | Skin sloughing covering <10% BSA with associated signs (e.g., erythema, purpura, epidermal detachment and mucous membrane detachment) syndrome is thought to be a hyper | Skin sloughing covering 10 -<br>30 % BSA with associated signs<br>(e.g., enythema, purpura,<br>epidermal detachment and<br>mucous membrane<br>detachment)<br>sensitivity complex affecting the s | Death Rin and the |
| nucous membranes. | | | | | |
| Telan giecta sia | Telangiectasias covering < 10 %<br>BSA | Telangie ctasias covering >10 %<br>BSA; associated with<br>psychosocial impact | | - | - |
| Definition: A disorder characteri | zed by local dilatation of small vess | els resulting in red discoloration o | of the skin or mucous membranes. | | 8<br> |
| Toxic epidermal necrolysis | | | | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| Definition: A disorder characteri<br>mucous membranes. | ্<br>zed by greater than 30% total body | rskin area separation of dermis. T | he syndrome is thought to be a hy | persensitivity complex affecting th | e skin and th |
| Urticaria | Urticarial Lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesion's covering 10 -<br>30 % BS A; oral intervention<br>indicated | Urticarial lesions covering >30 %<br>BSA; Mintervention indicated | | ē<br>ē |
| Definition: A disorder characteri | zed by an itchy skin eruption charac | cterized by wheals with pale inter | iors and well-defined red margins. | | |
| Skin and suboutaneous tissue<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin va sive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

CARTISTEM® 

| | V. | Social circumstar | nces | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | - 5 |
| Menopause | Menopause occurring at age 46 | - 45 | Menopause occurring before age 40 years of age | | |
| Definition: A disorder character<br>Social circumstances - Other, | ized by the permanent cessation of<br>Asymptomatic or mild | menses, usually defined by 12 co<br>Moderate; minimal, local or | Severe or medically significant | n a woman over 46 years of age.<br>Life-threatening consequences; | Death |
| specify | symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | urgent intervention indicated | 3 8860/04/2 |
| | | | disabling; limiting self care ADL | | |

CTCAE 4.0 - May 28, 2009 : Skin and subcutaneous tissue disorders 74 CTCAE 4.0 - May 28, 2009 : Social circumstances 75 CTCAE 4.0 - May 28, 2009 : Surgical and medical procedures 76

CARTISTEM® 

| | | Surgical and medical p | l procedures | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Surgical and medical procedures - Other, specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations<br>only; intervention not<br>indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately life-<br>threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Life-threatening<br>consequences; urgent<br>intervention indicated | Death |

CARTISTEM® 

| | Vascular disorders | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Capillary leak syndrome | - | Symptomatic; medical intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | zed by leakage of intra vascular flui<br>: syndromes, low-flow states, ischei | | | 경우 이 10 원인 이 아이를 보고 있습니다. 일본 이 전 보고 있는 것이 하고 하고 있다. | |
| Flushing | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical<br>intervention indicated; limiting<br>instrumental ADL | Symptomatic, associated with<br>hypotension and/or tachycardia;<br>limiting self care ADL | | - |
| Definition: A disorder characteri | zed by episodic reddening ofthe fa | ce. | I. | | |
| Hematoma | Mild symptoms; intervention not indicated | Minimally in vasive evacuation or aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a localized collection of bloo | id, u sually clotted , in an organ , sp: | ace, or tissue, due to a break in th | e wall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by an uncomfortable and temp | orary sensation of intense body wa | armth , flushing , sometime s accom | panied by sweating upon cooling. | 0 |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic BP 140 - 159 mm Hg or diastolic BP 90 -99 mm Hg); medical intervention indicated; recurrent or persistent (>24 hrs); symptomatic increase by >20 mm Hg (diastolic) orto >140,90 mm Hg if previously WNL; monotherap y indicated. Pediatric: recurrent or persistent (>24 hrs) BP >ULN; monotherap y indicated | Stage 2 hypertension (systolic BP >= 160 mm Hg or diastolic BP >= 100 mm Hg); medical intervention indicated; more than one drug or more intensive therapythan previously used indicated Pediatric: Same as adult | Life-threatening consequences (e.g. malignant hypertension, transient or permanent neurologic de foit, hypertensive crisis); urgent intervention indicated Pediatric: Same as a dult | Death |
| Definition: A dispersor sharmstori | I<br>zed by a pathological increase in bl | | <br>ion in the blood proceum exceeding | l<br>na 140 ovor 00 mm Ha | E. |
| Hypotension | Asymptomatic, intervention not<br>indicated | Non-urgent medical intervention<br>indicated | Medical intervention or hospitalization indicated | Life-threatening and urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a blood pressure that is belo | ow the normal expected for an indi | vidual in a given environment. | | 81 |
| Lymph leakage | | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention in dicated | Death |
| | zed by the loss of lymph fluid into th<br>T | No. 1970 - 1970 | · | | |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery<br>skin texture; papillary formation;<br>limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL | | - |
| Definition: A disorder characteri | zed by excessive fluid collection in: | tissues that causes swelling. | T 2 | | |
| Lymphocele | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | | - |
| Definition: A disorder characteri | zed by a cystic lesion containing lyr | nph. | 0 V | | 0 |
| Peripheral ischemia | | Brief (<24 hrs) episode of<br>ischemia managed non-<br>surgically and without<br>permanent deficit | Recurring or prolonged (>=24<br>hrs) and/or in vasive intervention<br>indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| T. | zed by impaired circulation to an ex | I. | | | |
| Phlebitis | 1- | Present | - | -8 | + |
| PRINCIPAL STREET, STRE | zed by inflammation of the wall of a | vein. | Ť | | 1 |
| Superficial thrombophlebitis | to an institution of | Present | lo | 13 | - |
| Definition: A disorder characteri | zed by a blood clot and inflammatio | n involving a superficial vein of the | e extremities. | | |

CTCAE 4.0 - May 28 , 2009 : Vascular disorders

CARTISTEM® 

| Vascular disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1. | 2 | 3 | 4 | 5 |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening consequences;<br>urgent multi-modality<br>intervention indicated (e.g.,<br>lysis, thrombectomy, surgery) | Death |
| Definition: A disorder character<br>cough, orthopnea and headach | ized by obstruction of the blood flow | in the superior vena cava. Sign: | s and symptoms include swelling ar | nd cyanosis of the face, neck, and | upperarn |
| Thrombo embolic e vent | Ven ous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | Thrombosis (e.g.,<br>uncomplicated pulmonary<br>embolism [venous], non-embolic<br>cardiac mural [arterial]<br>thrombus), medical intervention<br>indicated<br>a distal site via the blood stream. | Life-threatening (e.g., pulmonary embolism, cerebrovascular event, arterial insufficiency); hemodynamic or neurologic instability; urgent intervention indicated | Death |
| Va sculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening; evidence of peripheral or visceral ischemia; urgent intervention indicated | Death |
| Definition: A disorder character | ized by inflammation involving the w | all of a vessel. | | | |
| Msoeral arterial ischemia | | Brief (<24 hrs) episode of<br>ischemia managed medically<br>and without permanent deficit | Prolonged (>=24 hrs) or recurring symptoms and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a decrease in blood supply ( | due to narrowing or blockage of: | a visceral (mesenterio) arteny. | | ** |
| Vascular disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>nonin va sive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not imme diately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

CARTISTEM® 



CTCAE 4.0 - May 28, 2009 : Vascular disorders 78

NIH Publication No. 03-5410 Revised May 2009 Reprinted May 2009



CARTISTEM® 

**CONFIDENTIAL:** These all contents herein are the sole property of MEDIPOST Co., Ltd. Any reproduction or distribution of this document without the written consent of MEDIPOST Co., Ltd is prohibited. Copyright © 2017 MEDIPOST Co., Lt

## APPENDIX 5. IDMC charter

## 1. Composition of Data Safety Monitoring Boards (DSMB)

In the present clinical trial study for Evaluation of Safety and Exploratory Efficacy of CARTISTEM®, Data Safety Monitoring Boards (DSMB) consists of 3 members who are experts in the area of orthopedics, cell therapies or biostatistics. The members will be independent from the sponsor, IRB, regulatory agencies, principal investigator, co-principal or sub-principal investigator, site investigator, site sub-investigator, steering committee membership, advisory board membership, CEC membership, clinical care of the study subjects, or any other capacity related to the present clinical trial operations.

## 2. Frequency of DSMB meetings

DSMB meets periodically to review aggregate and individual subject data related to safety, data integrity and overall conduct of the trial. DSMB meetings will be organizational face-to-face and quarterly teleconferences. However, given the small sample size for the present clinical study, the DSMB meetings will be flexible and based on enrollment of patients.

According to the schedule, the DSMB meetings will be required 1) for protocol revision, 2) before the dosage B started and 3) to review a draft final report after 12 month follow-up period.

## 3. Information to be reviewed at each meeting

In order for the DSMB members to review all the information at each meeting, guidance for the conduct of safety and effectiveness analyses, protocol modification if applicable, and guidelines/stopping rules will be established prior to the DSMB's first evaluation of data. The DSMB will review data unblinded fashion.

The DSMB will also consider data from other studies or external sources during its deliberations, if available, as these results may have a profound impact on the status of the patients and design of the present study.

CARTISTEM® 